#### NRG ONCOLOGY Radiation Therapy Oncology Group

#### **RTOG 1115**

(ClinicalTrials.gov NCT #: 01546987)

Phase III Trial of Dose Escalated Radiation Therapy and Standard Androgen Deprivation Therapy (ADT) with a GnRH Agonist vs. Dose Escalated Radiation Therapy and Enhanced ADT with a GnRH Agonist and TAK-700 for Men with High Risk Prostate Cancer

Amendment 3: June 12, 2018

#### **RTOG 1115**

# PHASE III TRIAL OF DOSE ESCALATED RADIATION THERAPY AND STANDARD ANDROGEN DEPRIVATION THERAPY (ADT) WITH A GNRH AGONIST VS. DOSE ESCALATED RADIATION THERAPY AND ENHANCED ADT WITH A GNRH AGONIST AND TAK-700 FOR MEN WITH HIGH RISK PROSTATE CANCER

This trial is part of the National Clinical Trials Network (NCTN) program, which is sponsored by the National Cancer Institute (NCI). The trial will be led by NRG Oncology with the participation of the network of NCTN organizations: the Alliance, ECOG-ACRIN, and SWOG.

Study Chairs (12Jun2018)

| Study Chairs (12Jun2018) | |
|---|---|
| Principal Investigator/Medical Oncology | Radiation Oncology Co-Chair |
| M. Dror Michaelson, MD, PhD | Daniel Hamstra, MD, PhD |
| Massachusetts General Hospital | William Beaumont Hospital |
| 32 Fruit Street, Yaw 7E | 18101 Oakwood Blvd. |
| Boston, MA 02114 | Dearborn, MI 48124 |
| Phone: 617-726-1594/Fax: 617-726-3440 | Phone: 313-593-3773/Fax: 313-593-8844 |
| E-mail: dmichaelson1@partners.org | E-mail: <u>Daniel.Hamstra@Beaumont.org</u> |
| Brachytherapy Co-Chair | <u>Urology Co-Chair</u> |
| François Bachand, MD, FRCPC | Viraj Master, MD PhD |
| Radiation Oncology | Emory University |
| BC Cancer Agency | Emory Clinic Building B-1400 |
| Center for Southern Interior | 1365 Clifton Road, NE |
| 399 Royal Avenue | Atlanta, GA 30322 |
| Kelowna, BC | Phone: 404-778-4898 |
| V1Y 5L3 | E-mail: virajmaster@gmail.com |
| Phone: 250-979-6645/Fax: 250-712-3911 | |
| E-mail: FBachand@bccancer.bc.ca | |
| Outcomes Co-Chair | Fatigue Co-Chair |
| Deborah Watkins Bruner, RN, PhD, FAAN | Mylin A. Torres, MD |
| Nell Hodgson Woodruff School of Nursing | Department of Radiation Oncology |
| Emory University | Emory University School of Medicine |
| 1520 Clifton Road, Room 232 | 1365-C Clifton Road Northeast |
| Atlanta, GA 30322 | Clinic C Suite 3012 |
| Phone: 404-712-9695/Fax: 404-727-8514 | Atlanta, GA 30322 |
| E-mail: deborah.w.bruner@emory.edu | Phone: 404-778-3473/Fax: 404-778-4139 |
| | E-mail: matorre@emory.edu |
| Translational Research Co-Chair | Medical Physics Co-Chair |
| Philip J. Saylor, MD | Robert E. Wallace, PhD |
| Massachusetts General Hospital Cancer Center | Cedars-Sinai Medical Center |
| 55 Fruit Street, Yaw 7E | Department of Radiation Oncology |
| Boston, MA 02114 | 8700 Beverly Boulevard |
| Phone: 617-724-4000/Fax: 617-726-8685 | Los Angeles, CA 90048 |
| E-mail: psaylor@partners.org | Phone: 310-423-1113 |
| | E-mail: robert.wallace@cshs.org |

#### **RTOG 1115**

Study Chairs (continued)

<u>Senior Statistician</u> James J. Dignam, PhD

NRG Oncology Statistical and Data Management Center & The University of Chicago Biological

Sciences

1818 Market Street, Suite 1720

Philadelphia, PA 19103

Phone: 215-574-3174/Fax: 215-928-0153

E-mail: dignamj@nrgoncology.org

Radiation Oncology Co-Chair/ECOG

Neha Vapiwala, MD

Perelman Center for Advanced Medicine

Radiation Oncology

3400 Civic Center Boulevard Fourth Floor West Pavilion Philadelphia, PA 19104

Phone: 215-662-2337

E-mail: vapiwala@uphs.upenn.edu

#### **Protocol Agent**

| Agent | Supply | NSC # | IND # |
|---------------------------|------------|-------|--------|
| TAK-700 | Millennium | N/A | 115368 |
| Leuprolide<br>Goserelin | Commercial | N/A | Exempt |
| Buserelin<br>Triptorelin | | | |
| Flutamide<br>Bicalutamide | | | |

#### **Participating Sites:**

□ U.S. and Canada

#### **Document History**

| | Version/Update Date | Broadcast Date |
|-------------|---------------------|--------------------|
| Amendment 3 | June 12, 2018 | N/A |
| Closure | | September 30, 2014 |
| Amendment 2 | April 16, 2014 | June 17, 2014 |
| Update | February 4, 2014 | February 4, 2014 |
| Amendment 1 | December 17, 2013 | February 4, 2014 |
| Update | February 5, 2013 | February 5, 2013 |
| Update | August 9, 2012 | August 9, 2012 |
| Update | May 2, 2012 | May 2, 2012 |
| Update | May 1, 2012 | May 1, 2012 |
| Activation | February 10, 2012 | May 1, 2012 |

#### NRG Oncology 1-800-227-5463, ext. 4189

This protocol was designed and developed by NRG Oncology. It is intended to be used only in conjunction with institution-specific IRB approval for study entry. No other use or reproduction is authorized by NRG Oncology nor does NRG Oncology assume any responsibility for unauthorized use of this protocol.

#### **RTOG 1115**

PHASE III TRIAL OF DOSE ESCALATED RADIATION THERAPY AND STANDARD ANDROGEN DEPRIVATION THERAPY (ADT) WITH A GNRH AGONIST VS. DOSE ESCALATED RADIATION THERAPY AND ENHANCED ADT WITH A GNRH AGONIST AND TAK-700 FOR MEN WITH HIGH RISK PROSTATE CANCER

| CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION (12Jun2018) | | |
|---|---|---|
| To submit site registration documents: | For patient enrollments: | Submit study data directly to the Lead Cooperative Group unless otherwise specified in the protocol: |
| Regulatory documentation can be submitted to the CTSU via: ONLINE: Regulatory Submission Portal (Sign in at www.ctsu.org, and select the Regulatory Submission sub-tab under the Regulatory tab.) | Please refer to the patient enrollment section for instructions on using the OPEN system. Contact the CTSU Help Desk with any OPEN-related questions at ctsucontact@westat.com. | Data collection for this study will be done exclusively through Medidata Rave. Please see the data submission section of the protocol for further instructions. Do not submit study data or forms to CTSU Data Operations. Do not copy the CTSU on data submissions. |

The most current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>. Access to the CTSU members' web site is managed through the Cancer Therapy and Evaluation Program - Identity and Access Management (CTEP-IAM) registration system and requires user log on with CTEP-IAM username and password.

- For patient eligibility or treatment-related questions Contact the Study PI of the Lead Protocol Organization
- For questions unrelated to patient eligibility, treatment, or data submission contact the CTSU Help Desk by phone or e-mail:
- CTSU General Information Line 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

For detailed information on the regulatory and monitoring procedures for CTSU sites please review the CTSU Regulatory and Monitoring Procedures policy located on the CTSU members' website <a href="https://www.ctsu.org">https://www.ctsu.org</a> > education and resources tab > CTSU Operations Information > CTSU Regulatory and Monitoring Policy

The CTSU Web site is located at https://www.ctsu.org

The following Cooperative Groups have endorsed this trial: ECOG: Co-Chair: Neha Vapiwala, MD. ECOG members will enroll patients to this study via the Cancer Trials Support unit (CTSU).

#### **Table of Contents**

| | 1115 | |
|---|---|---|
| | MA | |
| | BILITY CHECKLIST | |
| 1.0 | INTRODUCTION | |
| 1.1 | Background | 12 |
| 1.2 | Adjuvant/concurrent/neoadjuvant ADT with Radiation Therapy | |
| 1.3 | Safety of Proposed Therapy | |
| 1.4 | Prostate Cancer Survivorship | |
| 1.5 | Fatigue | |
| 2.0 | OBJECTIVES | |
| 2.1 | Primary Objective | |
| 2.2 | Secondary Objectives | |
| 3.0 | PATIENT SELECTION | |
| 3.1 | Conditions for Patient Eligibility | |
| 3.2 | Conditions for Patient Ineligibility) | 18 |
| 4.0 | PRETREATMENT EVALUATIONS/MANAGEMENT | |
| 4.1 | Required Evaluations/Management | |
| 5.0 | REGISTRATION PROCEDURES | |
| | ess Requirements for OPEN, Medidata Rave®, and TRIAD | |
| 5.1 | Pre-Registration Requirements for IMRT Treatment Approach | |
| 5.2 | Pre-Registration Requirements for 3DCRT Treatment Approach | |
| 5.3 | Pre-Registration Requirements for Brachytherapy Treatment Approach | ۱ ک |
| 5.4<br>5.5 | Digital RT Data Submission to RTOG Using TRIADRegulatory Pre-Registration Requirements) | |
| 5.6 | OPEN Registration | |
| 6.0 | RADIATION THERAPY | |
| 6.1 | Two Stage Radiation Plan | |
| 6.2 | Technical Factors | |
| 6.3 | EBRT Localization, Simulation, and Immobilization | |
| 6.4 | Treatment Planning/Target Volumes | |
| 6.5 | Critical Structures | |
| 6.6 | Treatment Verification | |
| 6.7 | Quality Assurance | |
| 6.8 | Dose Specifications/Technical Considerations: LDR Brachytherapy Boost | |
| 6.9 | Dose Specifications/Technical Considerations: HDR Brachytherapy Boost | |
| 6.10 | | |
| 6.11 | • | |
| 6.12 | | |
| 7.0 | DRUG THERAPY | |
| 7.1 | Treatment | |
| 7.2 | LHRH agonists (such as leuprolide, goserelin, buserelin, triptorelin) | 36 |
| 7.3 | Eulexin (flutamide) | 37 |
| 7.4 | Casodex (bicalutamide) | 37 |
| 7.5 | Study Drug (TAK-700) Administration (TAK-700, IND # 115368) | 38 |
| 7.6 | TAK-700 Dose Modification and Supportive Care Guidelines | 38 |
| 7.7 | Excluded Concomitant Medications and Procedures | |
| 7.8 | Precautions and Restrictions | |
| 7.9 | Blinding and Unblinding | |
| 7.10 | 1 5 5 | |
| 7.11 | | |
| 7.12 | | |
| 7.13 | Storage, Handling, and Accountability | 42 |

| 7.14 | Supply | 43 |
|---|---|---|
| 7.15 | Modality Reviews | 44 |
| 7.16 | Adverse Events | 45 |
| 7.17 | CTEP-AERS Adverse Event Reporting Requirements | 46 |
| 8.0 | SURGERY | 47 |
| 9.0 | OTHER THERAPY | 48 |
| 9.1 | Permitted Supportive Therapy | 48 |
| 9.2 | Non-permitted Supportive Therapy | |
| 10.0 | TISSUE/SPECIMEN SUBMISSION | |
| 10.1 | Tissue/Specimen Submission | |
| 10.2 | Specimen Collection for Translational Research (Mandatory) | |
| 10.3 | Specimen Collection for Tissue Banking and Translational Research (Strongly Recommendational Research (Strongly Recommendation Recommendation | |
| ` | 7/13) | |
| 10.4 | Storage Conditions | 51 |
| 10.5 | Submit materials for Tissue Banking and Translational Research | |
| 10.6 | Reimbursement | |
| 10.7 | Confidentiality/Storage | |
| 11.0 | PATIENT ASSESSMENTS | |
| 11.1 | Study Parameters | |
| 11.2 | PROMIS-Fatigue Short Form | |
| 11.3 | Health Related Quality of Life (HRQOL) Assessments | |
| 11.4 | Criteria for Discontinuation of Protocol Treatment | |
| 12.0 | DATA COLLECTION | |
| 12.1 | Summary of Data Submission | |
| 12.2 | Summary of Dosimetry Digital Data Submission | 58 |
| 13.0 | STATISTICAL CONSIDERATIONS | |
| 13.1 | Primary Endpoint | |
| 13.2 | Secondary Endpoints | |
| 13.3 | Sample Size Determination | |
| 13.4 | Randomization | |
| | Analysis Plan | |
| 13.6 | Gender and Minorities | |
| KEFEF | RENCES | 67 |
| | IDIX I, STUDY PARAMETER TABLE: PRE-TREATMENT ASSESSMENTS (12/17/13) | |
| | IDIX II | |
| | IDIX III | |
| | IDIX IV | |
| | IDIX V | |
| | IDIX VI | 08 |
| | II II A VIII | χu |

#### **RTOG 1115**

Phase III Trial of Dose Escalated Radiation Therapy and Standard Androgen Deprivation Therapy (ADT) with a GnRH Agonist vs. Dose Escalated Radiation Therapy and Enhanced ADT with a GnRH Agonist and TAK-700 for Men with High Risk Prostate Cancer

#### **SCHEMA**

(12/17/13)

| 11/10/ | | T |
|---|---|---|
| Risk Groups 1. Gleason ≥ 9, PSA ≤ 150, any T-stage 2. Gleason 8, PSA < 20, and ≥ T2 3. Gleason 8, PSA ≥ 20-150, any T-stage 4. Gleason 7, PSA ≥ 20-150, any T-stage | R A N D O M I Z E (1:1) | Arm 1: Androgen Deprivation Therapy: GnRH agonist for 24 months with concurrent oral antiandrogen until completion of radiation + Dose Escalated Radiation: To start 8-10 weeks after initiation of ADT. Initially, 45 Gy to prostate and pelvic lymph nodes delivered with 3DCRT/IMRT with a boost to be provided with IMRT, LDR implant, or HDR implant. |
| Type of RT Boost 1. IMRT 2. Brachytherapy (LDR using PPI or HDR) | | Arm 2: Androgen Deprivation Therapy: GnRH agonist for 24 months with concurrent oral antiandrogen until completion of radiation + TAK-700 twice daily for 24 months |
| ADT Started Prior to Registration 1. No 2. Yes | | + <u>Dose Escalated Radiation</u> : To start 8-10 weeks after initiation of ADT. Initially, 45 Gy to prostate and pelvic lymph nodes delivered with 3DCRT/IMRT with a boost to be provided with IMRT, LDR implant, or HDR implant. |
| | <ol> <li>Gleason ≥ 9, PSA ≤ 150, any T-stage</li> <li>Gleason 8, PSA &lt; 20, and ≥ T2</li> <li>Gleason 8, PSA ≥ 20-150, any T-stage</li> <li>Gleason 7, PSA ≥ 20-150, any T-stage</li> <li>Type of RT Boost</li> <li>IMRT</li> <li>Brachytherapy (LDR using PPI or HDR)</li> <li>ADT Started Prior to Registration</li> <li>No</li> </ol> | 1. Gleason ≥ 9, PSA ≤ 150, any T-stage 2. Gleason 8, PSA < 20, and ≥ T2 3. Gleason 8, PSA ≥ 20-150, any T-stage 4. Gleason 7, PSA ≥ 20-150, any T-stage Type of RT Boost 1. IMRT 2. Brachytherapy (LDR using PPI or HDR) ADT Started Prior to Registration 1. No |

See pre-registration requirements in Section 5.0. See Section 7.0 for details/doses of study drug.

#### Patient Population: (See Section 3.0 for Eligibility)

Histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days prior to registration at high risk for recurrence as determined by one of the following combinations:

| Gleason score | | <u>PSA</u> | | <u>T-Stage</u> |
|---------------|-----|--------------------|-----|----------------|
| <u>&gt;</u> 9 | and | <u>&lt;</u> 150 | and | Any |
| 8 | and | < 20 | and | <u>&gt;</u> T2 |
| 8 | and | <u>&gt;</u> 20-150 | and | Any |
| 7 | and | <u>&gt;</u> 20-150 | and | Any |

Required Sample Size: 900

### **ELIGIBILITY CHECKLIST** (4/16/14)

| |
|---|
| NRG Oncology Institution # RTOG 1115 Case # |
| 1(Y) Does the patient have a histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days prior to registration? |
| 2(Y) Was a history/physical examination done within 60 days prior to registration? |
| 3(Y) Did the patient have clinically negative lymph nodes within 90 days prior to registration demonstrated by imaging (abdominal <u>and/or</u> pelvic CT or MRI) which if deemed equivocal or questionable the nodes are less than 2.0 cm or negative nodes per nodal sampling or dissection? |
| 4(Y) Did a bone scan demonstrate no distant metastases (M0) within 90 days prior to registration (18F-Na PET is an acceptable substitute)—and if the bone scan was equivocal were plain films negative? |
| 5(Y) Was the study entry (baseline) PSA performed with an FDA approved assay within 180 days prior to registration and prior to the start of any hormone ablation therapy? |
| 6N/Y Was ADT started prior to registration (must be 50 days or less from registration)? If yes: Date started Drug(s) started Please note: If patient has started ADT prior to registration, he is not eligible to participate in the quality of life component of this study. |
| 7(N) Did the patient have testosterone administered within 90 days prior to registration? |
| 8(Y) Is the patient's performance status 0 or 1 documented within 21 days prior to registration? |
| 9(Y) Is the patient's age 18 years or greater? |
| <ul> <li>10(Y) Has a CBC with differential been obtained within 14 days prior to registration demonstrating adequate bone marrow function as follows?</li> <li>Absolute neutrophil count (ANC) ≥ 1800 cells/mm³</li> <li>Platelets ≥ 100,000 cells/mm³</li> <li>Hemoglobin ≥ 8.0 g/dl</li> </ul> |
| 11. Y) Has a serum creatinine with a value of <2.0 ng/dL and a creatinine clearance (calculated can |

- be used) showing 40 mL/min been obtained within 21 days prior to registration?
- (Y) Has a total bilirubin with a value of < 1.5x the institutional ULN and an ALT or AST < 2.5x the institutional ULN been obtained within 21 days prior to registration?
- 13. (Y) Has serum testosterone been obtained within 21 days prior to registration?
- (Y) Has a chemistry panel (including sodium, potassium, chloride, bicarbonate (carbon dioxide), BUN, glucose, calcium, magnesium and phosphorus) and liver studies (including albumin and alkaline phosphatase) been obtained within 21 days prior to registration?
- (Y) Has a fasting glucose, fasting insulin, lipid panel (cholesterol, triglyceride, HDL, LDL), and Hemoglobin A1C been obtained within 21 days prior to registration?

#### NRG Oncology Institution # RTOG 1115 Case #

## ELIGIBILITY CHECKLIST (12/17/13) 

| 16(Y) Has a screening calculated ejection fraction been obtained by multiple gated acquisition (MUGA) scan or by echocardiogram (ECHO) demonstrating a result of ≥ to institutional lower limit of normal? |
|---|
| 17(Y) Has a baseline ECG been obtained within 180 days prior to registration? |
| 18(Y/N/A) If the patient is a man of child-producing potential has he agreed to use effective contraception while on treatment and for at least 120 days after treatment has been completed? |
| 19(Y) Is the patient able to provide study specific informed consent prior to study registration? |
| 20(Y) Does the patient demonstrate a high risk for prostate cancer recurrence as determined by one of the following combinations? |
| Gleason score ≥ 9 and PSA ≤ 150 and Any T-stage |
| Gleason score 8 and PSA < 20 and T-stage ≥ T2 |
| Gleason score 8 and PSA ≥ 20-150 and Any T-stage |
| Gleason score 7 and PSA ≥ 20-150 and Any T-stage |
| What is the Gleason score? |
| What is the PSA value? |
| What is the T-stage? |
| 21(N) Is the PSA value > 150? |
| 22(N) Is there evidence of metastatic disease? |
| 23(N) Are there pathologically positive pelvic lymph nodes or pelvic lymph nodes > 2.0 cm demonstrated by imaging (CT or MR)? |
| 24(N) Has the patient had a radical prostatectomy, cryosurgery for prostate cancer or a bilateral orchiectomy for any reason? |
| 25(N) Has the patient had a prior invasive malignancy (except non-melanoma skin cancer) unless disease free or not requiring systemic therapy for a minimum of 3 years? |
| 26(N) Has the patient had prior systemic chemotherapy for prostate cancer? |
| 27(N) Has the patient had prior radiotherapy, including brachytherapy, to the region of the prostate that would result in overlap of radiation therapy fields? |
| 28(N) Has the patient had previous hormonal therapy for > 50 days prior to registration? |
| 29(N) Does the patient have a known hypersensitivity to TAK-700 or related compounds or |

#### NRG Oncology Institution # RTOG 1115 Case #

# ELIGIBILITY CHECKLIST (12/17/13) 

| 30(N) Has the study entry PSA been obtained during either of the following time frames: |
|---|
| 10 day period following a prostate biopsy or following the initiation of hormonal therapy? |
| 31 (N) Does the patient have a history of adrenal insufficiency? |
| <ul> <li>(N) Does this patient have any severe or active co-morbidities as defined by the following?</li> <li>A major surgical procedure within 14 days prior to registration</li> <li>Ongoing arrhythmias (greater than grade 2); thromboembolic events or any other cardiac condition (such as pericardial effusion, etc.) within 6 months prior to registration</li> <li>Class III or IV heart failure per New York Heart Association classification</li> <li>ECG abnormalities: <ul> <li>-Q-wave infarction unless identified more than 6 months prior to registration</li> <li>-QTc interval greater than 460 msec</li> <li>Chronic liver disease (bilirubin &gt; 1.5 x ULN; ALT or AST &gt; 2.5x ULN)</li> <li>Serious infection within 14 days prior to registration</li> <li>Unstable symptomatic ischemic heart disease</li> <li>History of myocardial infarction</li> </ul> </li> </ul> |
| 33(N) Does the patient have a history of Cushing's syndrome? |
| 34(N) Does the patient have a history of severe chronic renal disease demonstrated by a serum Creatinine > 2.0 mg/dl and a Creatinine clearance of < 40 mL/min? |
| 35(N) Has the patient had chronic treatment with glucocorticoids within the last year? |
| 36(N) Does the patient have uncontrolled hypertension despite appropriate medical therapy characterized by a blood pressure of greater than 150 mm Hg systolic and 90 mm Hg diastolic at two separate measurements no more than 60 minutes apart within 21 days prior to registration? |
| 37(N) Does the patient have uncontrolled nausea, vomiting or diarrhea (grade 3 or greater) despite appropriate medical therapy at the time of registration? |
| 38(N) Does the patient have a known gastrointestinal disease or procedure that might interfere with the oral absorption or tolerance of TAK-700, including difficulty swallowing tablets at the time of registration? |
| 39(Y) Even if surgically sterilized (vasectomy), does the patient agree to practice effective barrier contraception during the entire study treatment period and for (4) months after the last dose of study drug or abstain from intercourse completely? |

### <u>ELIGIBILITY CHECKLIST</u> (12/17/13) (2/4/14) 

### The following questions will be asked at Study Registration: IMRT CREDENTIALING IS REQUIRED BEFORE REGISTRATION

| | 1. | Institutional person randomizing case. |
|---|---|---|
| (Y) | 2. | Has the Eligibility Checklist been completed? |
| (Y) | 3. | In the opinion of the investigator, is the patient eligible? |
| | 4. | Date informed consent signed |
| | 5. | Patient's Initials (First Middle Last) |
| | 6. | Verifying Physician |
| | 7. | Patient ID |
| | 8. | Date of Birth |
| | 9. | Race |
| | 10. | Ethnicity |
| | 11. | Gender |
| | 12. | Country of Residence |
| | 13. | Zip Code (U.S. Residents) |
| | 14. | Method of Payment |
| | 15. | Any care at a VA or Military Hospital? |
| | 16. | Calendar Base Date (date hormone ablation to start—if hormones started prior to registration use today's date) |
| | 17. | Randomization date |
| (Y/N) | 18. | Have you obtained the patient's consent for his or her tissue to be kept for use in research to learn about, prevent, treat, or cure cancer? |
| (Y/N) | 19. | Have you obtained the patient's consent for his or her blood to be kept for use in research to learn about, prevent, treat, or cure cancer? ( <b>Note</b> : Blood collection is mandatory for patients participating in QOL). |
| (Y/N) | 20. | Have you obtained the patient's consent for his or her tissue to be kept for use in research about other health problems (for example: causes of diabetes, Alzheimer's disease, and heart disease)? |
| (Y/N) | 21. | Have you obtained the patient's consent for his or her blood to be kept for use in |

## ELIGIBILITY CHECKLIST (4/16/14) 

| | research about other health problems (for example: diabetes, Alzheimer's disease, or heart disease). ( <b>Note</b> : Blood collection is mandatory for patients participating in QOL). |
|---|---|
| (Y/N) 22. | Have you obtained the patient's consent to allow someone from this institution to contact him or her in the future to take part in more research? |
| Note: If the patient st component. | Did the patient agree to participate in the quality of life component? If no, please specify the reason from the following: 1. Patient refused due to illness 2. Patient refused for other reason: specify 3. Not approved by institutional IRB 4. Tool not available in patient's language 5. Other reason: specify tarted ADT prior to registration, then he cannot participate in the quality of life |
| 24. | Risk group (specify): 1. Gleason ≥ 9, PSA ≤ 150, any T-stage 2. Gleason 8, PSA < 20, and ≥ T2 3. Gleason 8, PSA ≥ 20-150, any T-stage 4. Gleason 7, PSA ≥ 20-150, any T-stage |
| (N/Y) 25. | Androgen deprivation therapy (ADT) started prior to registration? If yes, treatment start date (Must be ≤50 days from registration): |
| 26. | RT Modality for boost (specify): 1. IMRT 2. LDR Permanent Prostate Implant (PPI) Boost 3. HDR Boost |
| ( N/Y) 27. | Use of IMRT |
| and dated checklist us | st must be completed in its entirety prior to web registration. The completed, signed, sed at study entry must be retained in the patient's study file and will be evaluated NCI/NRG Oncology audit. |
| Completed by | Date |

#### 1.0 INTRODUCTION

#### 1.1 Background

Prostate cancer is the most common cancer in men. Androgen deprivation therapy (ADT) with gonadotropin releasing hormone (GnRH) agonists is the foundation of advanced prostate cancer treatment and is given as neoadjuvant/concomitant/adjuvant treatment with radiation for intermediate and high risk localized disease. GnRH agonist therapy causes cessation of gonadal androgen production, resulting in a reduction in serum testosterone levels by more than 95% and estrogen levels by approximately 80%. Adrenal androgen synthesis accounts for most of the small persistent level of serum androgens.

TAK-700 is an oral, selective nonsteroidal inhibitor of (Keating 2006, Eri 1995) lyase that blocks synthesis of both gonadal and adrenal dehydroepiandrosterone sulfate (DHEA) and androstenedione. TAK-700 has been shown to further reduce serum testosterone levels in men already maintained on a GnRH agonist. In Phase I and II clinical trials in men with advanced prostate cancer, TAK-700 has demonstrated notable efficacy with excellent tolerability (Dreicer 2010a, Dreicer 2010b). The most common adverse effects have included fatigue, nausea and constipation, and are generally mild in nature. TAK-700 has been administered alone to a maximum recommended dose of 300 mg BID, and together with low-dose prednisone to a maximum dose of 600 mg BID. In two ongoing, pivotal phase III trials, TAK-700 is being administered at either 400 mg BID along with 5 mg daily of prednisone (metastatic prostate cancer) or 300 mg BID without prednisone (nonmetastatic prostate cancer).

#### 1.2 Adjuvant/concurrent/neoadjuvant ADT with Radiation Therapy

Risk stratification of patients prior to primary therapy for prostate cancer yields important prognostic information and can be used to guide therapeutic choices. Three factors that are independently associated with relapse risk are clinical tumor stage, Gleason score, and pretreatment PSA level (Chism, 2004, D'Amico 2002, Levegrun 2002, Pisansky 1997, Symon 2003). Prostate cancer is categorized as high risk if it features extraprostatic extension (T3), Gleason > 8, or PSA > 20. Standard-of-care for men with high risk disease treated with external beam radiation is 2 – 3 years of ADT with a GnRH agonist based on phase III trials demonstrating an overall survival benefit (Bolla 1997, Pilepich 2005, Mohler 2010). Recently reported data from an EORTC trial comparing 6 months of ADT to 3 years of ADT for men with locally advanced disease showed a significant 5 year overall survival advantage for the longer term ADT group (15.2% vs. 19.0% mortality) (Bolla 2009). Efforts to achieve further benefit through intensified systemic therapy for this patient population led to RTOG 05-21, a randomized phase III trial in which adjuvant docetaxel chemotherapy was added to standard radiation and neoadjuvant/ concomitant/adjuvant ADT. RTOG 05-21 has completed accrual, but analysis is still several years away.

Though standard ADT with a GnRH agonist has clearly been shown to improve the efficacy of radiation therapy, no trial has yet built upon this foundation with the use of more profound androgen deprivation in this clinical setting. We propose to examine the combination of radiation with enhanced ADT using a GnRH agonist and TAK-700. This combination of hormonal agents has been shown to suppress serum testosterone to undetectable levels. Given the survival benefit conferred by lowering serum androgens with 2-3 years of GnRH agonist treatment in combination with radiation for high risk prostate cancer, we hypothesize that further lowering of serum androgens will produce additional clinical benefit.

#### 1.3 Safety of Proposed Therapy

Based upon experience from phase I and ongoing II and III trials, TAK-700 is generally well tolerated when given in combination with a GnRH agonist. Adverse events that have been observed to occur frequently include fatigue, nausea, constipation, anorexia and vomiting (Dreicer 2010a, Dreicer 2010b) The most prominent safety concerns are primarily related to the risk of hypertension and electrolyte abnormalities secondary to mineralocorticoid excess, an effect that has been observed with other lyase inhibitors (Attard 2005, Attard 2008). However, this has generally not been a concern in early trials with TAK-700. In this study, electrolytes including serum potassium will be monitored regularly.

No completed study has examined the combination of TAK-700 with a GnRH agonist and concurrent radiation. Though the tolerability of this combination is anticipated to be similar to that of radiation with concurrent GnRH agonist therapy, the absence of unexpected adverse events must be verified and is a co-primary endpoint of the study. Formal toxicity assessment will be carried out after follow-up of 200 patients (100 per treatment arm) through six months of therapy. Adverse events will be measured by NCI

CTCAE criteria and compared between arms. The trial will be halted if unacceptable levels of toxicity are found among patients randomized to TAK-700 relative to standard ADT, with threshold criteria for excess incidence derived from observed adverse event data from similar patients who underwent radiation and ADT per the control arm of this trial. If the toxicity profile is acceptable as defined in <a href="Section 13.5.7">Section 13.5.7</a>, the trial will continue to full accrual. Quality of life measured by the EPIC (32 item) and EQ-5D (5 item) questionnaires and fatigue measured by the Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Scale also will be examined as supporting information regarding tolerability of TAK-700. In addition to this early safety assessment and continuous CTCAE adverse event monitoring throughout the trial, detailed studies with respect to both short and long term potential adverse consequences of TAK-700 will be conducted, as described in <a href="Sections 1.4">Sections 1.4</a> and <a href="1.5">1.5</a>.

#### 1.4 Prostate Cancer Survivorship

A major consideration in the treatment of prostate cancer is achievement of a satisfactory risk-benefit ratio with respect to treatment. While men with disease meeting disease stage criteria here are deemed high-risk and thus candidates for multimodality therapy including 2-year androgen deprivation, their likelihood to non-cancer morbidity and mortality may still exceed their prostate cancer mortality risk, and thus it is necessary to carefully assess the totality of impacts treatment may exert, including adverse consequences. These are considered in a series of studies as follows.

#### **1.4.1** Metabolic Consequences of Androgen Deprivation

Androgen deprivation therapy (ADT) can be accomplished with medical or surgical castration. This hypogonadism produces several well-described treatment-related adverse effects including insulin resistance, elevated lipoproteins, and weight gain.(Smith, Finkelstein et al. 2002; Smith, Lee et al. 2006; Saylor and Smith 2009) Consistent with these adverse effects, GnRH agonist treatment has been associated with increased risk for diabetes and cardiovascular disease.(Keating, O'Malley et al. 2006; Saigal, Gore et al. 2007; Allibhai 2008; Keating, O'Malley et al. 2010; Saylor, Keating et al. 2011) The metabolic impact of the more profound hypogonadism produced by an androgen biosynthesis inhibitor in combination with GnRH agonist therapy has not yet been evaluated.

Castrate testosterone is defined as serum testosterone < 50 ng/dL. TAK-700 is an androgen biosynthesis inhibitor that further reduces serum testosterone in men with castrate testosterone levels due to GnRH agonist therapy.(Dreicer, Agus et al. 2010) Testosterone measurement using widely-available radioimmunoassays and chemiluminescent testing is notably imprecise when measuring testosterone levels at the low end of the spectrum.(Fitzgerald and Herold 1996; Taieb, Mathian et al. 2003; Wang, Catlin et al. 2004) We therefore plan to measure ontreatment testosterone using liquid chromatography tandem mass spectrometry (LC/MS/MS), a technique that maintains precision when testosterone levels are below 50 ng/dL.(Taieb, Mathian et al. 2003; Wang, Catlin et al. 2004) It is expected that nadir testosterone will be lower among men who receive TAK-700 in addition to a GnRH agonist. Serum testosterone levels drawn at intervals throughout the 24 months of ADT will be analyzed to investigate whether there is lower cumulative androgen exposure during those 24 months, a putative mechanism of the proposed therapy.

The metabolic impact of this lower androgen exposure will be evaluated in several ways. Glycemic parameters, lipid profiles, and body mass index (BMI) will be serially evaluated during systemic treatment and during follow-up. Insulin resistance is an independent risk factor for cardiovascular disease and is present in about one fourth of adults in the general population.(Despres, Lamarche et al. 1996; Pyorala, Miettinen et al. 1998) Existing data demonstrate that standard ADT with a GnRH agonist decreases insulin sensitivity(Smith, Lee et al. 2006) and is associated with an increased incidence of type 2 diabetes.(Allibhai 2008; Keating, O'Malley et al. 2010) We will investigate whether long-term treatment with TAK-700 increases the incidence of insulin resistance, prediabetes, or diabetes. Standard ADT with a GnRH agonist causes increases in total cholesterol, triglycerides, and high density lipoprotein (HDL).(Eri, Urdal et al. 1995; Dockery, Bulpitt et al. 2003; Smith, Lee et al. 2008) We will investigate whether long-term treatment with TAK-700 results in higher lipid levels. Finally, prospective studies have demonstrated that one year of GnRH agonist therapy increases total body weight by approximately 2%.(Smith, Finkelstein et al. 2002; Smith 2004) We will

investigate whether long-term treatment with TAK-700 results in higher body mass index when compared to GnRH agonist monotherapy.

#### 1.4.2 Androgen Recovery after Treatment

Withdrawal of GnRH agonist therapy usually leads to recovery of androgen production to noncastrate levels, though the timing of this recovery is quite variable. Among studies that have described the recovery of androgen production after ADT, median time to normalization of serum testosterone varied greatly. (Hall, Fritzsch et al. 1999; Nejat, Rashid et al. 2000; Pickles, Agranovich et al. 2002; Gulley, Figg et al. 2005; Kaku, Saika et al. 2006; Gulley, Aragon-Ching et al. 2008) One study reported normalization within a median of 15.4 weeks in men who had received six months of ADT(Gulley, Aragon-Ching et al. 2008) while another reported a median of 24 months to testosterone normalization in men who had received a median of 30 months of ADT.(Kaku, Saika et al. 2006) Androgen recovery after blockade of both gonadal and adrenal androgen synthesis using a GnRH agonist with TAK-700 has not yet been described. In this phase III trial, the timing of androgen recovery after cessation of ADT will be important to the interpretation of the primary results. If the experimental arm is found to have superior overall survival when compared to the control arm, it will be essential to also know the kinetics of androgen recovery. We hypothesize that recovery of testosterone to above the accepted threshold for supplementation in the general population will be similar in the two treatment arms. We will measure serum testosterone during the first 5 years of follow-up after cessation of systemic therapy.

#### 1.4.3 Evaluation of Clinical and Chronic Disease Outcomes

Clinical outcomes that have been shown to be associated with GnRH agonist therapy include new diagnosis of diabetes, osteoporotic fracture, coronary artery disease, myocardial infarction, stroke, pulmonary embolism, and deep vein thrombosis. Post-hoc analyses of clinical outcomes among men who participated in RTOG clinical trials (trials 85-31(Efstathiou, Bae et al. 2008), 86-10(Roach, Bae et al. 2008), and 92-02(Efstathiou, Bae et al. 2008)) have been important in clarifying these risks as they found no association between GnRH agonist treatment and cardiovascular mortality. Unfortunately, those trials were not designed to assess non-fatal cardiovascular events or other clinical endpoints relevant to prostate cancer survivorship. The proposed study presents an important opportunity to formally collect data on these clinical outcomes in a large prospective trial.

It is not known whether more intensive androgen deprivation with a GnRH agonist and an androgen biosynthesis inhibitor is associated with additional risk for these outcomes. The proposed study provides an ideal setting in which to examine this possibility as it is a randomized controlled trial with long term follow-up. Long term safety of such novel hormonal agents cannot optimally be evaluated in clinical trials in patients with more advanced disease because such patients suffer from more substantial cancer disease burden and more commonly move on promptly to subsequent therapies.

Abiraterone acetate is another androgen biosynthesis inhibitor that recently has been shown to improve survival in men with metastatic CRPC after failure of first line chemotherapy. (de Bono, Logothetis et al. 2011) With the current and planned development of TAK-700 and other agents in this class, it is likely that increasing numbers of men will be exposed to such enhanced hypogonadism, and for increasing durations. The risks for adverse clinical outcomes as a consequence of systemic therapy among prostate cancer survivors is a particularly important issue among men treated with curative intent. This study will rigorously measure the incidence of important adverse clinical outcomes and chronic diseases among men treated with standard ADT with those treated with the combination of a GnRH agonist with TAK-700.

#### 1.5 Fatigue (12Jun2018)

A second key facet of risk-benefit evaluation for prostate cancer evaluation is patient reported outcomes relating to well-being, with fatigue being principal among these in prostate cancer. A comprehensive evaluation of fatigue is thus an integral component of this clinical trial.

Fatigue has been described as the most frequent and distressing symptom related to cancer and its treatment (Bower 2005). Radiotherapy-induced fatigue is a common early side effect reported by 80% of

patients during treatment (Jereczek-Fossa 2001). There is evidence that cancer-related fatigue (CRF) has profound effects on ability to function in usual roles and activities and can linger for months or years after treatment completion (Lilleby 1999; Monga 1999; Monga 2005; Truong 2006). Following RT and/or ADT, approximately one third of prostate cancer survivors report clinically relevant fatigue one year post treatment (Storey et al. 2011, Kyrdalen et al., 2010). The high prevalence of this symptom in persons treated for prostate cancer, as well as its association with poor quality of life, mark it as a significant problem that requires further scientific study.

The etiology of fatigue, its correlates, and prevalence in the context of prostate cancer treatment are poorly understood. RT field size (whole pelvis vs. prostate only RT), ADT, and TAK-700 have been associated with the development of fatigue. (Danjoux 2007, Beard et al. 1997, Fransson 2010, Saad et al. 2011, Agust et al. 2011). During prostate RT, fatigue has been found to increase significantly with the most severe fatigue being reported the last week of RT. (Jereczek-Fossa 2001; Truong 2006; Beard 1997; Danjoux 2007; Prue 2006, Fransson 2010). However, a significant increase in fatigue between baseline and all follow-up time points, including end of RT, 3 months, 1 year, 3 years, and 5 years following RT has been noted in prostate cancer patients (Fransson et al. 2010). For example, five years after RT, 66% of living patients had fatigue, while only 41% reported fatigue at baseline (Fransson et al. 2010). Patients who continued to undergo ADT for bone metastasis had the highest levels of fatigue. Other studies of prostate cancer patients support the notion that ADT has been independently associated with higher fatigue levels. When measured at baseline and 3 months post neoadjuvant ADT alone, fatique increased in as many as two thirds of patients all before the first day of RT. (Stephens 2007; Stone 2000). In men receiving both ADT and RT, fatigue appears to be considerably worse than in men receiving RT alone. (Voermen et al. 2006) Kyrdalen et al (2010) found that 40% of >1 year prostate cancer survivors on ADT reported chronic fatigue, while only 20% of men who discontinued ADT reported fatigue at the same time point. Men who discontinued ADT had a fatigue rate comparable to men treated with RT alone and to age-matched controls from the general population. Like ADT, TAK-700 is associated with higher fatigue levels. In Phase I and II clinical trials in men with metastatic prostate cancer treated with TAK-700 [Saad et al. 2011, Agust et al. 2011] (both are abstracts), the most common adverse effect was fatigue (16 of 26 patients) but only one patient developed grade 3 or higher fatigue. The effect of TAK-700 on fatigue levels in non-metastatic prostate cancer patients treated with ADT and RT is expected to be moderate, although there is no data at this time, only the clinical experience of the investigators.

In order to minimize the potential impact of various confounding factors on fatigue, a secondary endpoint of this study, the following key information regarding potential confounds will also be collected at the time of the PROMIS-fatigue short form (using limited questions to minimize patient burden): The Anxiety/Depression Item in the EQ-5D; Overall Sleep Quality: Item from Pittsburgh Sleep Quality Index (Buysse 1989); 1 item (Q3) of the Pittsburgh Sleep Quality Index (PSQI), a self-rated questionnaire which measures sleep quality and disturbances over a 1-week or 1-month time period; and Participants' level of physical activity will be assessed using 3-items from the Godin Leisure-Time Exercise Questionnaire (GLTEQ) [Godin 1986; Gionet 1989]. Please see Section 11.0 for further details.

#### 1.5.1 Correlation of Circulating Proinflammatory Cytokines to Fatigue

The etiology of fatigue, its correlates, and prevalence in the context of prostate cancer treatment are poorly understood. There is growing evidence that pro-inflammatory cytokines play a role in cancer-related fatigue (CRF) and fatigue from other chronic illnesses (Schubert 2007). Most of the research has been generated in breast cancer patients, and the most commonly implicated cytokines are IL-1, IL-6, TNF alpha, sTNFR2, and IFN alpha (Ryan 2007). These cytokines will be measured in the proposed study of prostate cancer patients in addition to NF-Kappa B DNA binding which has been found by our group to be elevated in fatigued women undergoing breast RT (Torres 2011). Additionally, SNPs in the promoters of cytokine genes, IL6, IL1, and TNF alpha have been associated with fatigue in breast cancer survivors (Collado-Hidalgo 2008) and prostate cancer patients (Aouizerat 2009, Miaskowski 2010). These SNPs found in genes integral to the inflammatory response will be assessed in the proposed study, as they may identify patients at risk for fatigue development. RT and ADT may initiate a constellation of molecular events that include activation of the inflammatory signaling molecule, nuclear factor kappa B (NF-kB) as well as the local and peripheral release of inflammatory cytokines (Anscher 2005). Work by Raison et al. (2009) and others have demonstrated that peripherally elaborated inflammatory cytokines can enter the brain and

activate a central inflammatory response that is associated with fatigue.(Capuron 2007) Studies have shown that the development of fatigue during radiation therapy for prostate cancer is significantly correlated with increases in peripheral inflammatory markers including interleukin (IL)-1 receptor antagonist (IL-1ra), IL-6 and c-reactive protein (CRP).(Bower 2009) In contrast, the effect of hormonal therapy on inflammatory markers is less well known. Small studies have shown altered cytokine expression by prostate tumors after hormonal therapy (Sugihara 1998), but levels of systemic cytokines after hormonal therapy for prostate cancer are not well described. Fatigue, however, is a well-known complication of hormonal therapy for prostate cancer and has been independently associated with increased inflammation (Peters 2008). Activation of the inflammatory response may be a fundamental consequence of ADT and RT leading to fatigue. Indeed, the combination of these two treatments may result in a more persistent and prolonged fatigue compared to the series evaluating fatigue after radiation alone, with as many as 32% of patients experiencing fatigue at the completion of radiation and a substantial number experiencing fatigue as late as 6.5 weeks after completion of radiation (Stone 2000). Given its primary importance in regulating the inflammatory response, NF-kB may play a prominent role in the link between cancer treatment and subsequent fatique. (Bower In press, Torres preliminary data 2011)

It will be strongly recommended that patients consent to having a blood sample sent for storage to the RTOG Biospecimen Resource. Blood will be collected from patients enrolled on this protocol at baseline, 1 year, and 2.5 years after therapy begins to follow trends in inflammatory biomarkers that may correlate with fatigue levels. The specimens will be collected and processed according to the RTOG specimen processing guidelines and must be clearly labeled with the patient identification number. Specimens from participating institutions will be banked in the RTOG Biospecimen Resource for future translational analyses. The buffy coat will be isolated from each sample and the DNA extracted. Anticipated analyses for collected specimens include circulating markers that may correlate to patient reported outcomes. An example of one anticipated analysis is the evaluation of plasma cytokines for correlation to fatigue as measured by the PROMIS instrument in patients enrolled on this trial. Examples of inflammatory markers that will be tested include CRP, NF- kappa B, TNF alpha, IL-1, IL-1ra, sTNFR2, and IL-6.

#### 1.5.2 Genetic Predictors of Fatigue

Evidence that specific genetic variants are associated with the development of such adverse effects arises from several studies. In one case/control study, 141 prostate cancer patients treated with radiotherapy were screened for SNPs in TGFB1 (Burri in press). Those subjects who possessed either the T/T genotype at position -509, the C/C genotype at position 869 or the G/C genotype at position 915 were significantly associated with the development of a decline in erectile function compared with those who did not have these genotypes. In addition. patients with the -509 T/T genotype had a significantly increased risk of developing late rectal bleeding compared with those who had either the C/T or C/C genotype at this position. These subjects were also genotyped for SNPs in SOD2, XRCC1, and XRCC3 (Damaraju 2006). Patients possessing the XRCC1 rs25489 G/A genotype were more likely to develop erectile dysfunction following irradiation compared to patients who had the G/G genotype. The estimated CAG haplotype frequency for XRCC1 was significantly higher in men with late rectal bleeding than in men without late rectal bleeding. In addition, patients who possessed the SOD2 rs4880 C/T genotype exhibited a significant increase in grade 2 late rectal bleeding compared to patients who had either the C/C or T/T genotype for this SNP. Furthermore, patients possessing the combination of the SOD2 rs4880 C/T genotype and XRCC3 rs861539 C/T genotype experienced a significant increase in grade 2 late rectal bleeding compared to patients without this particular genotypic arrangement. Another important study reported that possession of SNPs in the LIG4, ERCC2, and CYP2D6 was significantly associated with the development of clinical toxicity, including urinary morbidity, in patients treated with radiotherapy for prostate cancer (Dudbridge 2006). Taken together, the results of these studies provide a strong basis for the role of genetic factors in the ability to predict which prostate cancer patients will exhibit adverse radiotherapy responses. Thus, the hypothesis that forms the basis for this study is that SNPs and/or CNVs in certain genes are associated with the development of fatigue after radiotherapy for prostate cancer. This effect may be further exacerbated by profound androgen deprivation via agents such as TAK-700.

It will be strongly recommended that patients consent to having a blood sample sent for storage to the RTOG Biospecimen Resource. The buffy coat will be isolated from each sample and the DNA extracted. The specimens will be collected and processed according to the RTOG specimen processing guidelines. Anticipated analyses include evaluation of single nucleotide polymorphisms (SNPs) and copy number variants (CNVs) through screening DNA samples derived from case and matched control subjects using Affymetrix 6.0 microarrays. Genes to be investigated for SNPs and CNVs include TNFAIP1, IL6, IL6R, CRP, IL1R1, IL1A, IL1B. Case subjects will be patients that represent the 20% of patients in this study exhibiting the highest levels of fatigue as defined and measured by the PROMIS instrument used in this study while controls will be the 20% of patients who reported the lowest levels of fatigue as quantified using PROMIS. The goal of this study will be to identify SNPs and CNVs associated with the development of fatigue in prostate cancer patients following radiotherapy.

#### 2.0 OBJECTIVES

#### 2.1 Primary Objective

To evaluate the difference in overall survival in men with clinically localized prostate cancer with unfavorable prognostic features between a) standard treatment (ADT + radiotherapy) and b) standard treatment with the addition of 24 months of TAK-700.

#### 2.2 Secondary Objectives (12Jun2018)

2.2.1 To characterize differences between the treatment groups with respect to incidence of unexpected grade ≥ 3 adverse events and/or clinically significant decrement in patient reported quality of life among subjects treated with TAK-700.

Additional secondary objectives are to compare the treatment groups with respect to:

- **2.2.2** Rates and cumulative incidence of biochemical control (freedom from PSA failure), local/regional progression, and distant metastases
- **2.2.3** Rate and cumulative incidence of clinical failure, defined as: PSA > 25 ng/ml, documented local disease progression, regional or distant metastasis, or initiation of androgen deprivation therapy
- **2.2.4** Prostate-cancer specific survival and other-cause mortality
- 2.2.5 Change in severity of fatigue as measured by the Patient-Reported Outcome Measurement Information System (PROMIS) fatigue short form
- 2.2.6 Changes in patient reported quality of life as measured by Expanded Prostate Cancer Index Composite (EPIC)
- 2.2.7 Assess quality adjusted survival using the EQ-5D (Will not be completed and is not part of the revised quality of life substudy per Amendment 3.)
- 2.2.8 Nadir and average serum testosterone at 12 and 24 months during treatment
- **2.2.9** Changes in hemoglobin A1C, fasting glucose, and fasting insulin during 24 months of systemic treatment and during the first three years of follow-up
- 2.2.10 Changes in fasting lipid levels during 24 months of treatment and during the first three years of follow-up
- 2.2.11 Changes in body mass index (BMI) during 24 months of treatment and during the first three years of follow-up
- **2.2.12** Incidence of adverse events ascertained via CTCAE version 4.
- 2.2.13 Rate of recovery of testosterone to >230 ng/dL (accepted threshold for supplementation) after 12 and 24 months of follow-up
- 2.2.14 Median time to recovery of testosterone to >230 ng/dL during the first five years of follow-up
- **2.2.15** Cumulative incidence of relevant clinical survivorship endpoints including new diagnosis of type 2 diabetes, coronary artery disease, myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis, or osteoporotic fracture

#### 3.0 PATIENT SELECTION

#### NOTE: PER NCI GUIDELINES, EXCEPTIONS TO ELIGIBILITY ARE NOT PERMITTED

#### 3.1 Conditions for Patient Eligibility (4/16/14)

For questions concerning eligibility, please contact the study data manager.

**3.1.1** Histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days prior to registration at high risk for recurrence as determined by one of the following combinations:

| Gleason score | | PSA | | T-Stage |
|---------------|-----|--------------------|-----|----------------|
| <u>&gt;</u> 9 | and | <u>&lt;</u> 150 | and | Any |
| 8 | and | < 20 | and | <u>&gt;</u> T2 |
| 8 | and | <u>&gt;</u> 20-150 | and | Any |
| 7 | and | <u>≥</u> 20 – 150 | and | Any |

- **3.1.2** History/physical examination within 60 days prior to registration.
- **3.1.3** Clinically negative lymph nodes as established by imaging (abdominal <u>and/or</u> pelvic CT or abdominal <u>and/or</u> pelvic MRI), nodal sampling, or dissection within 90 days prior to registration.
  - Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are < 2.0 cm.</li>
- **3.1.4** No distant metastases (M0) on bone scan within 90 days prior to registration (18F-Na bone scan is an acceptable substitute).
  - Equivocal bone scan findings are allowed if plain films are negative for metastasis.
- **3.1.5** Baseline serum PSA value performed with an FDA-approved assay (e.g., Abbott, Hybritech), obtained prior to any LHRH or anti-androgen therapy, within 180 days of randomization.
- 3.1.6 Androgen deprivation therapy (ADT), such as LHRH agonists (e.g., goserelin, leuprolide), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g., DES), or surgical castration (orchiectomy), may have been started prior to registration, provided that registration is within 50 days of beginning ADT. Please note: If the patient has started ADT he will not be eligible to participate in the quality of life component of this study.
- **3.1.7** Prior testosterone administration is allowed if last administered at least 90 days prior to registration.
- **3.1.8** Zubrod Performance Status 0-1 within 21 days prior to registration
- **3.1.9** Age ≥ 18
- **3.1.10** CBC/differential obtained within 14 days prior to registration on study, with adequate bone marrow function defined as follows:
  - Absolute neutrophil count (ANC) ≥ 1,800 cells/mm<sup>3</sup>
  - Platelets ≥ 100.000 cells/mm<sup>3</sup>
  - Hemoglobin ≥ 8.0 g/dl (<u>Note</u>: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
- **3.1.11** Serum creatinine < 2.0 mg/dl and creatinine clearance (can be calculated) > 40 mL/minute within 21 days prior to registration
- **3.1.12** Bilirubin < 1.5x ULN and ALT or AST < 2.5x ULN within 21 days prior to registration
- **3.1.13** Serum testosterone within 21 days prior to registration
- **3.1.14** Chemistry (including sodium, potassium, chloride, bicarbonate (carbon dioxide), BUN, glucose, calcium, magnesium and phosphorous) and liver panels (including albumin and alkaline phosphatase) obtained within 21 days prior to registration
- **3.1.15** Fasting glucose, fasting insulin, lipid panel (cholesterol, triglyceride, HDL, LDL), and Hemoglobin A1C within 21 days prior to registration
- **3.1.16** Screening calculated ejection fraction of ≥ to institutional lower limit of normal by multiple gated acquisition (MUGA) scan or by echocardiogram ECHO.
- **3.1.17** Baseline ECG within 180 days prior to registration
- **3.1.18** Patients, even if surgically sterilized (ie, status post vasectomy), who:
  - (a) Agree to practice effective barrier contraception during the entire study treatment period and for 4 months (120 days) after the last dose of study drug, or
  - (b) Agree to completely abstain from intercourse.
- 3.1.19 Patient must be able to provide study-specific informed consent prior to study entry.
- 3.2 Conditions for Patient Ineligibility (12/17/13)
- **3.2.1** PSA > 150
- **3.2.2** Definite evidence of metastatic disease.
- **3.2.3** Pathologically positive lymph nodes or nodes > 2.0 cm on imaging.
- **3.2.4** Prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy for any reason.
- **3.2.5** Prior invasive malignancy (except non-melanoma skin cancer) unless disease-free or not requiring systemic therapy for a minimum of 3 years.

- **3.2.6** Prior systemic chemotherapy for prostate cancer (Note that prior chemotherapy for a different cancer is allowed, per Section 3.2.5).
- **3.2.7** Prior radiotherapy, including brachytherapy, to the region of the prostate that would result in overlap of radiation therapy fields.
  - Any patient undergoing brachytherapy must have transrectal ultrasound confirmation of prostate volume <60 cc, AUA score ≤15 within 60 days of registration, and no history of prior transurethral resection of the prostate (TURP); prior TURP is permitted for patients who receive EBRT only).
- **3.2.8** Previous hormonal therapy for > 50 days (see Section 3.1.6).
- **3.2.9** Known hypersensitivity to TAK-700 or related compounds
- **3.2.10** A history of adrenal insufficiency
- **3.2.11** History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 [NCI CTCAE, version 4.02] (U.S. Department of Health and Human Services, National Institutes of Health National Cancer Institute, 2009), thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (eg, pericardial effusion restrictive cardiomyopathy) within 6 months prior to registration. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
- 3.2.12 New York Heart Association Class III or IV heart failure (see Appendix IV).
- **3.2.13** ECG abnormalities of:
  - (a) Q-wave infarction, unless identified 6 or more months prior to screening
  - (b) QTc interval > 460 msec
- **3.2.14** Patients who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
- **3.2.15** Prior allergic reaction to the drugs involved in this protocol.
- **3.2.16** Study entry PSA obtained during the following time frames:
  - (a) 10-day period following prostate biopsy;
  - (b) following initiation of hormonal therapy.
- 3.2.17 Cushing's syndrome
- **3.2.18** Severe chronic renal disease (serum creatinine > 2.0 mg/dl and confirmed by creatinine clearance < 40 mL/minute)
- **3.2.19** Chronic liver disease (bilirubin > 1.5x ULN, ALT or AST > 2.5x ULN)
- **3.2.20** Chronic treatment with glucocorticoids within one year
- **3.2.21** Uncontrolled hypertension despite appropriate medical therapy within 21 days prior to registration (blood pressure of greater than 150 mm Hg systolic and 90 mm Hg diastolic at 2 separate measurements no more than 60 minutes apart during Screening visit)
- **3.2.22** Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel.
- **3.2.23** Major surgery within 14 days prior to registration
- **3.2.24** Serious infection within 14 days prior to registration
- **3.2.25** Uncontrolled nausea, vomiting, or diarrhea (CTCAE grade ≥ 3) despite appropriate medical therapy at the time of registration
- **3.2.26** Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-700, including difficulty swallowing tablets

#### 4.0 PRETREATMENT EVALUATIONS/MANAGEMENT

NOTE: This section lists baseline evaluations needed before the initiation of protocol treatment that do not affect eligibility.

- 4.1 Required Evaluations/Management (12/17/13) (2/4/14)
- **4.1.1** Review of medications at time of registration [drug names and dosages, frequency, route, start dates (at least the year that the drug was started), etc.]
- 4.1.2 Completion of the Patient-Reported Outcome Measurement Information System (PROMIS)-Fatigue Short Form, Expanded Prostate Cancer Index Composite (EPIC), and EuroQol (EQ-5D) is required for the patients who have consented to participate in the optional quality of life assessment (up to a maximum of 458 patients). However, patients participating in the QOL assessment may not have started LHRH or other anti-androgen therapy prior to enrollment and completing the QOL forms.
- 4.1.3 Any patient undergoing brachytherapy must have transrectal ultrasound confirmation of prostatic volume < 60 cc and American Urologic Association (AUA) symptom index composite score ≤ 15 within 60 days of registration. If a patient is thought to be a poor brachytherapy candidate based on anatomy at the time of</p>

ultrasound, he may still participate in the study but must receive EBRT only per protocol guidelines. If a patient is deemed an inadequate brachytherapy candidate after he has already been enrolled on the protocol, he may be switched to EBRT administered per protocol guidelines, but this will result in a protocol deviation.

#### **4.1.4** Height and weight

#### **5.0 REGISTRATION PROCEDURES** (12JUN2018)

Food and Drug Administration (FDA) regulations and National Cancer Institute (NCI) policy require all individuals contributing to NCI-sponsored trials to register and to renew their registration annually. To register, all individuals must obtain a Cancer Therapy Evaluation Program (CTEP) Identity and Access Management (IAM) account (<a href="https://ctepcore.nci.nih.gov/iam">https://ctepcore.nci.nih.gov/iam</a>). In addition, persons with a registration type of Investigator (IVR), Non-Physician Investigator (NPIVR), or Associate Plus (AP) (i.e., clinical site staff requiring write access to OPEN, RAVE, or TRIAD or acting as a primary site contact) must complete their annual registration using CTEP's web-based Registration and Credential Repository (RCR) (https://ctepcore.nci.nih.gov/rcr). Documentation requirements per registration type are outlined in the table below.

| Documentation Required | IVR | NPIVR | АР | А |
|---|---|---|---|---|
| FDA Form 1572 | V | V | | |
| Financial Disclosure Form | • | V | • | |
| NCI Biosketch (education, training, employment, license, and certification) | • | • | V | |
| HSP/GCP training | V | V | • | |
| Agent Shipment Form (if applicable) | • | | | |
| CV (optional) | • | • | • | |

An active CTEP-IAM user account and appropriate RCR registration is required to access all CTEP and CTSU (Cancer Trials Support Unit) websites and applications. In addition, IVRs and NPIVRs must list all clinical practice sites and IRBs covering their practice sites on the FDA Form 1572 in RCR to allow the following:

- Added to a site roster
- Assigned the treating, credit, consenting, or drug shipment (IVR only) tasks in OPEN
- Act as the site-protocol PI on the IRB approval

Additional information can be found on the CTEP website at < <a href="https://ctep.cancer.gov/investigatorResources/default.htm">https://ctep.cancer.gov/investigatorResources/default.htm</a> >. For questions, please contact the RCR Help Desk by email at < RCRHelpDesk@nih.gov >.

TRIAD, the American College of Radiology's (ACR) image exchange application, will be used for dosimetry digital treatment data submission on this trial. See below for information on installing TRIAD for submission of digital RT data prior to enrolling patients.

#### 5.1 Pre-Registration Requirements for IMRT Treatment Approach (4/16/14)

5.1.1 In order to utilize IMRT on this study, the institution must have met specific technology requirements and have provided baseline physics information. Instructions for completing these requirements or determining if they already have been met are available on the Imaging and Radiation Oncology Core (IROC) Houston QA Center [formerly the Radiological Physics Center (RPC)] web site. Visit <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a> and select "Credentialing" and "Credentialing Status Inquiry". The institution or investigator must update or complete a new IMRT Facility Questionnaire (available on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>) and send it to NRG Oncology for review prior to entering any cases.

An IMRT phantom study with IROC Houston must be successfully completed (if the institution has not previously met this IMRT credentialing requirement). Instructions for requesting and irradiating the phantom are available on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>; select "Credentialing" and "NRG". Upon review and successful completion of the phantom irradiation, IROC Houston will notify both the registering institution and NRG Oncology that the institution has completed this requirement. Subsequently, NRG Oncology will notify the institution that the IMRT credentialing requirement has been met.

#### **5.2** Pre-Registration Requirements for 3DCRT Treatment Approach (4/16/14)

- **5.2.1** Only institutions that have met the technology requirements and that have provided the baseline physics information that are described in 3D-CRT Quality Assurance Guidelines may enter patients onto this study.
- 5.2.2 A new or updated Facility Questionnaire (one per institution, available on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>) is to be sent to NRG Oncology for review prior to entering any cases. NRG Oncology will notify the institution when all requirements have been met and the institution is RT credentialed to enter patients onto this study. Institutions that have previously enrolled patients on 3D-CRT trials of this same disease site may enroll patients on this study without further credentialing.

#### 5.3 Pre-Registration Requirements for Brachytherapy Treatment Approach (4/16/14)

#### 5.3.1 Brachytherapy

Institutions must be credentialed by IROC Houston prior to registering any cases to this study. The credentialing materials may be found on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a> under the "credentialing" tab. Upon review and successful completion, IROC Houston will notify both the registering institution and NRG Oncology that the institution has successfully completed this requirement. NRG Oncology will notify the institution when all requirements have been met and the institution is RT credentialed to enter subsequent patients onto this study.

#### **5.3.2** Brachytherapy Credentialing

Radiation Oncologists and Physicists are credentialed as a team for LDR brachytherapy (seed dependent), CT planned HDR brachytherapy, and TRUS planned HDR brachytherapy. The following can be found on the IROC Houston web site at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a> and must be completed for each technique and/or seed:

- Knowledge Assessment Questionnaire to be submitted to IROC Houston.
- Facility Questionnaire to be submitted to IROC Houston.
- 2 Benchmark Cases to be submitted to IROC Houston.
- A recent clinical case treated per protocol and a completed Implant Dosimetry Data Form to be submitted to IROC Houston and electronically sent to NRG Oncology (see <u>Section 12.2</u>)

If an institution has been credentialed for a previous NRG Oncology/RTOG LDR prostate brachytherapy trial (RTOG 0526, RTOG 0815), RTOG HDR prostate brachytherapy trial for CT planned HDR, and/or RTOG HDR prostate brachytherapy trial for TRUS planned HDR, and the radiation oncologist and physicist team are the same as on the approved credentialing request, and the institution is using the same seed model and planning system as on the approved credentialing request, then they do not have to be re-credentialed for that modality for this trial with the exception of completing the Knowledge Assessment Form specific to this protocol.

- A change of physician will require submission of the Knowledge Assessment Form and Clinical Test Case.
- A change in physicist will require submission of the Knowledge Assessment Form and the Benchmark Cases.
- A change in either the treatment planning computer or brachytherapy source model will require resubmission of only the Benchmark Cases.

Brachytherapy sources to be used on this protocol must be listed on the joint RPC/AAPM source registry at <a href="http://irochouston.mdanderson.org">http://irochouston.mdanderson.org</a>; select "brachy sources".

#### 5.4 Digital RT Data Submission to NRG Oncology Using TRIAD

TRIAD is the American College of Radiology's (ACR) image exchange application. TRIAD provides sites participating in NRG Oncology clinical trials a secure method to transmit DICOM RT and other objects. TRIAD anonymizes and validates the images as they are transferred.

#### **TRIAD Access Requirements:**

- Site physics staff who will submit images through TRIAD will need to be registered with The Cancer Therapy Evaluation Program (CTEP) and have a valid and active CTEP Identity and Access Management (IAM) account. Please refer to <u>Section 5.0</u> above for instructions on how to request a CTEP-IAM account.
- To submit images, the site physics user must have been assigned the 'TRIAD site user' role on the relevant Group or CTSU roster.
- RAs are able to submit standard of care imaging through the same method.

#### **TRIAD Installations:**

When a user applies for a CTEP-IAM account with proper user role, he/she will need to have the TRIAD application installed on his/her workstation to be able to submit images. TRIAD installation documentation can be found on the NRG Oncology/RTOG website Core Lab tab.

This process can be done in parallel to obtaining your CTEP-IAM account username and password.

If you have any questions regarding this information, please send an e-mail to the TRIAD Support mailbox at TRIAD-Support@acr.org.

#### **5.5 Regulatory Pre-Registration Requirements** (12Jun2018)

**5.5.1** This study is supported by the NCI Cancer Trials Support Unit (CTSU).

Each investigator or group of investigators at a clinical site must obtain IRB approval for this protocol and submit IRB approval and supporting documentation to the CTSU Regulatory Office before they can enroll patients.

Assignment of site registration status in the CTSU Regulatory Support System (RSS) uses extensive data to make a determination of whether a site has fulfilled all regulatory criteria including but not limited to the following:

- An active Federal Wide Assurance (FWA) number
- An active roster affiliation with the Lead Network or a participating organization
- A valid IRB approval
- Compliance with all protocol specific requirements.

In addition, the site-protocol Principal Investigator (PI) must meet the following criteria:

- Active registration status
- The IRB number of the site IRB of record listed on their Form FDA 1572
- An active status on a participating roster at the registering site.

Sites participating on the NCI CIRB initiative that are approved by the CIRB for this study are not required to submit IRB approval documentation to the CTSU Regulatory Office. For sites using the CIRB, IRB approval information is received from the CIRB and applied to the RSS in an automated process. Signatory Institutions must submit a Study Specific Worksheet for Local Context (SSW) to the CIRB via IRB Manager to indicate their intent to open the study locally. The CIRB's approval of the SSW is then communicated to the CTSU Regulatory Office. In order for the SSW approval to be processed, the Signatory Institution must inform the CTSU which CIRB-approved institutions aligned with the Signatory Institution are participating in the study.

#### **Downloading Site Registration Documents:**

Site registration forms may be downloaded from the RTOG 1115 protocol page located on the CTSU members' web site. Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the members' area using your CTEP-IAM username and password

- Click on the Protocols tab in the upper left of your screen
- Either enter the protocol # in the search field at the top of the protocol tree, or
- Click on the By Lead Organization folder to expand
- Click on the NRG Oncology link to expand, then select trial protocol #RTOG-1115.
- Click on LPO Documents, select the Site Registration Documents link and download and complete the forms provided

#### Requirements for RTOG 1115 site registration:

- IRB approval (For sites not participating via the NCI CIRB; local IRB documentation, an IRB-signed CTSU IRB Certification Form, Protocol of Human Subjects Assurance Identification/IRB Certification/Declaration of Exemption Form, or combination is accepted)
- CTSU RT Facilities Inventory Form (if applicable)
- IRB/REB approved consent (English and native language versions\*)
   \*Note: Institutions must provide certification/verification of IRB/REB consent translation to NRG Oncology (described below).

#### Non-English Speaking Canadian and Non-North American Institutions

Translation of documents is critical. The institution is responsible for all translation costs. All regulatory documents, including the IRB/REB approved consent, must be provided in English and in the native language. Certification of the translation is optimal but due to the prohibitive costs involved NRG Oncology will accept, at a minimum, a verified translation. A verified translation consists of the actual REB approved consent document in English and in the native language, along with a cover letter on organizational/letterhead stationery that includes the professional title, credentials, and signature of the translator as well as signed documentation of the review and verification of the translation by a neutral third party. The professional title and credentials of the neutral third party translator must be specified as well.

### Submit completed forms along with a copy of your IRB Approval and Informed Consent to the CTSU Regulatory Office, where they will be entered and tracked in the CTSU RSS:

Regulatory Submission Portal: www.ctsu.org (members' area) → Regulatory Tab → Regulatory Submission

When applicable, original documents should be mailed to: CTSU Regulatory Office 1818 Market Street, Suite 3000 Philadelphia, PA 19103

Check the status of your site's registration packets by querying the RSS site registration status page of the members' section of the CTSU web site. (Note: Sites will not receive formal notification of regulatory approval from the CTSU Regulatory Office.)

Go to <a href="https://www.ctsu.org">https://www.ctsu.org</a> and log in to the members' area using your CTEP-IAM username and password;

- Click on the Regulatory tab at the top of your screen;
- Click on the Site Registration tab;
- Enter your 5-character CTEP Institution Code and click on Go.

#### **5.5.2** Pre-Registration Requirements FOR CANADIAN INSTITUTIONS

In addition to the requirements above, Canadian institutions also must complete and submit to the Regulatory Submission Portal: www.ctsu.org (members' area) → Regulatory Tab → Regulatory Submission

- Health Canada's Therapeutic Products Directorates' Clinical Trial Site Information Form,
- Qualified Investigator Undertaking Form, and
- · Research Ethics Board Attestation Form.

#### **5.5.3** Pre-Registration Requirements for the Initial Shipment of TAK-700:

#### **U.S. and Canadian Institutions**:

All pre-registration requirements must be met before registering the first case. Institutions must electronically complete (versus hand write) a Study Agent Shipment Form (SASF) available on the NRG Oncology/RTOG web site, <a href="www.rtog.org">www.rtog.org</a>, under protocol-specific materials/regulatory resources. U.S. and Canadian institutions must fax the SASF to the CTSU Regulatory Office (Fax 215-569-0206) as soon as the individual responsible for the study agent has been identified. The completed SASF document also may be e-mailed to the CTSU at <a href="mailto:CTSURegulatory@ctsu.coccg.org">CTSURegulatory@ctsu.coccg.org</a>.

#### **5.6 OPEN Registration** (12/17/13)

#### **5.6.1** OPEN Registration Instructions

Patient registration can occur only after evaluation for eligibility is complete, eligibility criteria have been met, and the study site is listed as 'approved' in the CTSU RSS. Patients must have signed and dated all applicable consents and authorization forms.

Patient enrollment will be facilitated using the Oncology Patient Enrollment Network (OPEN). OPEN is a web-based registration system available on a 24/7 basis. All site staff will use OPEN to enroll patients to this study. OPEN can be accessed at <a href="https://open.ctsu.org">https://open.ctsu.org</a> or from the OPEN tab on the CTSU members' web site <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

Prior to accessing OPEN site staff should verify the following:

- All eligibility criteria have been met within the protocol stated timeframes. Site staff should
  use the registration forms provided on the group or CTSU web site as a tool to verify
  eligibility.
- All patients have signed an appropriate consent form and HIPPA authorization form (if applicable).

#### Access requirements for OPEN:

- See Section 5.0 for obtaining a CTEP-IAM account.
- To perform registrations, the site user must have been assigned the 'Registrar' role on the relevant Group or CTSU roster.
- To perform registrations on protocols for which you are a member of NRG Oncology, you
  must have an equivalent 'Registrar' role on the NRG Oncology roster. Role assignments
  are handled through the Groups in which you are a member.
- To perform registrations to trials accessed via the CTSU mechanism (i.e., non-Lead Group registrations) you must have the role of Registrar on the CTSU roster. Site and/or Data Administrators can manage CTSU roster roles via the new Site Roles maintenance feature under RSS on the CTSU members' web site. This will allow them to assign staff the "Registrar" role.

The OPEN system will provide the site with a printable confirmation of registration and treatment information. Please print this confirmation for your records.

Further instructional information is provided on the CTSU members' web site OPEN tab or within the OPEN URL. For any additional questions contact the CTSU Help Desk at 1-888-823-5923 or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>.

5.6.2 In the event that the OPEN system is not accessible, participating sites can contact web support for assistance with web registration: <a href="websupport@acr.org">websupport@acr.org</a> or call the Registration Desk at (215) 574-3191, Monday through Friday, 8:30 a.m. to 5:00 p.m. ET. The registrar will ask the site to fax in the eligibility checklist and will need the registering individual's e-mail address and/or return fax number. This information is required to assure that mechanisms usually triggered by the OPEN web registration system (e.g., drug shipment and confirmation of registration) will occur.

#### **6.0 RADIATION THERAPY** (12/17/13) (2/4/14)

TRIAD, the American College of Radiology's (ACR) image exchange application, will be used for dosimetry digital treatment data submission. See <a href="Section 5.0">Section 5.0</a> for information on installing TRIAD for submission of digital RT data PRIOR TO ENROLLING PATIENTS.

In both arms, radiotherapy should begin within 8-10 weeks after the date of the first LHRH agonist injection.

Note: There is no difference in radiation requirements between arms as the randomized question is in regard to hormonal therapy. However, as this protocol allows for treatment with EBRT exclusively or EBRT + a brachytherapy boost (at the discretion of the treating physician) this must be specified at the time of study enrollment. Because patients are stratified by type of boost treatment delivered (IMRT vs. brachytherapy), if a patient who was originally intended to receive brachytherapy be found, post-enrollment, to be a poor brachytherapy candidate based on transrectal ultrasound examination, he may be switched to external beam radiotherapy administered per protocol guidelines, but this will result in a protocol deviation. Therefore, it is strongly recommended to obtain ultrasound assessment of prospective brachytherapy patients before enrollment on this study.

When an IMRT (rather than brachytherapy) boost is used to meet the dose constraints, the composite EBRT plan (see Sections 6.4 - 6.5) that includes Phases 1 and 2 must be generated and summed at the beginning of the patient's treatment to verify adherence to the required dose constraints. In the case of an inability to meet normal tissue dose-constraints on the summed plan a decrease in PTV dose to achieve normal tissue sparing is recommended (see Section 6.5).

#### **6.1** Two Stage Radiation Plan (12/17/13)

**6.1.1 Phase 1**: Whole pelvis including prostate and seminal vesicles

Acceptable Treatment Modalities:

3D-CRT or IMRT

Prescription Dose (See Table 1):

45 Gy to cover 98% of PTV

- Minimum dose within PTV 95% of prescribed dose and for a volume that is 0.03 cc
- Maximum dose within the PTV 110% of prescribed dose and for a volume that is 0.03 cc

Table 1: 3D-CRT and IMRT Dose Objectives for Phase 1 – Pelvic and Prostate Radiation

| Phase 1 | Dose, | Volume, | Per | Variation |
|---|---|---|---|---|
| PTV_4500 | Gy | cc or | Protocol | Acceptable |
| | | %PTV | | included in range of |
| Coverage | $D_{Rx}^{I}(V_{\%})$ | 98% | equals 45 | 44 to 46 |
| Minimum | $D_{Min}^{I}(V_{cc})$ | 0.03cc | not less | 40.5 to |
| Dose | | | than 42.8 | 42.8 |
| Maximum | $D_{Max}^{I}(V_{cc})$ | 0.03cc | not more | 49.5 to 54 |
| Dose | | | than 49.5 | |
| Homogeneity | D <sup>I</sup> <sub>PTV_4500</sub> | V(49.5Gy) | not more | |
| | _ | | than 10% | |
| D <sub>Max</sub> in | | | In | |
| Patient | | | PTV_4500 | |

Note: Dosimetric and/or volumetric parameters falling outside the Per Protocol and Variation Acceptable specifications are classified as Deviation Unacceptable.

#### **6.1.2** Phase 2: Reduce volume to boost prostate and proximal seminal vesicles

Acceptable Treatment Modalities:

IMRT or permanent prostate implant (PPI) brachytherapy or HDR brachytherapy

Prescribed Dose for IMRT boost (See Table 2):

34.2 Gy for IMRT to cover 98% of the PTV

- Minimum dose within PTV 95% of prescribed dose and for a volume that is 0.03 cc
- Maximum dose within the PTV 107% of prescribed dose and for a volume that is 0.03 cc

Prescription Dose for brachytherapy:

110 Gy for low dose rate PPI with I-125

100 Gy for low dose rate PPI with Pd-103

15 Gy in one fraction for HDR or two fractions of 10.5 Gy

Table 2: IMRT Dose Objectives for Prostate and Proximal Seminal Vesicle Boost

| Phase 2<br>PTV_7920 | Dose,<br>Gy | Volume,<br>cc or<br>%PTV | Per<br>Protocol | Variation Acceptable included in |
|---|---|---|---|---|
| | | 701 1 0 | | range of |
| Coverage | $D^{II}_{Rx}(V_{\%})$ | 98% | equals | 33.4 |
| | | | 34.2 | to 35 |
| Minimum | $D_{Min}^{II}(V_{cc})$ | 0.03cc | not less | 30.8 |
| Dose | | | than 32.5 | to 32.5 |
| Maximum | $D_{Max}^{II}(V_{cc})$ | 0.03cc | not more | 36.6 |
| Dose | | | than 36.6 | to 37.6 |
| Homogeneity | D <sup>II</sup> <sub>PTV_7920</sub> | V(36.6Gy) | not more | |
| | _ | | than 10% | |
| D <sub>Max</sub> in | | | In | |
| Patient | | | PTV_7920 | |

Note: Dosimetric and/or volumetric parameters falling outside the Per Protocol and Variation Acceptable specifications are classified as Deviation Unacceptable.

#### 6.2 Technical Factors

- **6.2.1** Either 3DCRT or IMRT may be used for phase 1 of either Arm 1 or 2. For 3DCRT treating the whole pelvis (WPRT), a minimum of 4-fields should be used and a 4 field plan is recommended. For IMRT, no specific field arrangement is required.
- **6.2.2** RT will be delivered with megavoltage equipment at energies ≥ 6 MV. Typically, except for tomotherapy and VMAT techniques, 5 to 9 gantry angles are employed for the boost IMRT treatment.
- 6.2.3 Patients who receive brachytherapy as a boost component of their RT will undergo EBRT for Phase 1 implementing either 3DCRT or IMRT as described. The prostate and seminal vesicles will be treated to a dose of 45 Gy in 1.8 Gy fractions prescribed to a PTV dose as above.

#### 6.3 EBRT Localization, Simulation, and Immobilization (12/17/13)

Simulation will be CT-based in all cases. The use of urethral contrast at the time of simulation is not required to help identify the apex of the prostate. Rectal contrast is discouraged because it may distend the rectum and artificially displace the prostate in the anterior direction. Intravenous contrast is permitted but not required to assist in identifying the pelvic vessels. Patients will be positioned supine or prone on a flat tabletop and a customized thermoplastic immobilization cast or a molded foam cradle or similar immobilization for stabilization and setup reproducibility is suggested. The degree of bladder fullness should be made to duplicate the degree of fullness anticipated for daily treatment, i.e., if the patient is instructed to maintain a full bladder for treatment, he should be simulated as such (especially for cases in which image guidance is not implemented). The rectum should be kept as empty as possible; consider an enema 1-2 hours prior to simulation. CT images should be acquired at a slice thickness of ≤3 mm from the top of the iliac crests superiorly to the perineum inferiorly. Target volumes (Section 6.4) and normal critical structures (Section 6.4.4) will be defined in the slices in which they are visualized. The 3DCRT cases (Phase 1) must utilize "beam's eye view" representations to define final beam aperture.

**6.3.1** CT Slice Thickness, Dose Matrix Spatial Resolution, and DVH Fidelity

A CT slice thickness of 3mm with a linear dose matrix spatial resolution of 3mm, provides a dose voxel of 0.027cc, just sufficient to determine doses in  $V_{cc}$  = 0.03cc for compliance assessment via DVH analyses. Higher spatial resolution in imaging and in dose matrices improve the DVH analyses in the point-dose surrogate volume,  $V_{cc}$  = 0.03cc.

Imaging slice thickness  $\leq$  3mm Dose matrix resolution  $\leq$  3mm

For planning systems that calculate DVH by super-sampling of the dose matrix data, planners may find it useful to set the secondary DVH resolution in number of points sampling an object volume (i.e., PTV, OAR,...) to obtain a planning\_DVH\_ $V_{cc}$  smaller than 0.03cc. The lower bound on the number of sampling points is given by Object\_Volume(cc)/0.03cc. A factor of two to three increasing this number improves the fidelity of the DVH derived from the calculated dose matrix.

- **6.4** Treatment Planning/Target Volumes (4/16/14)
- 6.4.1 Patients treated with an IMRT boost (Phase 2) must have a composite treatment plan generated at the beginning of Phase 1 so that the final EBRT dose to critical structures is evaluated before any dose delivery has begun.

Dose for Phase 1 (CTV\_4500/PTV\_4500) will be 45.0 Gy at 1.8 Gy per fraction in both arms. Once Phase 1 is completed, a cone down boost to the prostate and proximal vesicles will be delivered in Phase 2 by any one of the three acceptable methods: IMRT, HDR or LDR permanent prostate implant. If an EBRT boost is planned, the prostate will receive 34.2 Gy at 1.8 Gy per fraction, for a total prostate dose of 79.2 Gy. For pelvic 3D-CRT, a 4-field technique, using opposed anterior-posterior and opposed lateral fields, is recommended. All fields should conform to the beam's-eye-view of the target. No specific field arrangement is required for IMRT, although typically 5-9 fields are used for fixed gantry treatment. Tomotherapy and VMAT also are allowed for IMRT treatment on this protocol. However, both of these techniques must be credentialed separately from general IMRT credentialing.

6.4.2 The definition of GTV, CTV and PTV will be in accordance with the ICRU Report #50: Prescribing, Recording, and Reporting Photon Beam Therapy.

#### <u>Phase 1 Pelvis, including prostate and seminal vesicles (Arms 1 and 2)</u> Gross Target Volume (GTV)

The GTV is defined by the physician as all known disease as defined by the planning CT, urethrogram, and clinical information. If a urethrogram is used, the GTV will encompass a volume inferiorly 5 mm superior to the tip of the dye and no less than the entire prostate. Prostate dimensions should be defined as visualized on CT scan.

#### Clinical Target Volume (CTV 4500)

The CTV 4500 will include the prostate and entire seminal vesicles (SeminalVesicle), the obturator. external iliac, proximal internal iliac and common iliac nodes (CTVn), using the vascular structures, up to a level corresponding to the top of L4-L5. Please refer to the pelvic nodal atlas at the RTOG Web site Node Prostate Lymph Volumes for http://www.rtog.org/CoreLab/ContouringAtlases/ProstatePelvicLymphNodes.aspx). The presacral nodes from L5-S1 to S3 may be included if desired depending on whether the dose constraints to the rectum are achievable (see Table 1). The CTV\_4500 will extend superiorly from L4-L5 to 0.5 cm below the tip of the urethral contrast dye (if used) and no less than the entire prostate gland. Lateral borders will be at least 1 cm from the pelvic brim. In the lateral fields, the external and internal iliac lymph nodes below the SI joints, and the posterior extension of the seminal vesicles should be covered. The usual posterior border is approximately S2-3, but CT anatomy should take precedence. The inferior extent of the external iliac lymph nodes is at the top of the femoral heads. The inferior extent of the obturator lymph nodes is at the top of the symphysis pubis. The CTV 4500 will include a 7 mm margin in 3-dimensions to the contoured iliac vessels, but not extend outside of the true pelvis, into the pelvic musculature nor into adjacent identifiable organs, such as the bladder, rectum or other bowel. Extension of the CTV into adjacent bone may be carved out.

#### Planning Target Volume

The PTV 4500 margins should be a minimum of 0.5 cm and a maximum of 1.5 cm in all dimensions.

#### <u>Phase 2 Prostate and Proximal Seminal Vesicles Boost with IMRT (Arms 1 and 2)</u> Gross Target Volume (GTV)

The expansion will be based on GTV in phase 1 above (see Section 6.4.2). Clinical Target Volume (CTV 7920)

The CTV\_7920 is the GTV plus areas considered to contain microscopic disease, delineated by the treating physician. The CTV 7920 includes the GTV (prostate) plus areas at risk for microscopic disease extension plus the proximal bilateral seminal vesicles. Only the proximal 1.0 cm of seminal vesicle tissue adjacent to the prostate shall be included in the clinical target volume. This 1.0 cm of seminal vesicles refers to both radial (in plane) and superior (out of plane) extent. If both prostate and seminal vesicle are visualized in the same CT slice, this seminal vesicle tissue will contribute to the 1.0 cm of tissue as seen on the CT simulation scan. For patients with clinical biopsy proven involvement of the seminal vesicles treatment of the entire seminal vesicles is acceptable as long as it does interfere with the ability to achieve dose constraints to the critical normal structures (see Section 6.5).

Planning Target Volume (PTV 7920)

The PTV 7920 will provide a margin around the CTV 7920 to compensate for the variability of treatment set up and internal organ motion. A range of 5-10 mm around the CTV is required to define each respective PTV. Individual selection of a PTV margin should be based on the institution's level of confidence in patient set-up and the availability of image guidance. Superior and inferior margins (capping) should be 5-10 mm depending on the thickness and spacing of the planning CT scan. Careful consideration should be made when defining the 5-10 mm margin in 3 dimensions.

#### Normal Critical Structures 6.4.3

Normal critical structures to be defined on the treatment planning CT scan will include the following: bladder, rectum (from its origin at the rectosigmoid flexure superiorly or the bottom of the SI joints, whichever is more inferior to the inferior-most extent of the ischial tuberosities), bilateral femora (to the level of ischial tuberosity), penile bulb, and skin. Any small bowel within the primary beam aperture should be defined as well. The normal tissues will be contoured and considered as solid organs. The bladder should be contoured from its base to the dome, and the rectum from the anus (at the level of the ischial tuberosities) for a length of 15 cm or to the rectosigmoid flexure. This generally is below the bottom of the sacroiliac joints. If IMRT is being used to treat the pelvic nodes, the potential bowel space (not just individual loops of bowel) where the small and large bowel may fall should be outlined. The borders are the abdominal wall anteriorly, pelvic sidewalls laterally (excluding the pelvic lymph node regions), superiorly to one cut above the last axial CT image on which the lymph nodes are outlined and inferiorly from the level of the top of CTV 4500 (outlining around the sides of the bladder near the top of the bladder to encompass the bowel that may fall into these regions). See the NRG Oncology/RTOG web site (http://www.rtog.org/CoreLab/ContouringAtlases/MaleRTOGNormalPelvisAtlas.aspx) to view the normal pelvis atlas for examples of target and normal tissue contours.

The following table summarizes the naming of targets and critical structures for submission of data to NRG Oncology via TRIAD.

**Note:** All required structures must be labeled as listed in the table below for digital RT data submission. Resubmission of data may be required if labeling of structures does not conform to the standard DICOM name listed.

| EBRT 1115 |
|---------------------|
| Standard DICOM Name |
| GTV |
| CTV_4500 |
| CTV_7920 |
| PTV_4500 |
| PTV_7920 |
| NonPTV |
| Femur_L |
| Femur_R |
| Bladder |
| PenileBulb |
| Rectum |
| External |
| BowelSpace |
| SeminalVesicle |
| CTVn |
| LDR |
| ETV |
| Rectum |
| Bladder |
| External |
| HDR |
| CTV |
| PTV |
| Prostate |
| SeminalVesicle |
| Urethra |
| Bladder |
| Rectum |
| External |

6.4.4 The PTV forms the entire target as described. 3D conformal beams will be shaped to include the entire PTV and minimize dose to surrounding critical structures as described. IMRT using inverse planning is permitted with constraints placed to adhere to critical structure dose limitations as defined below.

#### 6.5 Critical Structures

Critical structure dose constraints shall remain consistent with those represented in prior RTOG 3DCRT/IMRT prostate protocols (see Table 3 below).

**Table 3: Critical Structure Dose Constraints** 

| Normal organ<br>limit† | No more than 15% volume receives dose that exceeds | No more than<br>25% volume<br>receives dose<br>that exceeds | No more than<br>35% volume<br>receives dose<br>that exceeds | No more than<br>50% volume<br>receives dose<br>that exceeds |
|---|---|---|---|---|
| Bladder<br>Constraint | 80 Gy | 75 Gy | 70 Gy | 65 Gy |
| Rectum<br>Constraint | 75 Gy | 70 Gy | 65 Gy | 60 Gy |
| Penile Bulb | Mean dose less than or equal to 52.5 Gy | | | |

†Normal organ limit refers to the volume of that organ that should not exceed the dose limit.

While every effort should be made to deliver prescription doses to the PTV as specified while adhering to these constraints, it is recognized that certain anatomical factors may prevent this. As mentioned in Section 6.1, a prescription dose reduction to a level of 77.4 Gy or 75.6 Gy is permitted if constraints cannot be met at a prescription dose of 79.2 Gy. For purposes of compliance, up to a 5% absolute increase in the volume of critical structure receiving greater than the specified dose will be considered "variation acceptable," e.g. up to 20% of the rectum may receive a dose of > 75.6 Gy without a protocol deviation. Any increase in critical structure volume greater than 5% receiving more than the specified dose will be considered a "deviation unacceptable." It is at this point that a dose reduction to 77.4 Gy or 75.6 Gy should be implemented. The prescription dose should be the maximum deliverable up to 79.2 Gy while respecting the critical normal structure constraints. Of note, the penile bulb constraint is to be regarded as a guideline, and adherence to this should not, in any way, result in a reduction of the prescription dose or compromised dose coverage of the target volume.

#### **6.6 Treatment Verification** (12/17/13)

6.6.1 First day portal images of each field along with orthogonal isocenter verification images must be obtained. If modifications are made in field shaping or design, a portal image of each modified field along with orthogonal isocenter verification images are required on the first day's treatment of that field. Thereafter, weekly verification images of orthogonal isocenter views (anterior to posterior and lateral projection) are required.

**For IMRT** the intensity profiles of each beam must be independently verified and compared to the planned field intensity. Portal images are not required for IMRT but orthogonal verification images are required, just as for 3DCRT. Real-time ultrasound localization and on-line cone beam CT image guidance are important complements to conventional port films or portal imaging and should be used when available. When CBCT is not available for daily use, weekly port filming/imaging will be required on this study.

**6.6.2** Daily on-line target localization (kV or MV imaging with fiducials, trans-abdominal ultrasound, or other) or off-line adaptive approaches to account for interfraction organ motion and setup variability are permitted on this study but not required.

#### **6.7 Quality Assurance** (4/16/14)

#### **6.7.1** Compliance Criteria for Cases Treated with EBRT

Cases that are treated entirely with external beam radiation therapy must meet the criteria as stated in <u>Sections 6.1.1</u> and <u>6.1.2</u> (see also Tables 1 and 2) to be scored as per protocol. That is, each case will have to meet the requirements in these sections depending on the particular arm of the study selected during randomization. Both the Phase 1 and 2 requirements for a particular arm must be met in order to be scored as per protocol. If only one phase of treatment meets the requirement, the case will be scored with the lower score of either variation acceptable or deviation unacceptable. In addition, the critical structure dose constraints of <u>Section 6.5</u> and Table 3 must be met. In this case also, the patient's treatment will be scored lower when the critical structure score is lower.

The compliance criteria for the situation where the Phase 2 boost is accomplished with brachytherapy is given in Sections 6.8 and 6.9 below.

Acceptable <u>dose heterogeneity</u> for external beam treatment is summarized in Tables 1 and 2.
 The treating physician must carefully consider the tolerance dose/volume to each critical normal structure and unspecified tissue.

#### • Dose Distribution

IROC Philadelphia will display, and compare with isodose distributions for the axial and coronal planes through the planning target volume to verify correct digital submission and conversion. The submitted DVHs for the PTV will then be compared with those generated by NRG Oncology. Per protocol scoring will be considered for those cases in which 98% of the PTV receives the prescription dose.

• Elapsed Days During Radiotherapy

Per Protocol: 1 to 7 break days Variation Acceptable: 8 to 14 days Deviation Unacceptable: > 14 days

- 6.8 Dose Specifications/Technical Considerations: LDR Brachytherapy Boost (12/17/13) (2/4/14) Note: As this protocol allows for treatment with exclusively EBRT or EBRT + a brachytherapy boost (at the discretion of the treating physician) this must be specified at the time of study enrollment. If a patient who was originally intended to receive brachytherapy be found, postenrollment, to be a poor brachytherapy candidate based on transrectal ultrasound examination, he may be switched to EBRT administered per protocol guidelines, but this will result in a protocol deviation. Therefore, it is strongly recommended to obtain ultrasound assessment of prospective brachytherapy patients before enrollment on this study.
- 6.8.1 LDR, permanent seed, brachytherapy boost is permitted at the discretion of the treating radiation oncologist in conjunction with EBRT as described in <u>Section 6.2.3</u>. Implants will only be offered to patients with a prostate volume documented to be <60 cc by transrectal ultrasound examination, an AUA score ≤15, and no prior history of TURP (<u>Section 3.2.7</u>). The implant may be performed under either general or spinal anesthesia and will be performed following the EBRT portion of treatment no more than 4 weeks after its completion.

#### **6.8.2** Preplanning

This will be carried out prior to the procedure or intra-operatively via transrectal ultrasound examination. The prostate will be defined from base to apex in the axial plane at 5 mm slice intervals. The treatment length and prostate volume will be recorded. The CTV is the prostate gland and the proximal seminal vesicles (CTV\_7920). The PTV may be the same as the CTV or a 2-3 mm margin may be added anteriorly and up to 5 mm craniocaudally and laterally at the discretion of the treating physician.

#### **6.8.3** Isotope Selection

lodine-125 or Palladium-103 seeds may be used. The sources will be received and inventoried in accordance with state and federal regulations. If nonsterile loose sources or cartridges are used, at least 10% of the sources will be assayed in such a manner that direct traceability to either the National Institute of Standards and Technology (NIST), an Accredited Dosimetry Calibration Lab (ADCL) or for international participants, the national standards laboratory in their respective country, is maintained. NIST 1999 standards will be used. If sterile source assemblies or strands are used, alternatively non-stranded loose seeds equal to 5% of the total, or five seeds, whichever is fewer, may be ordered and assayed. Agreement of the average measured source strength shall agree with that indicated in the vendor's calibration certificate to within 5%. No measured source strengths should fall outside 10% of that indicated in the vendor's calibration certificate.

- For I-125, the allowable source strength for each seed is 0.277 U to .650 U (NIST 99 or later). For Pd-103 sources, this range is 1.29 U to 2.61 U (NIST 99 or later).
- The vendor's stated source strength shall be used in all dosimetry calculations. Calculations will be performed in accordance with NIST 1999 calibration standards, the point source formalism described in the report generated by AAPM Task Group 43 and subsequent published AAPM Subcommittee Reports. The AAPM's recommendations for Pd-103 dose specifications and prescription are being followed.

#### 6.8.4 Prescription Doses

The prescription dose for permanent seed interstitial boost will be **110 Gy for I-125 and 100 Gy for Pd-103**. Doses will be prescribed as minimal peripheral dose to the PTV.

#### **6.8.5** Postimplant Imaging

A pelvic x-ray with seed count verification will be obtained immediately postimplant. If the seed count does not match the number of seeds implanted, PA and lateral chest x-rays will be obtained to rule out

pulmonary seed migration. CT scan for postimplant dosimetric analysis will be obtained following implant completion. Use of a Foley catheter for this test is encouraged for accurate urethral dosimetry but not required. This may be obtained immediately postoperative on the day of the implant if desired but no later than 5 weeks postimplant. The use of intravesical contrast is encouraged. CT slices should be acquired at ≤3 mm thickness and should encompass the pelvis from, at minimum, the bottom of the sacroiliac joints superiorly to 2 cm caudal to the prostatic apex.

• Structures defined will include the prostate, bladder, and rectum. The rectum will be defined from the bottom of the sacroiliac joints to the ischial tuberosity and will extend to the outer surface of the visualized rectal wall. The postimplant, CT-defined prostate will be defined as the "evaluated target volume" (ETV) and will form the basis for dosimetric analysis.

#### 6.8.6 Dosimetry

Postimplant evaluation will be performed on equipment capable of providing structural and volume-based dosimetric assessment on both the target and critical structures. Volume acquisition will be based on contiguous axial CT slices as described above. Both target volume and critical structures will be contoured on each applicable axial slice. Isodose line displays and dose-volume histograms for all structures will be generated.

- The calculation grid should be set no larger than (2 mm x 2 mm x axial slice width).
- The planning system shall be capable of transmitting data via DICOM RT to TRIAD electronically.
- Guidelines established by the American Brachytherapy Society (Nag 2000) are to be followed.
  DVH-based analysis must be used in the postplan evaluation. The following values shall be
  reported. Vn is the percentage of the ETV that received at least n% of the prescription dose. Dm
  is the minimum dose received by m% of the ETV.
- Target coverage will be documented in terms of V100, V90, V80, D90.
- Dose uniformity will be expressed in terms of V150.
- The rectum will be defined from the bottom of the SI joints to the ischial tuberosity. The maximum rectal dose as well as the volume and percentage of rectum receiving > 100% of the prescription dose will be recorded.

**Note:** All required **LDR** Brachytherapy Boost structures must be labeled as listed in the table in <u>Section 6.4.3</u> for digital RT data submission. Resubmission of data may be required if labeling of structures does not conform to the standard DICOM name listed.

#### **6.8.7** Compliance Criteria

- <u>Per protocol</u>: D90 for the ETV is greater than 90% of the prescription dose but less than 130% of the prescription dose.
- *Variation acceptable*: D90 for the ETV is greater than 80% of the prescription dose, but less than 90% of the prescription dose, or greater than 130% of the prescription dose.
- Deviation unacceptable: D90 for the ETV is less than 80% of the prescription dose.

#### **6.8.8** Dosimetric Data to be Submitted to RTOG

- Copies of preimplant TRUS images with CTV and PTV annotated
- A copy of the implant record generated during the procedure
- A copy of the image taken after the procedure and a copy of the image or scout taken during the post implant CT
- A copy of the postimplant CT scan, ETV and bladder and rectum delineation and dosimetry calculations (must be submitted electronically)
- A copy of the postimplant dosimetry report that contains the information required in <u>Section 6.8.6</u> above.
- 6.9 Dose Specifications/Technical Considerations: HDR Brachytherapy Boost (4/16/14)

  Note: As this protocol allows for treatment with exclusively EBRT or EBRT + a brachytherapy boost (at the discretion of the treating physician) this must be specified at the time of study enrollment. If a patient who was originally intended to receive brachytherapy be found, postenrollment, to be a poor brachytherapy candidate based on transrectal ultrasound examination, he may be switched to EBRT administered per protocol guidelines, but this will result in a protocol deviation. Therefore, it is strongly recommended to obtain ultrasound assessment of prospective brachytherapy patients before enrollment on this study.

Type of HDR planning (CT or TRUS) must be specified at the time of enrollment. Any change of HDR planning technique must be reported to the HDR study co-chair Dr. Bachand in writing prior to the implant, otherwise the patient will no longer be eligible.

6.9.1 HDR brachytherapy boost is permitted at the discretion of the treating radiation oncologist in conjunction with EBRT as described in <u>Section 6.2.3</u>. Implants will only be offered to patients with a prostate volume documented to be <60 cc by transrectal ultrasound examination, AUA symptom index ≤15, and no prior history of TURP (<u>Section 3.2.7</u>). The implant may be performed during the EBRT portion of the treatment or within 2 weeks prior to its initiation or following its completion. The RT should start within 8-10 weeks following the first LHRH administration. The date of HDR brachytherapy implant will constitute the start of RT for those patients receiving implants prior to EBRT.

#### 6.9.2 CT Based HDR Brachytherapy

- All implants will be performed under transrectal ultrasound guidance. Epidural, spinal, or general
  anesthesia may be used. A 12-16 French Foley catheter should be inserted to allow visualization
  of the urethra. Posterior rows of catheters may be advanced into the seminal vesicles under
  TRUS guidance.
- At least 14 treatment catheters should be used to ensure adequate CTV coverage with acceptable dose heterogeneity.
- Fiducial markers identifying the prostatic base and apex could be placed at the time of the implant procedure unless previously placed for guidance of EBRT.
- The use of intraoperative cystoscopy can be used to ensure the absence of treatment catheters within the urethra or bladder. The cystoscope should be retroflexed within the bladder for visualization of the bladder neck. Light pressure on the treatment catheters should result in mucosal tenting confirming adequate coverage at the prostatic base.
- Patients will be treated with either a single implant-single HDR fraction, a single implant-2 HDR fractions delivered over 24 hours with a minimum of 6 hours in between or 2 implants-2 HDR fractions. For patients receiving 2 fractions over 2 implants, the insertions should be done 7 to 14 days apart. No EBRT treatment will be delivered on the day of HDR treatment.
- The treatment planning CT scan must be performed with the patients in the supine position with the Foley catheter in place. Metallic obturators, dummy ribbons and rectal tube or marker must be removed prior to the CT scan. If contrast material is used in the bladder, rectum or urethra, it should be diluted to 10% or less to minimize CT artifact. The scan must include all of the CTV with at least 9 mm superior and inferior margin, and the scan must include the tips of all the implanted catheters. The scan thickness must be ≤0.3 cm and the slices must be contiguous. The field of view (FOV) of axial CT slice should include all the critical structures and target volume on that slice while minimized the overall FOV size to approximately 20 x 20 cm. FOV does not need to include the contour of pelvis. The brachytherapy target volume and normal critical structures must be outlined on all CT slices including the prostate, seminal vesicles, urethra, bladder, and rectum.
- The evaluation of the quality of the implant will be based on the CT using criteria defined below (Section 6.9.10)
- Dwell times in positions located outside of the PTV should be turned down or off to minimize normal tissue irradiated. A dwell time optimization program based on implant geometry or an inverse planning algorithm may be used. Manual optimization is also accepted. An activation volume can be created around the CTV (not posteriorly), allowing optimization of the dwell times immediately outside the CTV/PTV.
- The Clinical Target Volume (CTV) is defined by the physician on the treatment planning CT scan. The CTV is the prostate gland plus any visualized extracapsular extension of tumor. The brachytherapy Planning Target Volume (PTV) is identical to the CTV.
- Critical structures to be defined include the bladder, rectum, and urethra, within the volume of
  interest defined in. The outermost extent of the bladder/rectal wall will define those structures with
  particular attention to bladder base. The urethra is defined by the outer surface of the Foley
  catheter.
- The volume of bladder and rectum receiving 75% of the prescription dose must be kept to less than 1 cc (V75 <1 cc) and the volume of urethra receiving 125% of the prescription dose must be kept to less than 1 cc (V125 <1 cc) and urethral V150 should be 0 cc (V150 = 0 cc). Attempts should be made to limit the volume of urethra receiving ≥115% of the prescription dose to

≤5%. Up to 10% will be considered variation acceptable. If the dose to normal critical structures cannot be kept below the specified level, we recommend readjusting the implant or repeating the implant procedure until a more optimal implant is obtained.

**Note:** All required **HDR** Brachytherapy Boost structures must be labeled as listed in the table in <u>Section 6.4.3</u> for digital RT data submission. Resubmission of data may be required if labeling of structures does not conform to the standard DICOM name listed.

#### **6.9.3** Compliance Criteria

The prescription dose and fractionation is at the discretion of the prescribing physician.

- Single implant-single fraction:
  - A prescription dose of 15 Gy will be delivered to the PTV.
- Single implant-2 fractions:

A prescription dose of 21 Gy will be delivered to the PTV in two equal fractions of 10.5 Gy. The first fraction of 10.5 Gy will be delivered as soon as possible following completion of the implant procedure and treatment planning. Both fractions must be delivered within a single 24-hour period and separated by a minimum of 6 hours. Overnight hospital stay is permitted between fractions if necessary.

#### • <u>2 implants-2 fractions</u>:

A prescription dose of 21 Gy will be delivered to the PTV in two equal fractions of 10.5 Gy, using one implant for each fraction. Both fractions of 10.5 Gy will be delivered as soon as possible following completion of the implant procedure and treatment planning. All catheters will be removed following completion of the treatment after each fraction. Both fractions must be separated by 7 to 14 days.

Ninety percent coverage of the PTV with the prescription dose is considered per protocol, 85% but <90% is considered variation acceptable, and <85% coverage is considered deviation unacceptable. Urethral dose above limits (V125 ≥ 1cc and V150 > 0 cc) is considered deviation unacceptable.

#### **6.9.4** Catheter Position Verification

Visual inspection of the catheters prior to delivery of each treatment is required. If readjustment is needed, the CT planning should be repeated. The physician may adjust the catheters if catheter displacement is identified prior to the treatment.

#### 6.9.5 Catheter Removal

After completion of the treatment all implant catheters will be removed.

#### **6.9.6** Data Submission

All data will be digitally submitted to the IROC Philadelphia and include CT data, normal critical structures, all PTV contours, and digital DVH data for all normal critical structures, the PTV for dose plan, a copy of the daily treatment chart for EBRT and Brachytherapy.

#### **6.9.7** Quality Assurance

Individual case review will be overseen by Dr. Bachand, the HDR brachytherapy study co-chair overseeing this subgroup of patients enrolled on this protocol, as specified in <u>Section 6.10.</u>

#### 6.9.8 TRUS Based HDR Brachytherapy

- All implants will be performed under transrectal ultrasound guidance. Epidural, spinal, or general anesthesia may be used.
- At least 14 treatment catheters should be used to ensure adequate CTV coverage with acceptable dose heterogeneity.
- The treatment planning TRUS must be performed with the patient in the supine position with the 12-16 French Foley catheter in place. Two sets of TRUS images are taken. The first set will be done prior to the insertion of implant catheters when the target volume and the urethra are visible. The second set of images is done after the insertion of the implant catheters and is used for treatment planning. The scan must include all of the CTV with at least 1 cm superior and inferior margin, and the scan must include the tips of all the implanted catheters. The scan thickness must be ≤0.3 cm and the slices must be contiguous. The brachytherapy target volume and normal critical structures must be outlined on all slices including the CTV, urethra and rectum.
- Both transrectal ultrasound scans, one prior to implant catheter insertion and one with catheters in place, must be submitted for each patient.
- Dwell times in positions located outside of the PTV should be turned down or off to minimize
  normal tissue irradiated. A dwell time optimization program based on implant geometry or
  an inverse planning algorithm may be used. Manual optimization is also accepted. An
  activation volume can be created around the CTV (not posteriorly), allowing optimization of the

dwell times immediately outside the CTV/PTV. A dwell time optimization program based on implant geometry or an inverse planning algorithm may be used. Manual optimization is also accepted.

- The Clinical Target Volume (CTV) is defined by the physician on the treatment planning CT scan. The CTV is the prostate gland plus any visualized extracapsular extension of tumor. The brachytherapy Planning Target Volume (PTV) is identical to the CTV.
- Critical structures to be defined using TRUS planning include the rectum and the urethra within
  the volume of interest defined above. The rectum is defined as the outermost extent of the rectal
  wall from the TRUS probe, the lateral boarders extends to the edge of the TRUS image. The
  urethra is defined by the outer surface of the Foley catheter and it is contoured as a solid
  structure.
- The volume of rectum receiving 80% of the prescription dose must be kept to less than 0.5 cc (V80 <0.5 cc) and the volume of urethra receiving 130% of the prescription dose should be 0 cc and the urethra D10 should be < 115%. Attempts should be made to limit the volume of urethra receiving ≥115% of the prescription dose to ≤5%.
- All TRUS based HDR treatment should be delivered with TRUS probe in the patient so the dosimetry may be accurately reproduced.

**Note:** All required **HDR** Brachytherapy Boost structures must be labeled as listed in the table in <u>Section 6.4.3</u> for digital RT data submission. Resubmission of data may be required if labeling of structures does not conform to the standard DICOM name listed.

#### 6.9.9 Compliance Criteria

The prescription dose and fractionation is at the discretion of the prescribing physician.

Single implant-single fraction:

A prescription dose of 15 Gy will be delivered to the PTV.

• Single implant-2 fractions:

A prescription dose of 21 Gy will be delivered to the PTV in two equal fractions of 10.5 Gy. The first fraction of 10.5 Gy will be delivered as soon as possible following completion of the implant procedure and treatment planning. Both fractions must be delivered within a single 24-hour period and separated by a minimum of 6 hours. Overnight hospital stay is permitted between fractions if necessary.

#### • 2 implants-2 fractions:

A prescription dose of 21 Gy will be delivered to the PTV in two equal fractions of 10.5 Gy, using one implant for each fraction. Both fractions of 10.5 Gy will be delivered as soon as possible following completion of the implant procedure and treatment planning. All catheters will be removed following completion of the treatment after each fraction. Both fractions must be separated by 7 to 14 days.

Ninety percent coverage of the PTV with the prescription dose is considered per protocol, 85% but <90% is considered variation acceptable, and <85% coverage is considered deviation unacceptable. Urethral dose above limits (V130 > 0 cc and D10 < 118%) is considered deviation unacceptable.</li>

#### 6.9.10 Catheter Removal

After completion of the treatment all implant catheters will be removed.

#### **6.9.11** Data Submission

All data will be digitally submitted to TRIAD and include both TRUS scans (with/without implant catheter), normal critical structures, all PTV contours, and digital DVH data for all normal critical structures, and the PTV for dose plan.

#### **6.9.12** Quality Assurance

Individual case review will be overseen by Dr. Bachand, the HDR brachytherapy study co-chair overseeing this subgroup of patients enrolled on this protocol, as specified in <u>Section 6.10</u>.

#### **6.10** R.T. Quality Assurance Reviews (4/16/14)

The study co-chairs for the respective RT modalities offered in this trial will oversee quality assurance reviews for patients treated in those respective fashions. These reviews will be ongoing and performed remotely. RT quality assurance reviews will be facilitated by IROC Philadelphia.

#### 6.11 Radiation Therapy Adverse Events

**6.11.1** All patients will be seen weekly by their treating radiation oncologist while undergoing EBRT. Any observations with respect to the following symptoms/side effects will be recorded:
- Bowel/rectal irritation manifesting as cramping, diarrhea, urgency, proctitis, or hematochezia
- Urinary frequency, urgency, dysuria, hematuria, urinary tract infection, or incontinence
- Radiation dermatitis
- **6.11.2** Clinical discretion may be used in managing radiotherapy-related side effects. Diarrhea/rectal frequency/urgency may be managed with diphenoxylate or loperamide. Bladder irritation may be mitigated with phenazopyridine. Urinary frequency/urgency can be managed with anticholinergic agents or alpha-blockers such as tamsulosin. Erectile dysfunction can be managed with phosphodiesterase (PDE) inhibitors such as sildenafil.

# 6.12 Radiation Therapy Adverse Event Reporting

See Section 7.17.

#### 7.0 DRUG THERAPY

**7.1** Treatment (12/17/13)

Androgen suppression (AS) must begin within 6 weeks after registration (if not started prior to registration) and will be administered in both Arms 1 and Arm 2. TAK-700 will begin at the same time as AS. Radiation therapy will begin 8-10 weeks after the initiation of AS and will be given as specified in <u>Section 6.0</u>.

For those who started LHRH therapy prior to enrollment, they must have started this <50 days prior to enrollment. In addition, the same goal of starting RT 8-10 weeks from the start of LHRH therapy will be maintained.

# **7.1.1** Arm 1

Patients on Arm 1 will receive standard AS with LHRH agonist and oral anti-androgen. LHRH agonist will continue for 24 months (cumulative 24 month total dose) from initiation. **Oral anti-androgen will be discontinued at the end of radiation therapy.** 

**7.1.2** Arm 2

Patients on Arm 2 will receive the same standard AS with LHRH agonist and oral antiandrogen as administered in Arm 1, but also will receive the study drug TAK-700 (for 2 years) as detailed in <a href="Section">Section</a> 7.5 below.

- 7.1.3 For patients on either Arm 1 or Arm 2 who began ADT prior to enrollment, if prior treatment was with LHRH agonist alone, an oral anti-androgen (plus or minus TAK-700) should be added at the time of enrollment.
- **7.2 LHRH agonists (such as leuprolide, goserelin, buserelin, triptorelin)** (12/17/13) Refer to the package insert for detailed pharmacologic and safety information.
- ,7.2.1 <u>Description</u>: LHRH agonists are long-acting analogs of the native LHRH peptide and are effective at reducing serum testosterone. Analogs approved by the FDA (or by Health Canada for Canadian institutions) can be used in this study.
- **7.2.2** Supply: Commercially available. (NOTE: Buserelin is not commercially available in the United States. It is commercially available for use in Canada and other countries outside of the United States.)
- **7.2.3** Storage: LHRH analogs should be stored as directed by the commercial supplier.
- 7.2.4 Administration: LHRH analogs are administered with a variety of techniques, including subcutaneous insertion of a solid plug in the abdominal wall (Zoladex), intramuscular injection (Lupron), subcutaneous injection (Eligard), or insertion of a long-acting cylinder that slowly releases the agent (Viadur). The manufacturer's instructions should be followed.
- 7.2.5 Toxicity: Consult the package insert for comprehensive toxicity information. Class-related toxicity is generally a manifestation of the mechanism of action and due to low testosterone levels. In the majority of patients testosterone levels increased above baseline during the first week, declining thereafter to baseline levels or below by the end of the second week of treatment. The most common side effect of LHRH analogs is vasomotor hot flashes; edema, gynecomastia, bone pain, thrombosis, and gastrointestinal disturbances have occurred. Potential exacerbations of signs and symptoms during the first few weeks of treatment is a concern in patients with vertebral metastases and/or urinary obstruction or hematuria which, if aggravated, may lead to neurological problems such as temporary weakness and/or paresthesia of the lower limbs or worsening of urinary symptoms. Other side effects include impotence and loss of libido, weight gain, depression, dizziness, loss of bone density, anemia, increased thirst and urination, unusual taste in the mouth, skin redness or hives, pain at injection site, and muscle

mass and strength loss, hair changes, penile length and testicular volume loss, increased cholesterol, hypertension, diabetes exacerbation, emotional lability, nausea, vomiting, and rarely allergic generalized rash and difficulty breathing.

# **7.3** Eulexin (flutamide)\_(12/17/13)

Refer to the package insert for detailed pharmacologic and safety information.

- 7.3.1 <u>Description</u>: Flutamide is a substituted anilide. It is a fine, light, yellow powder, insoluble in water but soluble in common organic solvents such as aromatic or halogenated hydrocarbons. Its concentration in plasma can be determined by gas chromatography. Flutamide is a nonsteroidal antiandrogen that is metabolized into a hydroxylated derivative, which effectively competes with the hydrotestosterone for androgen receptor sites.
- **7.3.2** Supply: Commercially available.
- **7.3.3** Storage: Flutamide should be stored at temperatures ranging from 20-30 °C (36 °-86 °F) and protected from excessive moisture.
- 7.3.4 Administration: The drug is administered orally at a dose of 250 mg (two 125-mg capsules) three times a day for a total daily dose of 750 mg. Flutamide will begin 8-10 weeks prior to radiotherapy and continue throughout radiotherapy. Administration will be suspended only if there is an apparent or suspected reaction to the drug. See Section 7.3.6. Flutamide will be terminated on the last day of radiotherapy. During radiotherapy interruptions, flutamide will be continued.
- 7.3.5 Toxicity: Consult the package insert for comprehensive toxicity information. The reported side effects of treatment include diarrhea and anemia. A high percentage of patients treated with flutamide alone developed gynecomastia within 2 to 8 months. There have been post-marketing reports of hospitalization, and, rarely, death due to liver failure in patients taking flutamide. Evidence of hepatic injury included elevated serum transaminase levels, jaundice, hepatic encephalopathy, and death related to acute hepatic failure. The hepatic injury was reversible after prompt discontinuation of therapy in some patients. Approximately half of the reported cases occurred within the initial 3 months of treatment with flutamide. Other side effects include impotence and loss of libido, fatigue, and rarely photosensitivity.
- 7.3.6 Dose Modifications: If gastrointestinal disturbances (cramps, diarrhea) occur prior to initiation of radiotherapy, flutamide will be withheld until the side effects subside; the drug will then be reintroduced at a dose of 250 mg/day and increased (at 3-day intervals) to 500 mg/day and then to 750 mg/day as tolerated. If gastrointestinal disturbances occur after administration of radiotherapy, it might be difficult to identify their cause. However, if severity of diarrhea exceeds the level commonly observed during pelvic irradiation, the toxicity will be ascribed to flutamide and the drug will be permanently discontinued. ALT will be measured pretreatment, then monthly during oral antiandrogen therapy. If ALT increases ≥ 2 x upper institutional limit of normal, flutamide must be discontinued. Elevated ALT values to < 2x the institutional upper limit of normal are subject to dose modifications or discontinuation of anti-androgen at the discretion of the treating physician.</p>

# **7.4** Casodex (bicalutamide) (12/17/13)

Refer to the package insert for detailed pharmacologic and safety information.

- 7.4.1 <u>Description</u>: Bicalutamide is a nonsteroidal antiandrogen, which has no androgenic or progestational properties. The chemical name is propanamide, N-[4-cyano-3(trifluoromethyl)phenyl]- 3- [(4-fluorophenyl)sulphonyl]- 2- hydroxy- 2- methyl, (+,-). Bicalutamide is a racemic mixture with the antiandrogen activity residing exclusively in the (-) or R-enantiomer. Bicalutamide has a long half-life compatible with once-daily dosing. Bicalutamide is well tolerated and has good response rates in phase II trials (Kennealey and Furr, 1991, Tyrrell 1994).
- **7.4.2** Supply: Commercially available.
- 7.4.3 Storage: Bicalutamide should be stored in a dry place at room temperature between 68°-77°F.
- 7.4.4 Administration: Bicalutamide is administered orally at a dose of one 50 mg tablet per day. Bicalutamide will begin 8-10 weeks prior to radiotherapy and continue throughout radiotherapy. Administration will be suspended only if there is an apparent or suspected reaction to the drug. Bicalutamide will be terminated on the last day of radiotherapy. During radiotherapy interruptions, bicalutamide will be continued.
- 7.4.5 <u>Toxicity</u>: Consult the package insert for comprehensive toxicity information. In animal experiments, birth defects (abnormal genitalia, hypospadias) were found in male offspring from female animals dosed with bicalutamide during pregnancy. Although offspring from male animals dosed with bicalutamide did not show any birth defects, patients enrolled in this trial are advised not to cause pregnancy nor donate sperm while receiving protocol therapy or during the first 3 months after cessation of therapy. The use of

barrier contraceptives is advised. The most frequent adverse events reported among subjects receiving bicalutamide therapy are breast tenderness, breast swelling, and hot flashes. When bicalutamide 50 mg was given in combination with an LHRH analog, the LHRH analog adverse event profile predominated with a high incidence of hot flashes (53%) and relatively low incidences of gynecomastia (4.7%) and breast pain (3.2%). Other side effects include impotence and loss of libido, fatigue, and rarely photosensitivity and diarrhea.

7.4.6 <u>Dose Modifications</u>: Bicalutamide should be discontinued in instances of chemical liver toxicity. ALT will be measured pretreatment and then monthly during antiandrogen therapy. If the ALT rises ≥ 2 x the institutional upper limit of normal, bicalutamide must discontinued. Elevated ALT values to < 2x the institutional upper limit of normal are subject to dose modifications or discontinuation of anti-androgen at the discretion of the treating physician.

# 7.5 Study Drug (TAK-700) Administration (TAK-700, IND # 115368) (12/17/13)

To supplement the toxicity information contained in this document, investigators must obtain the current version of the Investigator Brochure for comprehensive pharmacologic and safety information. The Investigator's Brochure is available on the NRG Oncology/RTOG web site under protocol-specific materials/regulatory resources.

# 7.5.1 Dose and Regimen

TAK-700 will initially be given at 300 mg BID (600 mg per day) orally, continuously for 2 years, beginning at the same time as androgen suppression (AS). See Section 7.6 for dose modification and supportive care guidelines. TAK-700 should be taken twice daily at the same time each day, but not less than 6 hours apart, and may be taken with or without food. Missed doses of study drug will not be made up. Patients will be given a diary to record study drug dosing. If a dose is missed, the missed dose will be recorded as "not taken." The next dose will be taken at the next scheduled time.

#### 7.6 TAK-700 Dose Modification and Supportive Care Guidelines (12/17/13)

The investigator should determine if an AE is related to TAK-700. Adverse events considered at least possibly related to TAK-700 may require a dose reduction (Table 7-1), a temporary hold, or permanent discontinuation.

Depending on the AE, following partial or complete resolution of symptoms, the dose of TAK-700 may be increased at 2-week intervals to the next higher dose level until the original dose level has been reached. Guidelines for modification of the dose based on the severity of the AE are provided in this section.

#### 7.6.1 Dose Levels for TAK-700

The TAK-700 dose levels to be applied for all dose modifications are defined in Table 7-1.

| Table 7-1 Dose Modifications for TAK-700 | |
|---|---|
| Dose Level TAK-700 Dose | |
| | (Tablets and Timing of Administration) |
| 0 | 300 mg BID (100 mg x 3 BID) |
| -1 | 200 mg BID (100 mg x 2 BID) |
| -2 None (dosing hold or temporary | |
| discontinuation) | |

#### 7.6.2 <u>Dose Modifications</u>

Dose modifications should be based on CTCAE version 4.0. Dose reduction for Grade 1 AEs is not required. Dose reduction for Grade 2 events should only be considered when the AE is judged by the investigator to be clinically intolerable. For TAK-700 Grade ≥2 AEs, the dose modification of TAK-700 should follow the Dose Reduction and Re-escalation guidelines (Sections 7.6.3 and 7.6.4, respectively). For events of fatigue, nausea, vomiting, diarrhea, and hypertension, refer to Section 7.6.6, Specific Guidelines for Possible TAK-700 Related Toxicities.

#### **7.6.3** Criteria for TAK-700 Initial Dose Reduction

Asymptomatic Grade 3 or 4 laboratory findings may not require dose modification (i.e. dose hold or reduction) especially if these are not considered to be clinically significant or related to study drug. The decision to modify the dose should be based on the investigator's clinical judgment.

Grade 3 or 4 AEs that are considered at least possibly related to study drug require a dosing hold, i.e. hold for a minimum of 2 weeks. The investigator should identify other potential causes of AEs. For a

clinically intolerable Grade 2 AE that is considered at least possibly related to study drug, the dose should be decreased by 1 dose level for 2 weeks.

Once the dose is reduced, reassessment is required at least every 2 weeks until the event is resolved or stabilized. However, the frequency of reassessment should be increased as clinically indicated. If the grade worsens at any time, the dose should be decreased in accordance with the guidelines for the worst grade.

#### **7.6.4** Criteria for TAK-700 Dose Re-escalation

#### Re-escalation for Grade 2 Intolerable Adverse Events

Re-escalation of TAK-700 after resolution or improvement of a Grade 2 intolerable AE will follow the criteria below:

- (1) If the AE grade improves to Grade 0, 1, or Grade 2 tolerable AE, re-escalate the dose by 1 level.
- (2) If the AE remains at intolerable Grade 2 or worsens to Grade > 3, hold TAK-700 for 2 weeks followed by a reassessment. Follow the re-escalation guidelines for Grade 3 or 4 AEs as defined below.

Reassess the AE after 2 weeks, or sooner if the AE worsens. Continue to reassess at least every 2 weeks until the event is resolved or stabilized. Continue to adjust the TAK-700 dose until the dose is optimally titrated. If the dose has been held for 6 weeks, TAK-700 should be discontinued permanently.

#### Re-escalation of TAK-700 Following a Grade 3 or 4 Adverse Event

Re-escalation following a Grade 3 or 4 AE will follow the criteria below:

- (1) If the AE grade improves to Grade 0, 1, or Grade 2 tolerable AE, re-escalate the TAK-700 dose by 1 level.
- (2) If the AE improves to Grade 2 but is still intolerable, hold dosing for another 2 weeks. Follow the reescalation guidelines for Grade 2 intolerable AEs as defined in Section 7.6.4.
- (3) If the AE is Grade 3 or 4 after 2 weeks, hold dosing for another 2 weeks and reassess again after 2 weeks.

Reassess the AE after 2 weeks, or sooner if the AE worsens. Continue to reassess at least every 2 weeks until the event is resolved or stabilized. Continue TAK-700 dose adjustment until the dose is optimally titrated.

#### **7.6.5** Criteria for Discontinuation of TAK-700

If the adverse event persists at ≥ Grade 3 for more than 6 weeks, permanently discontinue treatment with TAK-700. The TAK-700 dose may also be discontinued permanently if judged by the investigator to be clinically intolerable despite dose reduction, and the dose cannot be optimally titrated.

#### 7.6.6 Specific Guidelines for Possible TAK-700-Related Toxicities

This section provides the required dose modifications for study drugs and recommended clinical management of patients who experience AEs that are considered by the investigator to be related to TAK-700.

#### Fatigue

Grade 2 to Grade 3 fatigue has occurred in some patients receiving TAK-700 without concomitant prednisone. Less severe Grade 1 or Grade 2 fatigue has been reported in some men receiving concomitant prednisone; other factors such as acute androgen deprivation may also contribute to symptoms.

Dose modification for Grade 2 fatigue is optional but may be helpful by slowing the induction to full androgen deprivation. Grade 3 fatigue should be treated according to the general outlines in <u>Section 7.6.2</u>, including initial hold and re-introduction of TAK-700 with subsequent titration at 2 week intervals to the patient's tolerated dose level.

#### Gastrointestinal Adverse Events

In previous and ongoing clinical studies, episodic and not necessarily dose-related gastrointestinal toxicities have occurred.

#### Nausea and/or Vomiting

Grade 1 - No action required

Grade 2 – Concomitant antiemetics may initially be administered without dose reduction. If Grade 2 nausea or vomiting persists and is intolerable, dose reduction and re-escalation should follow Grade 2 Dose Reduction and Dose Re-escalation guidelines.

Grade 3 or 4 – Supportive care regimen should follow local standard of care. Follow Dose Reduction and Dose Re-escalation guidelines.

<u>Note</u>: It is possible that nausea and vomiting could be secondary to acute adrenal insufficiency. If nausea and vomiting occur in the setting of severe fatigue, prostration, or hypotension, blood should be obtained to check the electrolytes. Institutional standard of care should be followed in the presence of electrolytes imbalance. Even if the vomiting occurs shortly following the TAK-700 dose, no re-dosing of TAK-700 will be done.

#### Diarrhea

Prophylactic antidiarrheals will not be used in this protocol; however, patients will be treated according to institutional standard of care. Fluid intake should be maintained to avoid dehydration.

#### Hypertension

If new onset or worsening of established hypertension occurs and the potassium level is < 3.5 mEq/L, in the absence of other causes such as new diuretic therapy, it suggests a TAK-700-related mineralocorticoid syndrome. A plasma renin activity that is undetectable or low also suggests such a syndrome rather than a secondary cause. While addressing underlying factors or compliance with current antihypertensives, dose modification should be initiated according to the general guidelines outlined in Section 7.6.3.

If other causes are identified as the reason for new or worsening hypertension, the investigator should follow the institution's local standard of care treatment and the dose of TAK-700 can be adjusted upwards in accordance with the general guidelines in <u>Section 7.6.3</u>.

#### Suspected or Possible Adrenal Insufficiency

If patients experience adrenal insufficiency, the adrenal insufficiency may have the more nonspecific manifestations of glucocorticoid insufficiency, rather than the more specific electrolyte abnormalities of mineralocorticoid insufficiency. Patients experiencing severe physiological stress (eg, surgery, severe infection) should be carefully monitored for adrenal insufficiency. Concomitant medications may complicate the picture of adrenal insufficiency, in particular in patients who are on beta-blockers or diuretics. Concomitant illness such as infection might similarly trigger or worsen symptoms of otherwise mild adrenal insufficiency. Grading of adrenal insufficiency should follow CTCAE criteria (version 4.0). In all cases, actions should include a thorough review for other possible causes or contributors to the presenting symptoms (eg, infection, anemia, or newly introduced concomitant medications).

# Abnormal Liver Enzymes

| Table 7-2 Management of Abnormal AST or ALT Bearing a Possible Relationship to TAK-700 Treatment | | |
|---|---|---|
| AST and/or ALT Elevation Grade (Per NCI CTCAE) | Concurrent Bilirubin Level | TAK-700 Dose Modification |
| Grade 1 | ≥ 1.5 x ULN | Hold until bilirubin resolves to < 1.5 ULN Dose at the next lower dose |
| Grade 2 | < 1.5 x ULN | Hold until ALT/AST resolve to Grade 1 Dose at the next lower dose level |
| Grade 2 | ≥ 1.5 x ULN | Discontinue TAK-700 |
| Grade ≥ 3 | Any | Discontinue TAK-700 |

Note: Following TAK-700 dose de-escalation due to AST/ALT and/or bilirubin abnormalities, no

re-escalation is permitted.

#### 7.6.7 Overdose

The maximum tolerated or efficacious dose for TAK-700 has not been determined. An overdose is defined as deliberate or accidental administration of study medication at a dose above that which is assigned to that individual subject. In the event of drug overdose, the principal investigator should be notified immediately and the patient observed closely for adverse effects. The patient should be treated symptomatically as appropriate, and the incident of overdose and related AEs and/or treatment-documented in the patient's medical record. Patients who may have overdosed and who have possible manifestations of adrenal insufficiency may be treated acutely with oral steroids as tolerated.

#### 7.7 Excluded Concomitant Medications and Procedures

The following medications and procedures are prohibited during the study:

- Any investigational agent other than TAK-700
- Other anticancer therapy, except for GnRH analogs, antiandrogens, and radiation therapy
- Hormonal therapies including estrogens or herbal products
- · Ketoconazole or aminoglutethimide
- Chronic use of systemic corticosteroids, such as oral prednisone
- Patients must be instructed not to take any medications, including over-the-counter products and vitamins, minerals and other dietary supplements, without first consulting with the investigator.

#### 7.8 Precautions and Restrictions

It is not known what effects TAK-700 has on human pregnancy or development of the embryo or fetus. Therefore, male patients should avoid impregnating a female partner. Patients should use effective methods of contraception through defined periods during and after study treatment as specified below. If a female partner of a male patient becomes pregnant during the male patient's participation in this study, this must be reported to Millennium Pharmacovigilance (or designee) immediately (see below). Every effort should be made to follow the pregnancy for the final pregnancy outcome (i.e. delivery, still birth, miscarriage).

Millennium Pharmacovigilance
SAE and Pregnancy Reporting Contact Information:
North America
PPD, Inc.
Safety and Medical Management, US
Fax: +1 888-488-9697

Hotline number (available 24/7): 1-800-201-8725

Male patients, even if surgically sterilized (eg, status postvasectomy) must agree to either practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from intercourse.

Nonclinical studies of TAK-700 biotransformation by human hepatic and intestinal microsomes indicate that CYP enzymes have only a minor role in the metabolism of TAK-700. Based on these findings, there is very low risk that the metabolism of TAK-700 will be affected by CYP-mediated interactions due to other drugs.

In vitro studies indicate that TAK-700 is a weak to moderate inhibitor of CYP1A2, 2C9, and 2C19 (Kis of 8.9, 15.4, and 19.4  $\mu$ mol/L, respectively). These findings indicate that TAK-700 has the potential to inhibit the metabolism of drugs that are substrates of CYP1A2 and may possibly inhibit the metabolism of drugs that are substrates of 2C9 and 2C19.

Drugs that are primarily metabolized by these CYP isoforms should be used with caution when administered concomitantly with TAK-700.

In vitro studies demonstrate that TAK-700 is a substrate for P-gp but the affinity of TAK-700 for P-gp is low. Studies show that TAK-700 was not an inhibitor of P-gp. Based on these findings, there is very low risk of a P-gp-based interaction of TAK-700 with other drugs.

No single-dose effect of TAK-700 on QTc interval has been observed in healthy male subjects, and no trend in QTc interval has been observed to date in patients with mCRPC in the open-label phase 1/2 TAK-700\_201 study. Until more data are available, patients with underlying cardiac rhythm abnormalities or in patients on other drugs that may affect the QTc interval should be monitored closely.

# 7.9 Blinding and Unblinding

This is an open-label study.

#### **7.10** Description of Investigational Agent (5/2/12)

TAK-700 is manufactured by Takeda Pharmaceutical Company, Ltd., Osaka, Japan. TAK-700 will be supplied as pale red film-coated tablets. Each tablet will contain 100 mg of TAK-700. Further details are provided in the TAK-700 Investigator's Brochure which is available on the RTOG web site under protocol-specific materials/regulatory resources.

#### 7.11 Preparation, Reconstitution, and Dispensation

TAK-700 is an antineoplastic agent, and as with other potentially toxic compounds, caution should be exercised when handling TAK-700.

# 7.12 Packaging and Labeling

TAK-700 supplied as 100 mg tablets packaged in high density polyethylene bottles with child-resistant cap and with a 3 gram desiccant. Each bottle will be labeled in accordance with all regulatory requirements appropriate for the country(ies) in which the study will be conducted.

#### **7.13** Storage, Handling, and Accountability (12/17/13)

TAK-700 supplied as 100-mg film-coated tablets should be stored in the original dispensing bottle at the conditions described in the product label. The drug supply must be kept in an appropriate, limited-access, secure place until it is dispensed to study enrollees, returned to the sponsor, or forwarded to the sponsor's designee for destruction. Drug supplies will be counted and reconciled at the site before being returned.

At the completion of the study, unused supplies will be destroyed at the site according to the institution's policy for drug destruction. Sites should complete the drug destruction form located on the NRG Oncology/RTOG website (<a href="www.rtog.org">www.rtog.org</a>) under protocol-specific materials/regulatory resources and send it to Biologics (see <a href="Section 7.14.1">Section 7.14.1</a> below for contact information).

The investigator must maintain 100% accountability for all study medication received and dispensed during his or her entire participation in the study. Proper drug accountability includes, but is not limited to:

- Continuously monitoring expiration dates if retest date is provided to the investigator.
- Frequently verifying that actual inventory matches documented inventory. Verifying that the drug accountability log is completed for the drug lot used to prepare each dose.
- Verifying that all containers used are documented accurately on the log.
- Verifying that required fields are completed accurately and legibly.

If any dispensing errors or discrepancies are discovered, the sponsor must be notified immediately. The investigator must maintain a current inventory (drug accountability log) of all study medication delivered to the site, inventory at the site, and patients' use records. This log must accurately reflect the drug accountability of the study medication at all times. The following information will be recorded at a minimum: protocol number and title, name of the investigator, site identifier and number, description of the study medication, expiry and/or retest date, date and amount dispensed, and the date and amount returned to the site by the patient, including the initials of the person dispensing and receiving the study medication. The log should include all required information as a separate entry for each patient to whom study medication is dispensed. At appropriate intervals, a representative from the sponsor will perform clinical study material accountability and reconciliation. The investigator will retain the original documentation regarding clinical study material accountability, return, and/or destruction. The investigator

will be notified of any expiry date or retest date extension of clinical study material during the study conduct. On expiry date notification from the sponsor or designee, the site must complete all instructions outlined in the notification, including segregation of expired clinical study material for return to the sponsor or its designee for destruction. In the event of expiry date extension of supplies already at the study site, supplies will be relabeled with the new expiry date at that site.

#### **7.14** Supply (5/1/12)

This study will be conducted under an IND to be held by RTOG (NRG Oncology) and will require FDA submission and approval as part of the IND. TAK-700 will be supplied to patients in the study free of charge.

The Study Agent Shipment Form [SASF; available on the NRG Oncology/RTOG web site, <a href="www.rtog.org">www.rtog.org</a>, under protocol-specific materials/regulatory resources] for U.S. and Canadian sites must be submitted to the CTSU Regulatory Office (Fax 215-569-0206) as soon as the individual responsible for the study agent has been identified. This must be done prior to registration of the institution's first case. The drug supply will not be shipped by Biologics, Inc. until the patient has been registered. Canadian shipments may require additional time. NRG Oncology will notify Biologics, Inc. to initiate each of these shipments after registration of the patient. Drug shipments may not be immediate if the protocol includes a delay in the initial dosing. Drug will be delivered in time for the patient's first dose.

#### **7.14.1** Biologics, Inc. TAK-700 Distribution

Upon receipt of patient registration/randomization, NRG Oncology will notify Biologics via e-mail. Biologics will then perform the following process:

- Confirm SASF and Registration/Randomization;
- Place call directly to the study site contact listed on the SASF confirming that the registration/randomization was received and to:
  - o Collect any additional patient or shipping information required per protocol;
  - o Arrange the date and time of arrival for the study drug;
  - Ship the initial shipment of study drug supply per protocol directly to SASF address; any discrepancies will be addressed with the CTSU.

Biologics, Inc. ships study drug the same day of receipt of patient registration/randomization if received before 2:00pm ET on Monday through Friday. Ambient drug like TAK-700 allows for Friday shipment with Monday delivery. Authorized and complete orders received after 2:00pm ET Monday through Friday will be processed and shipped the next business morning.

| TAK-700 Shipment Schedule | | | | |
|---|---|---|---|---|
| Patient<br>registered with<br>NRG Oncology | E-order<br>transmitted by<br>NRG Oncology | E-order<br>Received by<br>Biologics<br>(before 2PM ET) | Order shipped | Order received at site |
| Monday | Monday | Monday | Monday | Tuesday |
| Tuesday | Tuesday | Tuesday | Tuesday | Wednesday |
| Wednesday | Wednesday | Wednesday | Wednesday | Thursday |
| Thursday | Thursday | Thursday | Thursday | Friday |
| Friday | Friday | Friday | Friday | Monday |

All shipments are sent via *FedEx for Priority Overnight* delivery. Study Drug (TAK-700) is shipped in a Biologics, Inc. branded container appropriate to maintain temperature stability.

#### **Shipment Schedule**

**Initial shipment** – 18 Bottles of study drug to be taken continuously

6 months at 300mg (3 tabs/100mg each) PO BID

**Biologics places follow-up call** during month 5 for subsequent shipment of study drug **Subsequent shipment 2** – 18 Bottles of study drug to be taken continuously

6 months at 300mg (3 tabs/100mg each) PO BID

Biologics places follow-up call during month 11 for subsequent shipment of study drug Subsequent shipment 3 – 18 Bottles of study drug to be taken continuously

6 months at 300mg (3 tabs/100mg each) PO BID

Biologics places follow-up call during month 17 for subsequent shipment of study drug Subsequent shipment 4 – 18 Bottles of study drug to be taken continuously

6 months at 300mg (3 tabs/100mg each) PO BID

# For all drug shipments from Biologics, Inc.:

- Study Drug will be shipped in original manufacturers packaging. Bottles are placed in a Ziploc bag with a patient specific label adhered to the outside of the bag.
- Each shipment includes a patient label on the Ziploc bags with the following information:
  - The Study Number (i.e. RTOG 1115);
  - IND caution statement and/or local regulatory statements;
  - Drug identification (TAK-700)
  - **Expiration**
  - Storage conditions
  - Dosing instructions (Take as Directed per Protocol)
  - Subject ID number (e.g. 1115-YYY, where the study number and sequence number represents the unique patient identifier assigned by NRG Oncology at registration);
  - The patient's initials (i.e. first, middle, last)
  - A blank line for the site pharmacist to enter the patient's name;
  - Administration instructions (i.e. "Take xx tablets every day for xx days");
  - Storage instructions (i.e. "Store at controlled room temperature, xx degrees"):
  - Emergency contact instructions;
- Enclose a packing slip that includes the quantity of drug provided with a section to be completed once received by the site coordinator. This section includes confirmation of drug receipt, verification of package contents, and instruction to fax the completed packing slip to Biologics.
- Packages are tracked until confirmed delivered and delivery exceptions are managed with the highest level of urgency to ensure therapy start date adherence. Packing slips with the shipment tracking number included will be faxed to the designated site coordinator for all shipments.

Please contact the drug distributor, as listed below, directly for shipment tracking information and anticipated delivery dates or if a shipment has not been received by the expected date.

Unused supplies at the sites will be destroyed on site per local guidelines/standard operating procedures. Additional questions about supply and delivery should be directed to:

> Clinical Trial Services Biologics, Inc. 120 Weston Oaks Court Cary, NC 27513 (800) 693-4906

clinicaltrials@biologicstodav.com

#### **7.14.2** Study Agent Accountability

Drug accountability records must be maintained at all sites according to good clinical practices and NCI guidelines using the Investigational Agent Accountability Record (IAAR) form.

#### 7.15 Modality Reviews (2/4/14)

This study will undergo hormone therapy review for TAK-700. The Principal Investigator, M. Dror Michaelson, MD, PhD, will perform a Hormone Therapy Assurance Review of all patients who receive or are to receive TAK-700 in this trial. The goal of the review is to evaluate protocol compliance. The review process is contingent on timely submission of hormone treatment data as specified in Section 12.1. The

scoring mechanism is: per protocol; unacceptable deviation; not evaluable. A report is sent to each institution once per year to notify the institution about compliance for each case reviewed in that year.

# **7.16** Adverse Events (12Jun2018)

The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 will be utilized until March 31, 2018, for all AE reporting, CTEP-AERS, and case report forms. CTCAE version 5.0 will be utilized for CTEP-AERS reporting beginning April 1, 2018; all study case report forms will continue to use CTCAE version 4.0. All appropriate treatment areas should have access to a copy of CTCAE versions 4.0 and 5.0, which can be downloaded from the CTEP web site (https://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm).

Adverse events (AEs) that meet expedited reporting criteria defined in the table(s) below will be reported via the CTEP-AERS (CTEP Adverse Event Reporting System) application accessed via either the CTEP web site (<a href="https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613">https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613</a>).

#### 7.16.1 Adverse Events (AEs)

**Definition of an AE**: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product (attribution of unrelated, unlikely, possible, probable, or definite). (International Conference on Harmonisation [ICH], E2A, E6). [CTEP, NCI Guidelines: Adverse Event Reporting Requirements. February 29, 2012;

http://ctep.cancer.gov/protocolDevelopment/electronic applications/adverse events.htm]

7.16.2 Serious Adverse Events (SAEs) — Serious adverse events (SAEs) that meet expedited reporting criteria defined in the table in Section 7.17 will be reported via CTEP-AERS. SAEs that require 24 hour CTEP-AERS notification are defined in the expedited reporting table in Section 7.17. Contact the CTEP-AERS Help Desk if assistance is required.

**Definition of an SAE**: Any adverse drug event (experience) occurring at any dose that results in any of the following outcomes:

- Death:
- A life-threatening adverse drug experience;
- Inpatient hospitalization or prolongation of existing hospitalization;
- A persistent or significant disability/incapacity;
- A congenital anomaly/birth defect.
- Important medical events that may not result in death, be life threatening, or require hospitalization may be considered an SAE, when, based upon medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in the definition.

Due to the risk of intrauterine exposure of a fetus to potentially teratogenic agents, the pregnancy of a study participant, including a male patient's impregnation of his partner, must be reported via CTEP-AERS in an expedited manner.

#### **7.16.3** Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)

AML or MDS that is diagnosed as a secondary malignancy during or subsequent to treatment in patients on NCI/CTEP-sponsored clinical trials must be reported via the CTEP-AERS system within 30 days of AML/MDS diagnosis.

#### Secondary Malignancy

A secondary malignancy is a cancer caused by treatment for a previous malignancy (e.g., treatment with investigational agent/intervention, radiation or chemotherapy). A secondary malignancy is not considered a metastasis of the initial neoplasm.

CTEP requires all secondary malignancies that occur following treatment with an agent under an NCI IND/IDE be reported via CTEP-AERS. Three options are available to describe the event:

- Leukemia secondary to oncology chemotherapy (e.g., acute myelocytic leukemia [AML])
- Myelodysplastic syndrome (MDS)
- Treatment-related secondary malignancy

Any malignancy possibly related to cancer treatment (including AML/MDS) also should be reported via the routine reporting mechanisms outlined in each protocol.

# Second Malignancy

A second malignancy is one unrelated to the treatment of a prior malignancy (and is NOT a metastasis from the initial malignancy). Second malignancies require ONLY routine reporting via CDUS unless otherwise specified.

# 7.17 CTEP-AERS Adverse Event Reporting Requirements (4/16/14)

All serious adverse events that meet expedited reporting criteria defined in the reporting table below will be reported via CTEP-AERS, the CTEP Adverse Event Reporting System, accessed via the CTEP web site, <a href="https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613">https://eapps-ctep.nci.nih.gov/ctepaers/pages/task?rand=1390853489613</a>.

Submitting a report via CTEP-AERS serves as notification to NRG Oncology and satisfies NRG Oncology requirements for expedited adverse event reporting.

CTEP-AERS provides a radiation therapy-only pathway for events experienced that involve radiation therapy only. These events must be reported via the CTEP-AERS radiation therapy-only pathway.

In the rare event when Internet connectivity is disrupted, a 24-hour notification must be made to the NRG Oncology Office at 1-800-227-5463, ext. 4189, for instances when Internet fails. Once internet connectivity is restored, an AE report submitted by phone must be entered electronically into CTEP-AERS.

- CTEP-AERS 24-Hour Notification requires that a CTEP-AERS 24-hour notification is
  electronically submitted within 24 hours of learning of the adverse event. Each CTEP-AERS
  24-hour notification must be followed by a CTEP-AERS 5 Calendar Day Report. Serious
  adverse events that require 24 hour CTEP-AERS notification are defined in the expedited
  reporting table below.
- Supporting source document is not mandatory. However, if the CTEP-AERS report indicates
  in the Additional Information section that source documentation will be provided, then it is
  expected. If supporting source documentation accompanies an CTEP-AERS report, include
  the protocol number, patient ID number, and CTEP-AERS ticket number on each page, and
  fax supporting documentation to the NRG Oncology dedicated SAE FAX, 215-717-0990.
- A serious adverse event that meets expedited reporting criteria outlined in the following table
  but is assessed by the CTEP-AERS System as "expedited reporting NOT required" must still
  be reported to fulfill NRG Oncology safety reporting obligations. Sites must bypass the "NOT
  Required" assessment; the CTEP-AERS System allows submission of all reports regardless
  of the results of the assessment.

CTEP defines expedited AE reporting requirements for phase 3 trials as described in the table below. **Important:** All AEs reported via CTEP-AERS also must be reported on the AE section of the appropriate case report form (see <u>Section 12.1</u>).

Late Phase 2 and Phase 3 Studies: Expedited Reporting Requirements for Adverse Events that Occur on Studies under an IND/IDE within 30 Days of the Last Administration of the Investigational Agent/Intervention<sup>1, 2</sup>

#### FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

**NOTE:** Investigators <u>MUST</u> immediately report to the sponsor (NCI) <u>ANY</u> Serious Adverse Events, whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64)

An adverse event is considered serious if it results in ANY of the following outcomes:

- 1) Death
- 2) A life-threatening adverse event
- An adverse event that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) A congenital anomaly/birth defect.
- Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

<u>ALL SERIOUS</u> adverse events that meet the above criteria <u>MUST</u> be immediately reported to the NCI via CTEP-AERS within the timeframes detailed in the table below.

| Hospitalization | Grade 1<br>Timeframes | Grade 2<br>Timeframes | Grade 3 Timeframes | Grade 4 & 5<br>Timeframes |
|---|---|---|---|---|
| Resulting in<br>Hospitalization<br>≥ 24 hrs | | 10 Calendar Days | | 24-Hour 5 |
| Not resulting in<br>Hospitalization<br>≥ 24 hrs | Not r | required | 10 Calendar Days | Calendar Days |

**NOTE**: Protocol specific exceptions to expedited reporting of serious adverse events are found in the Specific Protocol Exceptions to Expedited Reporting (SPEER) portion of the CAEPR

# Expedited AE reporting timelines are defined as:

- "24-Hour; 5 Calendar Days" The AE must initially be reported via CTEP-AERS within 24 hours of learning of the AE, followed by a complete expedited report within 5 calendar days of the initial 24-hour report.
- "10 Calendar Days" A complete expedited report on the AE must be submitted within 10 calendar days of learning of the AE.

#### Expedited 24-hour notification followed by complete report within 5 calendar days for:

All Grade 4, and Grade 5 AEs

#### Expedited 10 calendar day reports for:

- Grade 2 adverse events resulting in hospitalization or prolongation of hospitalization
- · Grade 3 adverse events

Effective Date: May 5, 2011

# 8.0 SURGERY

Not applicable to this study

<sup>&</sup>lt;sup>1</sup>Serious adverse events that occur more than 30 days after the last administration of investigational agent/ intervention and have an attribution of possible, probable, or definite require reporting as follows:

<sup>&</sup>lt;sup>2</sup> For studies using PET or SPECT IND agents, the AE reporting period is limited to 10 radioactive half-lives, rounded UP to the nearest whole day, after the agent/intervention was last administered. Footnote "1" above applies after this reporting period.

#### 9.0 OTHER THERAPY

#### 9.1 Permitted Supportive Therapy

All supportive therapy for optimal medical care will be given during the study period at the discretion of the attending physician(s) within the parameters of the protocol and documented on each site's source documents as concomitant medication.

- **9.1.1** Anticonvulsants
- 9.1.2 Antiemetics
- 9.1.3 Anticoagulants
- 9.1.4 Antidiarrheals
- 9.1.5 Analgesics
- 9.1.6 Hematopoietic Growth Factors
- 9.1.7 Herbal products
- **9.1.8** Nutritional supplementation

#### 9.2 Non-permitted Supportive Therapy

Patients must be instructed not to take any medications, including over-the-counter products and vitamins, minerals and other dietary supplements, without first consulting with the investigator, as noted in <u>Section 7.7</u> above.

#### 10.0 TISSUE/SPECIMEN SUBMISSION

**NOTE:** Patients must be offered the opportunity to participate in the tissue/specimen submission component of the protocol. If the patient consents to participate in this component of the study, the site is required to submit the patient's specimens as specified below.

Sites are <u>not</u> permitted to delete the tissue/specimen submission component from the protocol or from the sample consent.

#### 10.1 Tissue/Specimen Submission

The NRG Oncology Biospecimen Bank at the University of California San Francisco acquires and maintains high quality specimens from NRG Oncology trials. Tissue from each block is preserved through careful block storage and processing. NRG Oncology encourages participants in protocol studies to consent to the banking of their tissue. The Biospecimen Bank provides tissue specimens to investigators for translational research studies. Translational research studies integrate the newest research findings into current protocols to investigate important biologic questions.

#### 10.2 Specimen Collection for Translational Research (Mandatory) (12/17/13)

For patients who have consented to participate in the tissue/blood component of the study (See sample consent).

#### 10.2.1 Specimen Submission

See Section 10.5 for the address information for sending specimens.

**10.2.2** Specimen Collection Summary for Translational Research (mandatory for all patients)

| Serum Specimens for Translational Research (mandatory for all patients) | | | |
|---|---|---|---|
| Specimens taken from patient: | Collected when: | Submitted as: | Shipped |
| SERUM for baseline and follow up Testosterone, processed as per local aboratory requirements | (1) Baseline/ pre-treatment: Within 21 days prior to treatment | Testing performed on site at local laboratory | Not applicable |
| Note: Collect restosterone in the a.m. at same time of day as collection of Fasting nsulin/Fasting Glucose/ Fasting Lipids/ Hemoglobin A1C | (2) At 30 months (3) Follow Up: Every 12 months for 3 years | | |

| SERUM for Testosterone (LC/MS/MS): 5 mL (no-additive redtop), processed as detailed in Appendix V Note: Collect testosterone in the a.m. at same time of day as collection of Fasting Insulin/Fasting Glucose/Fasting Lipids/Hemoglobin A1C | (a) At 12 months<br>(b) At 24 months | Frozen serum samples containing 0.5 mL per aliquot in 1 mL cryovials (five to ten) | Serum sent frozen on<br>dry ice via overnight<br>carrier to the NRG<br>Oncology<br>Biospecimen Bank |
|---|---|---|---|
| SERUM for Fasting Insulin: 5 mL (no-additive red- top), processed as detailed in Appendix V Note: Collect in the a.m. at same time of day as testosterone | (1) Baseline/ pre-treatment: Within 21 days prior to registration (2) During ADT: (a) At 12 months (b) At 24 months (3) Follow Up: Every 12 months for 3 years | Frozen serum samples containing <u>0.5 mL</u> per aliquot in 1 mL cryovials (five to ten) | Serum sent frozen on<br>dry ice via overnight<br>carrier to the NRG<br>Oncology<br>Biospecimen Bank |
| SERUM for Fasting Glucose/Fasting Lipids/Hemoglobin A1C, processed as per local laboratory requirements Note: Collect in the a.m. at same time of day as testosterone | (1) Baseline/ pre-treatment: Within 21 days prior to registration 2) During ADT: (a) At 12 months (b) At 24 months (3) Follow Up: Every 12 months for 3 years | Testing performed on site at local laboratory | Not applicable |

# 10.3 Specimen Collection for Tissue Banking and Translational Research (Strongly Recommended) (12Jun2018)

For patients who have consented to participate in the tissue/blood component of the study (See sample consent). Note: Plasma and whole blood collection is mandatory for patients participating in quality of life [QOL].

The following must be provided in order for the case to be evaluable for the NRG Oncology Biospecimen Bank:

- **10.3.1** One H&E stained slide (slide can be a duplicate cut stained H&E of the diagnostic slide (block); it does not have to be the diagnostic slide itself)
- 10.3.2 A corresponding paraffin-embedded tissue block of the tumor (the block must match the H&E being submitted) or 10-15 unstained sections cut onto positive charged slides from the tumor tissue block (must be from same block as H&E). Block or slides must be clearly labeled with the pathology identification number and block # that corresponds to the Pathology Report.
- **10.3.3** A Pathology Report documenting that the submitted block or slides contains tumor. The report must include the RTOG (NRG) protocol number and patient's case number. The patient's name and/or other identifying information should be removed from the report. The surgical pathology numbers and information must NOT be removed from the report.

- The submitted material must be from malignant tumor, not necrotic or fibrotic tissue. If the submitted material is reviewed and is not tumor, the site may be assessed a protocol violation.
- **10.3.4** A Specimen Transmittal Form clearly stating that tissue is being submitted for the NRG Oncology Biospecimen Bank; if for translational research, this should be stated on the form. The form must include the RTOG (NRG) protocol number and patient's case number.

# **10.3.5** Specimen Collection Summary for Tissue Banking and Translational Research (strongly recommended)

| Specimens for Tissue Banking and Translational Research (strongly recommended) *Note: Plasma and whole blood is mandatory for patients participating in QOL. | | | |
|---|---|---|---|
| Specimens taken from patient: | Collected when: | Submitted as: | Shipped: |
| Representative H&E stained slides of the primary tumor | Pre-treatment | H&E stained slide<br>Pre-treatment | Slide shipped ambient |
| A paraffin-embedded tissue block of the primary tumor taken before initiation of treatment or 10-15 unstained slides | Pre-treatment | Paraffin-embedded<br>tissue block or 15<br>unstained slides<br>(must match the H&E<br>slide being submitted) | Block or slides shipped ambient |
| PLASMA*: 5-10 mL of anticoagulated whole blood in EDTA tube #1 (purple/ lavender top) and centrifuge [For inflammatory cytokines and markers including CRP, NF- kappa B, TNF alpha, IL- 1, IL-1ra, sTNFR2, and IL-6] | (1) Pre-treatment (2) 1 year (12 months) after therapy starts (3) 2.5 years (30 months) after therapy starts | Frozen plasma<br>samples containing<br>0.5 mL per aliquot in 1<br>mL cryovials (five to<br>ten) | Plasma sent frozen on<br>dry ice via overnight<br>carrier to the NRG<br>Oncology Biospecimen<br>Bank |
| WHOLE BLOOD* for DNA: 5-10 mL of anticoagulated whole blood in EDTA tube #2 (purple/ lavender top) and mix [For SNPs and CNVs in TNFAIP1, IL6, IL6R, CRP, IL1R1, IL1A, IL1B] | Pre-treatment Note: If site missed this collection time point they may collect this specimen at any other time point instead but must note this on the Specimen Transmittal Form. | Frozen whole blood samples containing 1 mL in 1mL cryovials (three to five) | Whole blood sent<br>frozen on dry ice via<br>overnight carrier to the<br>NRG Oncology<br>Biospecimen Bank |
| PBMCs: 5-10ml of whole blood in EDTA purple/lavender top tube (tube #3). See Appendix VI for processing instructions. [For NF Kappa B] | (1) Pre-treatment (2) 1 year (12 months) after therapy starts (3) 2.5 years (30 months) after therapy starts | Frozen PBMC samples (one to two). See Appendix VI for study-specific processing instructions. | PBMC sent frozen on<br>dry ice via overnight<br>courier to the NRG<br>Oncology Biospecimen<br>Bank |

10.3.6 See Appendix V for the specimen collection kit and detailed collection instructions. See Appendix VI for detailed PBMC collection, processing, and shipping information. Note: Kits can be requested from the NRG Oncology Biospecimen Bank at NRGBB@ucsf.edu. Please include in the e-mail if you are requesting the complete kit or the kit without the PBMC processing component. PBMC processing components will not be shipped to sites that are unable to follow the PBMC processing instruction. The following materials must be provided to the NRG Oncology Biospecimen Bank: A Specimen Transmittal Form documenting the date of collection of the biospecimen; the RTOG protocol number, the patient's case number, time point of study, and method of storage, for example, stored at -80° C, must be included.

#### **10.4** Storage Conditions (5/1/12)

Store frozen specimens at -80°C (-70°C to -90°C) until ready to ship. Frozen specimens can be stored -80°C (-70°C to -90°C) for up to six months before shipping. If a -80°C freezer is not available:

Samples can be stored short term in a -20° C freezer (non-frost free preferred) for <u>up to one week</u> (please ship out Monday-Wednesday only; Canada: Monday-Tuesday).

OR:

Samples can be stored in plenty of dry ice for <u>up to one week</u>, replenishing daily (ship out Monday-Wednesday only; Canada: Monday-Tuesday).

OR:

Samples can be stored in liquid nitrogen vapor phase (ship out Monday-Wednesday only; Canada: Monday-Tuesday).

Please indicate on the Specimen Transmittal Form the storage conditions used and time stored.

# For PBMC Specimens Only:

Store frozen specimens immediately at -80°C. Samples must then be kept at -80°C during storage and shipping (please ship out Monday-Wednesday only; Canada: Monday-Tuesday)

If a -80°C freezer is not available: Samples can be stored in plenty of dry ice for <u>up to one week</u>, replenishing daily (ship out Monday-Wednesday only; Canada: Monday-Tuesday).

Please indicate on the Specimen Transmittal Form the storage conditions used and time stored. **See**Appendix VI for detailed PBMC collection, processing, and shipping information.

10.5 Submit materials for Tissue Banking and Translational Research as follows: (12Jun2018)

U. S. Postal Service Mailing Address: <u>For Non-frozen Specimens Only</u> NRG Oncology Biospecimen Bank
University of California San Francisco – Box 1800
Campus Box 1800
2340 Sutter Street, Room S341
San Francisco, CA 94143

Courier Address (FedEx, UPS, etc.): <u>For Trackable FFPE and ALL Frozen Specimens</u> NRG Oncology Biospecimen Bank University of California San Francisco 2340 Sutter Street, Room S341 San Francisco, CA 94115

Questions: 415-476-7864/FAX 415-476-5271; NRGBB@ucsf.edu

#### **10.6** Reimbursement (4/16/14)

Please note that with the start of the new NCI National Clinical Trials Network (NCTN) Program, NCI funds for reimbursement for protocol-specified biospecimen materials will be distributed per the requirements/methods specified by the new NCTN Program. This information will be made available with the other registration materials in the Oncology Patient Enrollment Network (OPEN) portal system. OPEN

will serve as the registration system for all patient enrollments onto NCI-sponsored NCTN trials, including this study, which will be transitioned into the new Program from the NCI-sponsored Cooperative Group Clinical Trials Program.

#### 10.7 Confidentiality/Storage

(See the Patient Tissue Consent Frequently Asked Questions, <a href="http://www.rtog.org/Researchers/BiospecimenResource/BiospecimenResourceFAQs.aspx">http://www.rtog.org/Researchers/BiospecimenResource/BiospecimenResourceFAQs.aspx</a> for further details.)

- **10.7.1** Upon receipt, the specimen is labeled with the RTOG (NRG) protocol number and the patient's case number only. The NRG Oncology Biospecimen Bank database only includes the following information: the number of specimens received, the date the specimens were received, documentation of material sent to a qualified investigator, type of material sent, and the date the specimens were sent to the investigator. No clinical information is kept in the database.
- **10.7.2** Specimens for tissue banking will be stored for an indefinite period of time. Specimens for the translational research component of this protocol will be retained until the study is terminated, unless the patient has consented to storage for future studies. If at any time the patient withdraws consent to store and use specimens, the material will be returned to the institution that submitted it.

#### **11.0 PATIENT ASSESSMENTS** (12/17/13)

#### 11.1 Study Parameters

See <u>Appendix I</u> for assessments and timeframes. See <u>Sections 11.1.1</u> and <u>11.1.2</u> below for details and/or exceptions to Appendix I.

- **11.1.1** Chemistry and liver panels (sodium, potassium, chloride, bicarbonate (carbon dioxide), BUN, creatinine, glucose, calcium, magnesium, phosphorus, albumin, AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin) will be checked monthly during ADT until three consecutive normal potassium values have been obtained, then the chemistry and liver panels will be spaced to every 3 months.
- **11.1.2** Collect blood for testosterone in the morning at the same time of day as collection of blood for Fasting Insulin/Fasting Glucose/ Fasting Lipids/Hemoglobin A1C.

#### 11.2 PROMIS-Fatigue Short Form (12/17/13)

<u>Note</u>: Patients must be offered the opportunity to participate in the correlative components of the study, such as quality of life (QOL) assessment. Participation in QOL is optional, with a goal of enrolling 458 patients in the QOL study. There is additional case credit and financial reimbursement to the institutions for participating in the QOL studies to take into account the additional time, effort, and cost involved. In addition, patients participating in the QOL studies may not have started anti-androgen therapy (either LHRH therapy or oral anti-androgens) prior to completing the QOL forms and getting baseline blood collection. Thus, patients who have started LHRH therapy prior to enrollment will be excluded from participating in the QOL studies.

If the patient consents to participate in the QOL component of the study, sites are required to administer the PROMIS, EPIC-26, and the EQ-5D assessments at baseline and as specified in <a href="Appendix I">Appendix I</a> of the protocol. Sites are <a href="not">not</a> permitted to delete the QOL component from the protocol or from the sample consent. Blood collection is <a href="mailto:mandatory">mandatory</a> for patients participating in the QOL.

The PROMIS Fatigue Scale (7 items) was developed by the Patient-Reported Outcome Measurement Information System (PROMIS), part of the NIH Roadmap Initiative, focused on developing a publicly available resource of standardized, accurate, and efficient patient-reported outcome (PRO) measures of symptoms, distress, and functioning. Two content domains of fatigue, experience and impact, were identified by a panel of experts. An item pool of 58 fatigue experience and 54 fatigue impact items were developed. The psychometric properties of these items were evaluated in a sample of 450 individuals from the general US population using classical test theory indices, monotonicity, and scalability. The expert panel selected the 10 best items in each domain. These 20 items were presented to a panel of clinical experts. Only one item was dropped because of redundancy. A preliminary fatigue short-form measure of 7 items was created using items selected for consistency in the response scale, broad coverage across the fatigue continuum (i.e., high to low), and good precision of measurement (discrimination function).

The following items are being measured due to the fact that sleep quality and exercise are documented confounders of fatigue:

Muscle weakness question (scale of 1-5, from none to very much)
Overall Sleep Quality: Item from Pittsburgh Sleep Quality Index (Buysse 1989):
Sleep quality will be measured by 1 item (Q3) of the Pittsburgh Sleep Quality Index (PSQI), a self-rated questionnaire which measures sleep quality and disturbances over a 1-week or 1-month time period.

| | Very | Fairly | Fairly | Very |
|---|---|---|---|---|
| | bad | bad | good | good |
| 1. During the past week, how would you rate your sleep quality overall? | 0 | 1 | 2 | 3 |

Participants' level of physical activity will be assessed using the three item Godin Leisure-Time Exercise Questionnaire (GLTEQ) [Godin 1986; Gionet 1989], which measures time spent per week in each of light, moderate, and vigorous activities. A score can be computed for each level of exercise. A total score is computed by summing the three levels weighted by their respective MET equivalents of 3, 5, and 9. The GLTEQ has good test-retest reliability and has shown convergent validity with both objective and other self-report measures of physical activity (Godin 1986; Gionet 1989).

The following questions are about your average weekly exercise. When answering the questions only count exercise that you do during free time (ignore exercise associated with your occupation and housework). Considering a typical week (7 days), how many times, on average, do you perform mild, moderate, or strenuous exercise? And when you engage in exercise, how long do you exercise, on average?

| | Times<br>Per Week<br><b>(a)</b> | Average Duration (b) |
|---|---|---|
| <ol> <li>Mild exercise – that is, minimal effort exercise that did not make you<br/>perspire, such as easy walking, yoga, bowling, lawn bowling,<br/>shuffleboard, or golf</li> </ol> | | mins. |
| 2. Moderate exercise – that is, exercise that is not exhausting and which made you perspire lightly, such as fast walking, tennis, easy bicycling, easy swimming, or popular and folk dancing | | mins. |
| 3. Strenuous exercise – that is, exercise that made your heart beat rapidly and made you sweat, such as running, aerobics classes, cross country skiing, vigorous swimming, or vigorous bicycling | | mins. |

#### 11.3 Health Related Quality of Life (HRQOL) Assessments (12/17/13)

Note: Patients must be offered the opportunity to participate in the correlative components of the study, such as quality of life (QOL) assessment. Participation in QOL is optional, with a goal of enrolling 458 patients in the QOL study. There is additional case credit and financial reimbursement to the institutions for participating in the QOL studies to take into account the additional time, effort, and cost involved. In addition, patients participating in the QOL studies may not have started anti-androgen therapy (either LHRH therapy or oral anti-androgens) prior to completing the QOL forms and getting baseline blood collection. Thus, patients who have started LHRH therapy prior to enrollment will be excluded from participating in the QOL studies.

If the patient consents to participate in the QOL component of the study, sites are required to administer the PROMIS, EPIC-26, and the EQ-5D assessments at baseline and as specified in <a href="Appendix I">Appendix I</a> of the

protocol. Sites are <u>not</u> permitted to delete the QOL component from the protocol or from the sample consent. **Blood collection is mandatory for patients participating in QOL.** 

The following instruments will be used to assess health related quality of life (HRQOL), including quality adjusted survival: the Expanded Prostate Cancer Index (EPIC)-26, and the EuroQol (EQ-5D) instrument. These outcomes measurements will be administered to 458 patients (229 in each arm). Of note, these are essentially the same instruments (and similar time points) that are being studied in two related trials, RTOG 0815 and 0924, which are currently accruing patients. In RTOG 0815, patients with "lower" intermediate risk prostate cancer all receive high dose RT and are randomized to +/- short term hormones. In RTOG 0924, patients with intermediate to high risk prostate cancer are randomized to +/- whole pelvic RT and are stratified by short (6 months) or long term (32 months) ADT. Ultimately, use of essentially the same instruments and time points in all three studies (RTOG 0815, RTOG 0924, and RTOG 1115) will create a large database of relevant information related to QOL, QAS, and fatigue issues in prostate cancer patients that will facilitate a large combined analysis in the future. The outcomes instruments in this study are as follows:

#### 11.3.1 Prostate Cancer-Specific Health-Related Quality of Life: EPIC-26

The Expanded Prostate Cancer Index Composite (EPIC) is a prostate cancer health-related quality of life (HRQOL) patient self-administered instrument that measures a broad spectrum of urinary, bowel, sexual, and hormonal symptoms related to radiotherapy and hormonal therapy (van Andel 2003;Wei 2000). To minimize patient burden, the abbreviated, validated EPIC-26 will be used (Szymanski 2010).

#### 11.3.2 Quality-Adjusted Survival Analysis: EuroQol (EQ-5D)

The EQ-5D is a patient self-administrated questionnaire that takes approximately 5 minutes to complete (Schulz 2002). The first part consists of 5 items covering 5 dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension can be graded on 3 levels: 1-no problems, 2-moderate problems, and 3-extreme problems. Health states are defined by the combination of the leveled responses to the 5 dimensions, generating 243 (3<sup>5</sup>) health states to which unconsciousness and death are added (Badia 1998).

The 5-item index score is transformed into a utility score between 0, "Worst health state," and 1, "Best health state." The index score or the cost-utility equation can be used in the quality adjusted survival analysis depending on the health state(s) of interest (Wu 2002). For this study we plan to report the multidimensional utilities for comparative purposes. The EQ-5D has been used across numerous disease sites (Milne 2006; Wildi 2004) and has been used to assess quality adjusted survival of prostate cancer screening and treatment (Essink-Bok 1998; Sandblom 2004; Sennfalt 2004).

#### 11.4 Criteria for Discontinuation of Protocol Treatment (12/17/13)

- Progression of disease;
- If radiation therapy begins more than 240 days after initiation of ADT. If protocol treatment is discontinued, follow up and data collection will continue as specified in the protocol.

# **12.0 DATA COLLECTION** (12/17/13)

This study will utilize Medidata Rave® for remote data capture (RDC) of all data. Access to the trial in Rave is granted through the iMedidata application (https://login.imedidata.com) to all persons with the appropriate roles in RSS. To access iMedidata/Rave see Section 5.0.

Each person responsible for data entry must be on the NRG Oncology roster in order to receive access to Medidata Rave®.

Upon initial site registration approval for the study in RSS (Regulatory Support System), all CRAs at participating sites will receive e-mail invitations from iMedidata (iMedidata-Notification@mdsol.com) to activate their account. Once an account is activated, eLearning modules will be available for Rave RDC instructions. Site users must complete all modules before access to data entry in Rave is granted. Further training opportunities will be communicated through the web site.

Users that have not previously activated their iMedidata/Rave accounts will also receive a separate invitation from iMedidata to activate their account. Account activation instructions are located on the CTSU website, Rave tab under the Rave resource materials (Medidata Account Activation and Study

Invitation Acceptance). Additional information on iMedidata/Rave is available on the CTSU website under the Rave tab at <a href="www.ctsu.org/RAVE/">www.ctsu.org/RAVE/</a> or by contacting the CTSU Help Desk at 1-888-823-5923 or by e-mail at <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>.

#### **12.1** Summary of Data Submission (12/17/13)

Adverse event data collection and reporting, which are required as part of every clinical trial, are done to ensure the safety of patients enrolled in the studies as well as those who will enroll in future studies using similar agents. Adverse events are reported in a routine manner at scheduled times during the trial using Medidata Rave. Additionally, certain adverse events must be reported in an expedited manner for timely monitoring of patient safety and care. The following sections provide information about expedited reporting. For this trial the *Adverse Event* forms are used for routine AE reporting in Rave.

| <u>Folder</u> | <u>Form/Item</u> | <u>Due</u> |
|---|---|---|
| Registration via the OPEN System | Subject Enrollment Form (1) | At time of registration |
| Enrollment When pushed into RAVE there will be 5 forms representing registration | <ul> <li>Demography Form (2)</li> <li>Step Information Form (3)</li> <li>Treatment Assignment Form (4)</li> <li>Eligibility Checklist Form (5)</li> </ul> | |
| Concomitant Medications | | Review at baseline and<br>then every 3 months<br>during treatment (24<br>months) for changes (in<br>frequency, dose,<br>additional drugs or<br>discontinuation of drugs) |
| PSA Measurements | | All required measurements will be collected in this folder—every 3 months during treatment; then every 6 months for 3 years; then annuallythe follow up form will prompt reporting of these measurements |
| Quality of Life (Optional for patients not previously on LHRH or oral anti-androgens. A total of 458 patients may participate in the QOL studies; when QOL accrual achieved this folder will not be available for future patients) | <ul> <li>EQ-5D (QF)</li> <li>EPIC-26 (FA)</li> <li>PROMIS (HP)</li> <li>PSQI/GLTEQ (QL)</li> </ul> | Collected at 5 time points (only if answer to quality of life participation = yes at registration): 1) Prior to the start of protocol hormone treatment (baseline); 2) Prior to RT; 3) During the last week of RT; 4) At one year (12 months) after the start of protocol treatment; 5) At 2.5 years (30 months) after the start of |

| <u>Folder</u> | Form/Item | <u>Due</u> |
|---|---|---|
| | | protocol treatment |
| Baseline Folder | <ul> <li>Patient History Form (formerly known as the A5; voluntary form completed by the patient or with help from site staff or family)</li> <li>Work Up Form</li> <li>Diagnostic Staging Form</li> <li>Prior Treatment Form</li> <li>Pathology Report Form (a copy of this report will be scanned and uploaded into RAVE)</li> <li>Chemistry Panel Form</li> <li>Liver Panel Form</li> <li>Fasting Lipid Panel Form</li> <li>CBC w/Differential Form</li> <li>Hemoglobin A1C Form</li> <li>Serum Testosterone Form</li> </ul> | Within 2 weeks after registration |
| Month 1 visit | Chemistry Panel Form Liver Panel Form | After 30 days of<br>hormonal treatment/<br>registration to the trial<br>For relevant labs<br>necessary during<br>hormonal treatment +/-<br>TAK700 |
| Month 2 visit | Chemistry Panel Form Liver Panel Form | After 60 days of hormonal treatment/ registration to the trial For relevant labs necessary during hormonal treatment +/- TAK700 |
| Follow-Up Folders Month 3 Month 6 Month 9 Month 12 Month 15 Month 18 Month 21 Month 24 | <ul> <li>Follow up Form – if Patient Contacted = "yes"</li> <li>Primary Cause of Death Form – if Patient's Vital Status = 'dead'</li> <li>Disease Assessment Form – if Documented clinical assessment = 'yes'</li> <li>New Primary Cancer Form – if New Primary Cancer = 'yes'</li> <li>Non-protocol Treatment Form – if patient started on non-protocol cancer therapy = 'yes'</li> <li>Complete Appropriate Lab Form – if labs performed = 'yes' (chemistry and liver panel forms every 3</li> </ul> | Every 3 months from the start of treatment/ registration to the trial during years 1 and 2 (to capture hormone +/- TAK-700 administration); |

| <u>Folder</u> | <u>Form/Item</u> | <u>Due</u> |
|---|---|---|
| | months and at 12 and 24 month visits fasting lipid panel form and hemoglobin A1C form will be added) • PSA Measurement Form – if PSA assessed = 'yes' • Adverse Event Form – if new or continuing adverse events = 'yes' • Concomitant Medication Form if Changes in Medication = 'yes' | |
| Hormonal Treatment<br>with or without TAK-700 | <ul> <li>Oral Antiandrogen Form</li> <li>LHRH Agonist Form</li> <li>Agent TAK700 Form</li> </ul> | Every 3 months (from<br>the start of hormonal<br>therapy/registration to<br>the trial) for 2 years |
| <ul> <li>Month 30 Visit</li> <li>Marks the start of follow up without treatment</li> <li>Questions answered as 'yes' generate additional forms—similar to 'filter questions' being asked</li> <li>Month 36 Month 42 Month 48 Month 54 Month 60 </li> <li>Month 72</li> <li>Start of annual visits</li> </ul> | <ul> <li>Follow up Form – if Patient Contacted = "yes"</li> <li>Primary cause of death form – if Patient's Vital Status = 'dead'</li> <li>Disease Assessment Form – if Documented clinical assessment = 'yes'</li> <li>New Primary Cancer Form – if New Primary Cancer = 'yes'</li> <li>Non-protocol Treatment Form – if patient started on non-protocol cancer therapy = 'yes'</li> <li>Complete Appropriate Lab Form – if labs performed = 'yes' (at 36, 48 and 60 month visits a chemistry panel form for fasting glucose; fasting lipids form; testosterone form and hemoglobin A1C form)</li> <li>PSA Measurement Form – if PSA assessed = 'yes'</li> <li>Adverse Event Form – if new or continuing adverse events = 'yes'</li> </ul> | therapy/registration to |

# 12.2 Summary of Dosimetry Digital Data Submission (4/16/14) Note: Submit digital RT data to TRIAD; see Section 5.0 for account access and installation instructions.

| <u>Form/Item</u> | <u>Due</u> |
|---|---|
| Preliminary Dosimetry Information Digital Data Submission — Treatment Plan submitted to IROC Houston via TRIAD account exported from treatment planning machine by Physics staff Digital data submission includes the following: • CT data, critical normal structures, all GTV, CTV, and PTV contours • Digital beam geometry for initial, boost and composite beam sets • Doses for initial, boost and composite sets of concurrently treated beams • Digital DVH data for all required critical normal structures, GTV, CTV, and PTVs for total dose plan Digital Data Submission Information (DDSI) → Upload confirmation email that digital data was submitted | Within 1 week of RT end (external beam RT +/-brachytherapy) |
| Final Dosimetry Information RT Treatment form [for EBRT +/- brachytherapy] Daily Treatment Record Please note: Daily Treatment Record will be uploaded via Rave to IROC Philadelphia NOTE: All Simulation and Portal Images will be kept by the Institution and only submitted if requested. LDR Brachytherapy Post-implant evaluation CT scan Post-implant structure set Post-implant plan Post-implant dose distribution RTOG Prostate Brachytherapy Protocol Compliance Form-Available | If applicable: 3-5 weeks post implant—submit listed items to TRIAD If applicable: 3-5 weeks post implant—submit listed items to TRIAD |
| | Preliminary Dosimetry Information Digital Data Submission — Treatment Plan submitted to IROC Houston via TRIAD account exported from treatment planning machine by Physics staff Digital data submission includes the following: • CT data, critical normal structures, all GTV, CTV, and PTV contours • Digital beam geometry for initial, boost and composite beam sets • Doses for initial, boost and composite sets of concurrently treated beams • Digital DVH data for all required critical normal structures, GTV, CTV, and PTVs for total dose plan Digital Data Submission Information (DDSI) → Upload confirmation email that digital data was submitted Final Dosimetry Information RT Treatment form [for EBRT +/- brachytherapy] Daily Treatment Record Please note: Daily Treatment Record will be uploaded via Rave to IROC Philadelphia NOTE: All Simulation and Portal Images will be kept by the Institution and only submitted if requested. LDR Brachytherapy Post-implant evaluation CT scan Post-implant structure set Post-implant tose distribution RTOG Prostate Brachytherapy |

| <u>Folder</u> | <u>Form/Item</u> | <u>Due</u> |
|---|---|---|
| | HDR Brachytherapy Implant CT scan Implant structure set Implant plan Implant dose distribution RTOG Prostate Brachytherapy Protocol Compliance Form-Available on the RPC website, http://irochouston.mdanderson.org NOTE: Copies of simulation and port films/images will be submitted to IROC Philadelphia ONLY if specifically requested. | |

#### 13.0 STATISTICAL CONSIDERATIONS

- 13.1 Primary Endpoint
- **13.1.1** Overall Survival (failure: death due to any cause)
- **13.2** Secondary Endpoints (12Jun2018)
- **13.2.1** Incidence of unexpected grade ≥ 3 adverse events and/or clinically significant decrement in patient reported quality of life among subjects treated with TAK-700
- **13.2.2** Rates and cumulative incidence of biochemical control (freedom from PSA failure), local/regional progression, and distant metastases
  - Biochemical failure will be defined by the Phoenix definition (PSA ≥ 2 ng/ml over the nadir PSA, the presence of local, regional, or distant recurrence, or the initiation of salvage androgen deprivation therapy) [Roach 2006].
  - Local failure will be defined as biopsy proven recurrence within the prostate gland.
  - Regional or distant metastasis will be defined as imaging or biopsy demonstrated evidence for recurrence in the pelvic lymph nodes (regional) or systemically. Biopsy is not required to define regional or distant metastasis; however, in absence of a rising PSA biopsy is encouraged.
- 13.2.3 General clinical treatment failure free interval (general clinical treatment failure [GCTF] is defined as: PSA > 25 ng/ml, documented local disease progression, regional or distant metastasis, or initiation of androgen deprivation therapy). Deaths prior to any of these events are treated as censoring for this endpoint.
- **13.2.4** Prostate cancer specific survival (failure: death due to prostate cancer) and other-cause survival (failure: death due to other causes)
- 13.2.5 Change in fatigue from baseline to 1 year, as measured by PROMIS
- **13.2.6** Changes in patient reported quality of life as measured by Expanded Prostate Cancer Index Composite (EPIC)
- 13.2.7 Assessment of quality adjusted survival using the EQ-5D (Will not be completed and is not part of the revised quality of life substudy per Amendment 3.)
- **13.2.8** Nadir and average serum testosterone at 12 and 24 months during treatment
- **13.2.9** Lipid profiles at 12 and 24 months
- 13.2.10 Fasting plasma glucose, fasting plasma insulin, and hemoglobin A1c at 12 and 24 months
- **13.2.11** Changes in body mass index (BMI) during 24 months of treatment and during the first three years of follow-up
- 13.2.12 Incidence of adverse events ascertained via CTCAE version 4
- **13.2.13** Rate of recovery of testosterone to >230 ng/dL (accepted threshold for supplementation) after 12 and 24 months of follow-up
- 13.2.14 Median time to recovery of testosterone to >230 ng/dL during the first five years of follow-up

**13.2.15** Cumulative incidence of relevant clinical survivorship endpoints including new diagnosis of type 2 diabetes, coronary artery disease, myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis, or osteoporotic fracture

#### **13.3** Sample Size Determination (12/17/13) (12Jun2018)

#### **13.3.1** Sample Size for Primary Endpoint

Patients with disease characteristics meeting the eligibility criteria for this study (Section 3.0) historically have 5-year survival of 78% and 8-year survival of 61.5%. We assume an annual hazard rate of 0.055, and aim to detect a 33% reduction in failure rate for the experimental arm. Assuming a two-sided alpha level of 0.05 (adjusted for interim analysis, see below), observation of 239 events is required for 85% statistical power to detect this effect. This relative hazard reduction implies an absolute survival difference of 7% at five years.

It is anticipated that patients can be accrued to this study at a rate of 30 per month. If 870 patients are accrued over 29 months, then the requisite events for definitive analysis would be accumulated after an additional 67 months, or 96 months from commencement of accrual. To account for a potential ineligibility and follow-up loss rate of 3%, 900 patients will be enrolled.

#### **13.3.2** <u>Statistical Power for Other Time to Event Endpoints</u>

Patients in this risk class have biochemical failure rates of approximately 8% per year between years 5 and 8. The trial will provide for detection of a 30% relative reduction in biochemical failure rate with statistical power approaching 90% at eight years. The distant failure rate for these patients is 2.0% per year. A 50% relative reduction in hazard of distant metastases for the experimental treatment group can be detected with statistical power of 88% at eight years.

# 13.3.3 <u>Statistical Power for Primary Survivorship Endpoints</u>

Hemoglobin A1c will be measured at baseline, 12 months and 24 months, with scores reflecting change from baseline compared at the follow-up time-points. A 0.1% difference in A1c between treatments would be considered of clinical interest. Given the precision of measurement in HB A1c in prior studies involving men receiving GnRH therapy (mean to standard error ratio greater than 10), power for detection of such differences would easily exceed 90%, even after controlling for multiple comparisons.

For diabetes/pre-diabetes incidence, the standard treatment frequency is expected to be in the range of 12-15%. Odds ratios of 1.5 or greater for the TAK-700 group will be detectable with power exceeding 80%.

#### 13.3.4 Statistical Power for Primary Quality of Life Endpoint

It is not anticipated that the entire trial participant cohort will be enrolled in the QOL correlative study. However, it is of interest to establish whether the addition of TAK-700 contributes to diminished quality of life scores and increased fatigue, and thus is desirable to have a sufficient sample to rule out smaller differences that would be considered clinically material. Fatigue, as measured by the PROMIS, will be the primary QOL analysis and therefore will be used in the sample size calculation. If we consider a 0.33 standard deviation effect size and a two-sided type I error = 0.05, we obtain a required sample size of 390 patients (195 patients per arm) for 90% power. To account for losses, such as ineligibility and non-compliance, 15% inflation in sample size is applied, resulting in 458 patients. A total of 458 patients enrolled in the study will participate in the QOL portion of the trial.

The study closed to accrual with 239 patients enrolled. Given this enrollment, it is assumed that there will be 130 patients evaluable at 1 year, with those not evaluable due to ineligibility, non-compliance and not consenting to this correlative study. With this sample size, a moderate effect size of 0.5 can be detected with 81% power using a two-sample test of the difference in means with a two-sided type I error = 0.05.

#### **13.3.5** Software for Sample Size Calculations

For the above calculations, the statistical software package EAST was used. Additional calculations verifying study duration and power for time to event endpoints were performed with user-written programs in the SAS statistical language.

#### 13.4 Randomization

Patients will be stratified before randomization by the composite risk score (based on Gleason score, PSA, and tumor stage) defined in <u>Section 3.1.1</u>, type of RT boost, and use of ADT prior to registration. Treatment arms will be balanced with respect to risk score via a permuted block procedure (Zelen 1974).

#### **13.5** Analysis Plan (12Jun2018)

#### 13.5.1 Primary Efficacy Endpoint

Primary analysis will include all eligible randomized patients with follow-up information, with patients included in the group to which they were assigned, regardless of whether they started treatment. Overall survival will be compared between treatment arms using the log-rank test (Mantel 1966). The Kaplan-Meier estimator will be used to estimate overall survival by treatment group (Kaplan 1958). Event times are measured from the date of study registration to the date of failure, or last follow up.

#### 13.5.2 Other Efficacy Endpoints

Cumulative probability over time of PSA failure, local/regional recurrence, distant metastases and clinical failure will be estimated via the cumulative incidence function, which correctly accounts for competing risks (Korn 1992). Primary putative treatment effect comparisons for these endpoints will be based on cause-specific hazards using logrank tests (Friedlin 2005, Dignam 2008). To evaluate differences specifically in cumulative incidence of these events, we may also employ Gray's test (Gray 1988).

If there are imbalances in covariates by treatment arm, then hazard regression models will be used to produce adjusted treatment effect estimates and tests. Appropriate models will be applied based on which metric is being examined (cause-specific hazard or cumulative incidence) [Prentice 1978, Fine 1999]. If model-specific assumptions are not met (for example, proportionality), then alternative approaches will be sought.

# 13.5.3 Longitudinal Quality of Life (QOL) and Patient Reported Outcome (PRO) Endpoints

The primary hypothesis of the QOL endpoints are that QOL and fatigue scores will not differ significantly between the control group and the experimental group receiving both a GnRH agonist and TAK-700. Quality of life will be measured with the prostate cancer-focused 32-question EPIC (The Expanded Prostate Cancer Index Composite) questionnaire and by the 5-question EQ-5D global quality of life assessment. Fatigue will be measured by the 7-question PROMIS (Patient-Reported Outcome Measurement Information System) fatigue short form questionnaire. The EPIC-26, PROMIS-fatigue short form, and EQ-5D will be collected at pretreatment (baseline), the week prior to starting RT, the last week of RT, and 1 year and 2.5 years after initiation of therapy.

The primary objective in the fatigue analysis is to determine the QOL differences at 1 year. The response will be the change of measurement from baseline for each measurement. Using the sample size specified in section 13.3.3 of 130 evaluable patients, we will have 64% statistical power assuming a type I error = 0.05 (with appropriate type I error control for multiplicity using the Bonferroni correction) to detect a standard deviation effect size of 0.5 between the treatment arms for the 4 domains of the EPIC.

For these investigations, a longitudinal analysis will be conducted that will focus on patterns of scores over time points (baseline, the week prior to starting RT, the last week of RT, and 1 year and 2.5 years after initiation of therapy) for the QOL and PRO instruments (EPIC, PROMIS and EQ-5D). Following descriptive statistics on assessments and tests of the primary endpoint of change from baseline to 1 year, repeated measures analysis of covariance (ANCOVA) will be used on scores for the assessment measures, where time points are considered the within-patient factor and treatment groups is considered the between-patient factor (Diggle 1994). While scales for the individual instrument questions are quantitative, they represent ordinal values on a bounded range rather than continuous quantities. Nonetheless, in aggregate these approximate continuous distributions, and appropriate transforms will be applied to improve consistency with model assumptions. The hierarchical analytic approach described below permits tests of omnibus hypotheses that control for multiple comparisons among time points and treatment groups. The analysis will be conducted as follows:

- The ANCOVA model will be used to carry out an omnibus test of the hypothesis that there is a common mean score across time point within the treatment groups:  $H_0$ :  $\mu_{it} = \mu_{i.}$ , where i = t treatment group 1 or 2, t = t time point (baseline, the week prior to starting RT, the last week of RT, 1 year and 2.5 years) and  $\mu_{it}$  is the mean score in treatment group i at time t.
- (2) If the hypothesis in (1) is rejected, individual comparisons of the post-RT and subsequent scores will be conducted within treatment groups. Additional modeling and graphical methods to determine trends or patterns of change in scores over time points will be conducted.

- (3) The ANCOVA model will be used to carry out an omnibus test of the hypothesis that there is a common mean score at each time point among the treatments:  $H_0$ :  $\mu_{it} = \mu_{.t}$ , where again  $\mu_{it}$  is the mean score in treatment group i at time t.
- (4) Assuming the result of the hypothesis test in (3) is significant (H<sub>0</sub> rejected), individual tests will be carried out to determine differences between treatment groups at specific time points. If there are no significant treatment differences identified in (3), an overall test of trend in scores can be aggregated over treatment groups. Additional modeling to characterize patterns of change over time will be conducted.

Information regarding potential confounds will be collected in a short form (QL) using limited questions to minimize patient burden. This information can be used to evaluate the potential impact of these confounding factors on fatigue. Patient responses to the following will be collected in the QL form: muscle weakness (one item), overall sleep quality as measured by one item from the Pittsburgh Sleep Quality Index (PSQI) [Buysse 1989] and level of physical activity as measured by the Godin Leisure-Time Exercise Questionnaire (GLTEQ) (Godin 1986; Gionet 1989). Anxiety/depression is also a potential confound with fatigue and patient responses to the anxiety/depression item in the EQ-5D can be used. At the same time points, the QL form (i.e., one item from the PSQI, 3 items from the GLTEQ, and one question regarding general muscle weakness) will be collected. In addition, in order to correlate fatigue with the cytokine changes, the PROMIS-fatigue short form (and the associated questions) will be collected at the following time points: at baseline, the week prior to starting RT, the last week of RT, 1 year and 2.5 years after therapy starts.

These confounding factors may be incorporated into the above hypothesis tests via the ANCOVA model. The effects of these covariates on scores may also be evaluated separately in exploratory analyses. Also note that baseline scores will be analyzed in relation to subsequent impairment or decline for both treatment groups (hypothesis (1) above). The use of change scores (relative to baseline) for the main analysis also may be explored to account for the influence of per patient conditions prior to undergoing treatment.

A certain degree of attrition from the study, due to both patient withdrawal and mortality, is expected. Characteristics of patients with missing data will be evaluated to identify imbalance in factors such as treatment, baseline scores, and other clinical and demographic features. In the absence of apparent systematic missing data patterns, data will be analyzed assuming that the observations are missing at random, employing appropriate methodology for this purpose (Little 1992). In the case of evidence for systematic patterns of missing data ('informative' missingness), alternative strategies for analyzing such data, depending on the pattern (e.g., intermittent versus complete dropout pattern) will be investigated (Wu 1988, Little 1992).

In this study, the addition of TAK-700 is hypothesized to improve overall survival (OS), without having a significant a negative impact on health related quality of life (HRQOL). As there are competing pros and cons of this treatment, it is useful to combine these factors into one equation to determine whether the potential benefits of this treatment (dose-escalated RT combined with short-term androgen deprivation), in terms of OS, outweigh the potential risks, in terms of negatively impacting on global HRQOL, compared to RT and ADT alone. Such a quality adjusted survival analysis can be invaluable for assisting in the decisions of future patients as well as clinicians faced with these treatment options.

Quality-adjusted survival can be defined by the weighted sum of different time episodes added up to a total quality-adjusted life-year [U= sum of quality (qi) of health states K times the duration (si) spent in each health state] (Glasziou 1990):

$$U = \sum_{i=1}^{K} q_i s_i$$

We will use Glasziou's multiple health-state (Q-TwiST) models to use the repeated measures of EQ-5D. Because Glasziou's method incorporates longitudinal QOL data into an analysis of quality-adjusted survival, the health stated model must be constructed on the following assumptions:

- A1) QOL is independent from treatment.
- A2) A health state is independent from previous states.
- A3) Proportionality of quality-adjusted duration and duration of the actual state of health

Assumption A1 can be checked by plotting QOL over time according to treatment, and the t-test can be used to compare the mean QOL scores of each treatment arm. Assumption A2 can be checked by comparing the QOL for patient groups in a given health state where the groups are defined by duration of previous health state experience using a regression model. Suitable checks for assumption A3 at minimum would be a simple plot. If data does not support these assumptions, we will use a method which uses the longitudinal QOL data directly. We will use the 5-item utility score in EQ-5D for the cost-utility analysis. We will use the Z-test to test the hypothesis that the cost-utility in the 2 treatment arms is the same at 1 year after initiation of treatment with a significance level of 0.05 and a 2-sided test. The remaining timepoints in which the EQ-5D is collected will also be assessed using similar longitudinal analysis techniques as described for the primary endpoint.

#### 13.5.4 Testosterone Kinetics

Comparison of testosterone levels at designated time points will be conducted via t-tests on baseline-corrected and appropriately transformed measurement values. Nonparametric tests to compare medians may also be conducted.

Time to recovery of testosterone to >230 ng/dL (accepted threshold for supplementation) after treatment will be estimated using time to event data methods. Specifically, the cumulative incidence of >230 ng/dL level achievement will be computed, accounting for competing events in the form of 1) interventions due to clinical failure that may suppress recovery and 2) deaths.

#### **13.5.5** Lipid Profiles, Glycemic Parameters, and Body Mass Index

Comparison of baseline-adjusted values for fasting glucose, fasting insulin, lipid levels, and hemoglobin A1c will be carried out between treatment groups at designated time points. Additionally, longitudinal models as described above may be used to characterize changes in these parameters over time within and between treatment groups. Body mass index will similarly be contrasted at specific time points and modeled as a function of time from treatment initiation.

#### **13.5.6** Clinical Survivorship Endpoints

Incidence rates (events/person years of exposure) and cumulative incidence over time of specific clinical events (type 2 diabetes, coronary artery disease, myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis, osteoporotic fracture) will be estimated by treatment arm. Poisson regression or other appropriate methods will be used to investigate the role of other explanatory risk factors in conjunction with treatment exposure.

#### 13.5.7 Trial Monitoring

#### Data Monitoring Committee

Phase III trials are required by NCI Cooperative Group Program Guidelines to be reviewed by a Data and Safety Monitoring Committee (DSMC). This study will be reviewed by the NRG Oncology Data Monitoring Committee (DMC) on a semi-annual basis.

This study will be monitored by the Clinical Data Update System (CDUS) version 3.0 (CDUS Abbreviated). Cumulative CDUS data will be submitted quarterly by electronic means. Reports are due January 31, April 30, July 31, and October 31.

# Interim Efficacy and Futility Analysis Plan

There will be three interim analyses of the primary hypotheses, at equally spaced increments of 25%, 50%, and 75% of the requisite events for definitive analysis. A conservative upper superiority bound, based on a Lan-DeMets approximation to the O'Brien and Fleming boundary (DeMets 1994) provides test criteria of Z > 4.33 at the first interim analysis, Z > 2.96 at the second interim analysis, and Z > 2.36 at the third interim analysis. At the final analysis, a test statistic of Z > 2.01 will be required to reject  $H_0$ .

Interim futility analysis will be based on the rule of Freidlin, Korn, and Gray (Freidlin 2010). This rule provides the opportunity to terminate early for evidence that the experimental arm will not prove superior, but protects against aggressive early termination for treatment effect sizes smaller than planned.

The following table summarizes the interim efficacy/futility monitoring schedule with respect to the primary endpoint:

| Analysis | Time<br>(month) | Prop. Cumulative Efficacy Total Total Events boundary | | | | _ | | boundary |
|---|---|---|---|---|---|---|---|---|
| | | events | (Both Arms) | Z> | P< | Z< | P> | |
| Interim 1 | 33 | 0.25 | 60 | 4.33 | 0.00001 | -1.64* | 0.05* | |
| Interim 2 | 54 | 0.50 | 120 | 2.96 | 0.0015 | 0.06 | 0.476 | |
| Interim 3 | 75 | 0.75 | 180 | 2.36 | 0.009 | 0.31 | 0.378 | |
| final | 96 | 1.00 | 239 | 2.01 | 0.022 | - | - | |

<sup>\*</sup> Early look for detriment in experimental arm, left-tail p < 0.05 will prompt stopping

In addition to the futility boundary for the primary endpoint, we will also implement a futility rule based on an intermediate endpoint for which evidence of efficacy is expected if there is eventual efficacy on the primary endpoint. Specifically, hormone deprivation agents that have shown favorable survival benefit typically demonstrate reductions in clinical outcomes such as time free from PSA progression or clinical failure (local, regional, or distant disease progression). Thus, early evidence of activity will be assessed by comparing the rate of general clinical treatment failure (GCTF, defined as time to any of the following events: PSA failure, local/regional recurrence, distant recurrence, hormone initiation) between treatment groups. The approach will involve testing for a difference in GCTF with adequately high power but a rather less stringent alpha level, following the strategy in multi-arm multi-stage clinical trials, where regimens are evaluated early based on intermediate endpoints to assure some level of activity before continuing to definitive endpoints (Sydes 2009).

Assuming an annual GCTF hazard rate of 0.125, a one-sided alpha of 0.10 and statistical power of 0.90, detection of a 40% reduction in GCTF hazard for patients receiving TAK-700 requires observation of 100 events. Because the most frequent GCTF event is PSA failure, and this event is delayed during active treatment, analysis will take place only on the cohort of patients consisting of those entering through the first 1.5 years (450 patients). This cohort will be observed for an additional 1.75 years, or to approximately 3.25 years from commencement of accrual, when the requisite number events for the above comparison will have been observed. At this time, GCTF will be compared between treatments, and if the null hypothesis of no difference in GCTF rate cannot be rejected in favor of a lower GCTF rate for patients receiving TAK-700 (one-sided 0.10 test), then discontinuation of the trial for futility will be considered. Within the time frame described above, there will be at least 80% power for any treatment difference equal to or greater than a 33% relative reduction in GCTF events. Results of this analysis will be reported only to the RTOG Data Monitoring Committee and not in any scientific forum or publication.

#### Interim Safety Analysis Plan

After the accrual and follow-up of 100 patients per treatment arm through completion of six months of therapy, adverse event (CTCAE) frequencies will be formally compared between treatment arms.

Analysis will focus on specific organ system class and specific adverse event types, in addition to frequency of grade 3 and higher adverse events overall (i.e., any type). Adverse events of interest are shown below, accompanied by expected frequencies for the control arm of this trial, based on observed rates in previous RTOG prostate cancer trials using prolonged androgen suppression.

| CTCAE (4.0) category | CTCAE specific | Expected % grade ≥3 or greater on standard ADT |
|---|---|---|
| Any | Any | 22.0 |
| Renal and urinary disorders | Any | 3.0 |
| Gastrointestinal disorders | Any | 3.6 |
| Reproductive system and | Any | 10.4 |
| breast disorders | | |
| General disorders and | Fatigue | 1.9 |
| administration site conditions | | |
| Vascular disorders | Hypertension | 0.0 |
| Metabolism and nutrition disorders | Hypokalemia | 0.0 |

Frequencies will be compared between treatment arms via Fisher's exact test. A one-sided criterion will be used to determine whether there is higher frequency of a given adverse event in the ADT+TAK700 arm. Including 200 patients with six months of follow-up (100 in each treatment group) and using a one-sided 0.01 alpha level, a 15% absolute increase in event types with expected frequency < 4% under standard ADT (for example, GU, GI, fatigue) can be detected with statistical power of 85% or greater. For those events with expected frequency in the range of 10%-25% in the control arm, statistical power for detecting a 25% absolute increase exceeds 85%. If there are imbalances between treatments in patient demographic or radiation treatment parameters that may affect adverse event rates, then stratification or modeling methods will be used.

In addition, scores for EPIC, EQ-5D, and PROMIS in this cohort will be compared between treatment groups, using the scheduled post-RT assessment. Differences will be assessed via t-tests on suitably transformed score sums, corrected for baseline values. A formal stopping criterion for these scores will not be specified.

# 13.5.8 Trial Reporting

The primary trial endpoint will be reported when specific criteria described in <u>Section 13.5.7</u> are met. In particular, when either the number of events for definitive analysis is reached or an interim analysis indicates that early stopping is warranted, then the primary endpoint will be considered eligible for reporting.

#### **13.5.9** Revised Sample Size, Statistical Power, and Analysis Plan

In June 2014, Millennium Pharmaceuticals informed NRG Oncology of their intention to no longer pursue development of the experimental agent (TAK-700) in prostate cancer. Subsequent discussion established that patients having entered the trial as of the accrual closure date would be provided assigned therapy to complete the regimen as described in 7.1.2. At trial accrual closure (September 30, 2014), 239 patients had been enrolled.

Statistical power for the primary and secondary endpoints will thus be compromised regardless of the length of follow-up time, and thus in order to frame completion of primary analysis that is practical with respect to time to reporting, a plan for seeking to obtain suitably reliable information on the effects of the intervention on PSA failure was developed, with a goal of reporting on the trial after 5 additional years of follow-up from accrual closure.

The assumed rate of PSA failure for the control arm is .08/year. With 239 patients accrued over 28 months (assuming 230 eligible and analyzed), additional follow-up (from September 2014) of 5 years will yield the following (based on projections computed as in Rubinstein, Gail, and Santner (1981)).

| | TAK- | TAK-700 Treatment Effect | |
|---|---|---|---|
| | HR 0.60 | HR 0.60 HR 0.55 HR 0.50 | |
| TAK-700 group failure rate | 0.048 | 0.044 | 0.040 |
| Number of events at 5 years | 70 67 65 | | |
| Power at 5 years* | 0.68 | 0.78 | 0.86 |

<sup>\*</sup> at one-sided alpha = 0.05

The PSA failure endpoint will be analyzed when 70 events have been observed, which is expected to occur relatively close to 5 years under any of these scenarios. If the relative reduction exceeds 40%, then power will be greater than 70% (at one-sided alpha = 0.05). For this number of events, if the relative reduction is 45%, power will reach 80%, and will reach 90% for a 50% reduction in PSA failure rate.

For the original primary endpoint (OS) and other secondary time to event endpoints, statistical power at the expected time of this first report is as follows. At the assumed failure rates, power for the originally planned detection of a 33% reduction in hazard of death would be approximately 28% (at two-sided alpha = 0.05). For distant metastasis, power to detect a 50% failure rate reduction would be approximately 32%.

At the time when PSA failure results are reported based on reaching the above criterion, these other endpoints will be reported. Confidence bounds will be provided for hazard ratio estimates and estimated percent event-free at specific time points, in order to illustrate the degree of uncertainty in these endpoints for which statistical power is less than desired. It will be determined at that time whether further (long-term) follow-up would be sufficiently informative towards evaluating the effect of experimental treatment

on these endpoints. At this time, it is not anticipated that a longer duration of follow-up would materially improve power or precision on estimates, given the low event rates for these endpoints.

#### 13.5.10 Revised Trial Monitoring Plan

Given the curtailed sample size and plan to report results when PSA failure data is mature, the interim monitoring plan will be revised. The trial will be evaluated for futility after one-half of the target of 70 events is observed. Efficacy will also be evaluated using an extreme boundary (consistent with an approximate 67% reduction in hazard), with the rationale being that early stopping for efficacy given the suboptimal sample size should only be considered in extraordinary circumstances.

The following table summarizes the interim efficacy/futility monitoring schedule with respect to the PSA failure endpoint:

| Analysis | Time (mo)<br>from trial | Prop.<br>Total | Cumulative<br>Total Events | Efficacy | boundary | Futil<br>bound | • |
|---|---|---|---|---|---|---|---|
| | start | events | (Both Arms) | Z> | P< | Z< | P> |
| Interim | 42 | 0.5 | 35 | 3.70 | 0.0001 | 0.00 | 0.5 |
| final | 84 | 1.00 | 70 | 1.65 | 0.05 | - | - |

#### 13.6 Gender and Minorities

Men of all races and ethnic groups are eligible for this study. Clinically important race/ethnicity differences are not expected from the intervention effect.

#### **Projected Distribution of Gender and Minorities**

| | | Gender | |
|-------------------------------------------|---------|--------|-------|
| Ethnic Category | Females | Males | Total |
| Hispanic or Latino | N/A | 27 | 27 |
| Not Hispanic or Latino | N/A | 873 | 873 |
| Ethnic Category: Total of all subjects | N/A | 900 | 900 |
| | | Gender | |
| Racial Category | Females | Males | Total |
| American Indian or Alaskan Native | N/A | 2 | 2 |
| Asian | N/A | 4 | 4 |
| Black or African American | N/A | 135 | 135 |
| Native Hawaiian or other Pacific Islander | N/A | 3 | 3 |
| White | N/A | 756 | 756 |
| Racial Category: Total of all subjects | N/A | 900 | 900 |

#### **REFERENCES (12JUN2018)**

Allibhai, S. M. D.-H., M.; Sutradar, R.; Fleshner, N.E.; Warde, P.; Cheung, A.M.; Paszat, L. (2008). "Impact of androgen deprivation therapy (ADT) on bone, cardiovascular, and endocrine outcomes: A propensity-matched analysis of 20,000 patients." J Clin Oncol(May 20 suppl; abstr 5012).

Anscher MS, Vujaskovic Z. Mechanisms and potential targets for prevention and treatment of normal tissue injury after radiation therapy. Semin Oncol. 2005;32(2 Suppl 3):S86-91.

Aouizerat BE, Dodd M, Lee K, West C, Paul SM, Cooper BA, et al. Preliminary evidence of a genetic association between tumor necrosis factor alpha and the severity of sleep disturbance and morning fatigue. Biol Res Nurs. 2009;11(1):27-41.

Attard G, Belldegrun AS, de Bono JS. Selective blockade of androgenic steroid synthesis by novel lyase inhibitors as a therapeutic strategy for treating metastatic prostate cancer. BJU Int 2005;96:1241-6.

Attard G, Reid AH, Yap TA, et al. Phase I clinical trial of a selective inhibitor of CYP17, abiraterone acetate, confirms that castration-resistant prostate cancer commonly remains hormone driven. J Clin Oncol 2008;26:4563-71

Badia X, Herdman M, Kind P. The influence of ill-health experience on the valuation of health. *Pharmacoeconomics*. 13:687-696, 1998.

Beard, C. J., Propert, K. J., Rieker, P. P., Clark, J. A., Kaplan, I., Kantoff, P. W., et al. (1997). Complications after treatment with external-beam irradiation in early-stage prostate cancer patients: a prospective multiinstitutional outcomes study. Journal of Clinical Oncology, 15(1), 223-229.

Bolla M, de Reijke TM, Van Tienhoven G, et al. Duration of androgen suppression in the treatment of prostate cancer. N Engl J Med 2009;360:2516-27.

Bolla M, Gonzalez D, Warde P, et al. Improved survival in patients with locally advanced prostate cancer treated with radiotherapy and goserelin. N Engl J Med 1997;337:295-300.

Bower, J.E. and J.E. Bower, Prevalence and causes of fatigue after cancer treatment: the next generation of research.[comment]. *Journal of Clinical Oncology*, 2005. 23(33): p. 8280-2.

Bower JE, Ganz PA, Irwin MR, Arevalo JM, Cole SW. Fatigue and gene expression in human leukocytes: increased NF-kappaB and decreased glucocorticoid signaling in breast cancer survivors with persistent fatigue. Brain Behav Immun. 2011;25(1):147-50.

Burri, RJ, Stock, RG, Cesaretti, JA, et al. Association of Single Nucleotide Polymorphisms in SOD2, XRCC1 and XRCC3 with Susceptibility for the Development of Adverse Effects Resulting from Radiotherapy for Prostate Cancer. Radiat Res, in press.

Buysse, D.J., et al., The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. *Psychiatry Research*, 1989. 28(2): p. 193-213.

Capuron L, Pagnoni G, Demetrashvili MF, Lawson DH, Fornwalt FB, Woolwine B, et al. Basal ganglia hypermetabolism and symptoms of fatigue during interferon-alpha therapy. Neuropsychopharmacology. 2007;32(11):2384-92.

Chism DB, Hanlon AL, Horwitz EM, Feigenberg SJ, Pollack A. A comparison of the single and double factor highrisk models for risk assignment of prostate cancer treated with 3D conformal radiotherapy. Int J Radiat Oncol Biol Phys 2004;59:380-5.

Collado-Hidalgo A, Bower JE, Ganz PA, Irwin MR, Cole SW. Cytokine gene polymorphisms and fatigue in breast cancer survivors: early findings. Brain Behav Immun. 2008;22(8):1197-200. PMCID: 2783767.

Damaraju, S, Murray, D, Dufour, J, *et al.* Association of DNA repair and steroid metabolism gene polymorphisms with clinical late toxicity in patients treated with conformal radiotherapy for prostate cancer. Clin Cancer Res, 2006; *12*(8): 2545-2554.

D'Amico AV, Cote K, Loffredo M, Renshaw AA, Schultz D. Determinants of prostate cancer-specific survival after radiation therapy for patients with clinically localized prostate cancer. J Clin Oncol 2002;20:4567-73.

Danjoux, C., Gardner, S., & Fitch, M. (2007). Prospective evaluation of fatigue during a course of curative radiotherapy for localised prostate cancer. Supportive Care in Cancer, 15(10), 1169-1176.

de Bono, J. S., C. J. Logothetis, et al. (2011). "Abiraterone and increased survival in metastatic prostate cancer." N Engl J Med 364(21): 1995-2005.

DeMets DL, Lan KK, 1994, Interim analysis: The alpha spending function approach, Statistics in Medicine 13: 1341-1352.

Despres JP, Lamarche B, Mauriege P, et al. Hyperinsulinemia as an independent risk factor for ischemic heart disease. N Engl J Med 1996;334:952-7.

Diggle PJ, Liang KY, Zeger SL. Analysis of longitudinal data. New York: Oxford University Press 1994.

Dignam JJ, Kocherginsky M. Choice and interpretation of statistical tests used when competing risks are present. J Clin Oncol 2008;26:4027-4034.

Dockery F, Bulpitt CJ, Agarwal S, Donaldson M, Rajkumar C. Testosterone suppression in men with prostate cancer leads to an increase in arterial stiffness and hyperinsulinaemia. Clin Sci (Lond) 2003;104:195-201.

Dreicer R, Agus D, MacVicar G, MacLean D, Zhang T, Stadler W. Safety, pharmacokinetics, and efficacy of TAK-700 in castration-resistant, metastatic prostate cancer: A phase I/II, open-label study. GU ASCO Proceedings 2010:103a.

Dreicer R, Agus D, MacVicar G, Wang J, MacLean D, Stadler W. Safety, pharmacokinetics, and efficacy of TAK-700 in metastatic, castration-resistant prostate cancer: A phase I/II, open-label study. J Clin Oncol 2010;28:3084a.

Dudbridge, F, Gusnanto, A, and Koeleman, BP Detecting multiple associations in genome-wide studies. Hum Genomics, 2006; 2(5): 310-317.

Efstathiou, J. A., K. Bae, et al. (2008). "Cardiovascular Mortality After Androgen Deprivation Therapy for Locally Advanced Prostate Cancer: RTOG 85-31." J Clin Oncol.

Efstathiou, J. A., K. Bae, et al. (2008). "Cardiovascular Mortality and Duration of Androgen Deprivation for Locally Advanced Prostate Cancer: Analysis of RTOG 92-02." Eur Urol.

Eri LM, Urdal P, Bechensteen AG. Effects of the luteinizing hormone-releasing hormone agonist leuprolide on lipoproteins, fibrinogen and plasminogen activator inhibitor in patients with benign prostatic hyperplasia. J Urol 1995;154:100-4.

Essink-Bot ML, de Koning HJ, Nijs HG, et al. Short-term effects of population-based screening for prostate cancer on health-related quality of life. J Natl Cancer Inst. 90:925-931, 1998.

Fine J, Gray R. A proportional hazards model for the subdistribution of a competing risks J Am Stat Assoc 1999;94:496-509.

Fitzgerald, R. L. and D. A. Herold (1996). "Serum total testosterone: immunoassay compared with negative chemical ionization gas chromatography-mass spectrometry." Clin Chem 42(5): 749-55.

Fransson P. Fatigue in prostate cancer patients treated with external beam radiotherapy: a prospective 5-year long-term patient-reported evaluation. J Cancer Res Ther. 2010;6(4):516-20.

Freidlin B, Korn EL, Gray R. A general inefficacy interim monitoring rule for randomized clinical trials. Clin Trials. 2010;7(3):197-208.

Freidlin B, Korn EL. Testing treatment effects in the presence of competing risks. Stat Med 2005;24:1703-1712.

Gionet, N.J. and G. Godin, Self-reported exercise behavior of employees: a validity study. *Journal of Occupational Medicine*, 1989. 31(12): p. 969-73.

Glasziou PP, Simes RJ, Gelber RD. Quality adjusted survival analysis. Stat Med. 9:1259-1276, 1990.

Godin, G., J. Jobin, and J. Bouillon, Assessment of leisure time exercise behavior by self-report: a concurrent validity study. *Canadian Journal of Public Health Revue Canadienne de Sante Publique*, 1986. 77(5): p. 359-62.

Gray RJ. A class of K-sample tests for comparing the cumulative incidence of a competing risk. *Ann Stat* 16:1141-1154, 1988.

Gulley, J. L., J. B. Aragon-Ching, et al. (2008). "Kinetics of serum androgen normalization and factors associated with testosterone reserve after limited androgen deprivation therapy for nonmetastatic prostate cancer." J Urol 180(4): 1432-7; discussion 1437.

Gulley, J. L., W. D. Figg, et al. (2005). "A prospective analysis of the time to normalization of serum androgens following 6 months of androgen deprivation therapy in patients on a randomized phase III clinical trial using limited hormonal therapy." J Urol 173(5): 1567-71.

Hall, M. C., R. J. Fritzsch, et al. (1999). "Prospective determination of the hormonal response after cessation of luteinizing hormone-releasing hormone agonist treatment in patients with prostate cancer." Urology 53(5): 898-902; discussion 902-3.

Jereczek-Fossa, B.A., H.R. Marsiglia, and R. Orecchia, Radiotherapy-related fatigue: how to assess and how to treat the symptom. A commentary. Tumori, 2001. 87(3): p. 147-51.

Kaku, H., T. Saika, et al. (2006). "Time course of serum testosterone and luteinizing hormone levels after cessation of long-term luteinizing hormone-releasing hormone agonist treatment in patients with prostate cancer." Prostate 66(4): 439-44.

Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc 53:457-481, 1958.

Keating NL, O'Malley AJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy for prostate cancer. J Clin Oncol 2006;24:4448-56.

Keating, N. L., A. J. O'Malley, et al. (2010). "Diabetes and cardiovascular disease during androgen deprivation therapy: observational study of veterans with prostate cancer." J Natl Cancer Inst 102(1): 39-46.

Korn EL, Dorey FJ. Applications of crude incidence curves. Stat Med 11:813-829, 1992.

Kyrdalen AE, Dahl AA, Hernes E, Hem E, Fossa SD. Fatigue in prostate cancer survivors treated with definitive radiotherapy and LHRH analogs. Prostate. 2010;70(13):1480-9.

Kyrdalen AE, Dahl AA, Hernes E, Cvancarova M, Fossa SD. Fatigue in hormone-naive prostate cancer patients treated with radical prostatectomy or definitive radiotherapy. Prostate Cancer Prostatic Dis. 2010;13(2):144-50.

Levegrun S, Jackson A, Zelefsky MJ, et al. Risk group dependence of dose-response for biopsy outcome after three-dimensional conformal radiation therapy of prostate cancer. Radiother Oncol 2002;63:11-26.

Lilleby, W., et al., Long-term morbidity and quality of life in patients with localized prostate cancer undergoing definitive radiotherapy or radical prostatectomy. *International Journal of Radiation Oncology, Biology, Physics*, 1999. 43(4): p. 735-43.

Little RJA. Regression with missing x's: A review. J Am Stat Assoc. 1992;87:1227-37.

Mantel N. Evaluation of survival data and two new rank order statistics arising in its consideration. *Cancer Chemotherapy Reports* 50(3): 163–70, 1966.

Miaskowski C, Dodd M, Lee K, West C, Paul SM, Cooper BA, et al. Preliminary evidence of an association between a functional interleukin-6 polymorphism and fatigue and sleep disturbance in oncology patients and their family caregivers. J Pain Symptom Manage. 2010;40(4):531-44. PMCID: 2952712.

Milne RJ, Heaton-Brown KH, Hansen P, Thomas D, Harvey V, Cubitt A. Quality-of-life valuations of advanced breast cancer by New Zealand women. Pharmacoeconomics. 2006;24(3):281-92.

Mohler J, Bahnson RR, Boston B, et al. NCCN clinical practice guidelines in oncology: prostate cancer. J Natl Compr Canc Netw 2010;8:162-200.

Monga, U., et al., Longitudinal study of quality of life in patients with localized prostate cancer undergoing radiotherapy. *Journal of Rehabilitation Research & Development*, 2005. 42(3): p. 391-9.

Monga, U., et al., Prospective study of fatigue in localized prostate cancer patients undergoing radiotherapy. *Radiation Oncology Investigations*, 1999. 7(3): p. 178-85.

Nejat, R. J., H. H. Rashid, et al. (2000). "A prospective analysis of time to normalization of serum testosterone after withdrawal of androgen deprivation therapy." J Urol 164(6): 1891-4.

Peters, CA, Stock, RG, Cesaretti, JA, et al. TGFB1 single nucleotide polymorphisms are associated with adverse quality of life in prostate cancer patients treated with radiotherapy. Int J Radiat Oncol Biol Phys, 2008; 70(3): 752-759.

Pickles, T., A. Agranovich, et al. (2002). "Testosterone recovery following prolonged adjuvant androgen ablation for prostate carcinoma." Cancer 94(2): 362-7.

Pilepich MV, Winter K, Lawton CA, et al. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys 2005;61:1285-90.

Pisansky TM, Kahn MJ, Bostwick DG. An enhanced prognostic system for clinically localized carcinoma of the prostate. Cancer 1997;79:2154-61.

Prentice RL, Kalbfleisch JD, Peterson AV Jr, Flournoy N, Farewell VT, Breslow NE. The analysis of failure times in the presence of competing risks. Biometrics. 1978;34:541-554.

Prue, G., Rankin, J., Allen, J., Gracey, J., & Cramp, F. (2006). Cancer-related fatigue: A critical appraisal. [Research Support, Non-U.S. Gov't, Review]. European Journal of Cancer, 42(7), 846-863. recommendations for permanent prostate Brachytherapy post-implant dosimetric analysis. *Int J Radiat Oncol Biol Phys*. 2000;1:221-230.

Pyorala M, Miettinen H, Laakso M, Pyorala K. Hyperinsulinemia predicts coronary heart disease risk in ealthy middle-aged men: the 22-year follow-up results of the Helsinki Policemen Study. Circulation 1998;98:398-404.

Raison CL, Borisov AS, Majer M, Drake DF, Pagnoni G, Woolwine BJ, et al. Activation of central nervous system inflammatory pathways by interferon-alpha: relationship to monoamines and depression. Biol Psychiatry. 2009;65(4):296-303. PMCID: 2655138.

Roach M, 3rd, Bae K, Speight J, *et al.* Short-term neoadjuvant androgen deprivation therapy and external-beam radiotherapy for locally advanced prostate cancer: long-term results of RTOG 8610. *J Clin Oncol* 2008;26:585-591.

Rubinstein LV, Gail MH, Santner TJ. Planning the duration of a comparative clinical trial with loss to follow-up and a period of continued observation. J Chronic Dis. 1981 34:469-79.

Ryan, J. L., J. K. Carroll, et al. (2007). "Mechanisms of Cancer-Related Fatigue." Oncologist 12(suppl 1): 22-34.

Saigal, C. S., J. L. Gore, et al. (2007). "Androgen deprivation therapy increases cardiovascular morbidity in men with prostate cancer." Cancer 110(7): 1493-500.

Sandblom G, Carlsson P, Sennfalt K, et al. A population-based study of pain and quality of life during the year before death in men with prostate cancer. Br J Cancer. 90:1163-1168, 2004.

Saylor, P. J., N. L. Keating, et al. (2011). "Gonadotropin-releasing hormone agonists and the risks of type 2 diabetes and cardiovascular disease in men with prostate cancer." Drugs 71(3): 255-61.

Saylor, P. J. and M. R. Smith (2009). "Metabolic complications of androgen deprivation therapy for prostate cancer." J Urol 181(5): 1998-2006; discussion 2007-8.

Sennfalt K, Carlsson P, Sandblom G, et al. The estimated economic value of the welfare loss due to prostate cancer pain in a defined population. Acta Oncol. 43:290-296, 2004.

Schubert, C., S. Hong, et al. (2007). "The association between fatigue and inflammatory marker levels in cancer patients: A quantitative review." Brain, Behavior, and Immunity 21(4): 413-427.

Schulz MW, Chen J, Woo HH, et al. A comparison of techniques for eliciting patient preferences in patients with benign prostatic hyperplasia. *J Urol.* 168:155-159, 2002.

Smith MR, Finkelstein JS, McGovern FJ, et al. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab 2002;87:599-603.

Smith MR, Lee H, Fallon MA, Nathan DM. Adipocytokines, obesity, and insulin resistance during combined androgen blockade for prostate cancer. Urology 2008;71:318-22.

Smith, MR, Lee, H, et al. (2006). Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab 91(4): 1305-8.

Smith MR. Changes in fat and lean body mass during androgen-deprivation therapy for prostate cancer. Urology 2004;63:742-5.

Stone, P., Hardy, J., Huddart, R., A'Hern, R., & Richards, M. (2000). Fatigue in patients with prostate cancer receiving hormone therapy. European Journal of Cancer, 36(9), 1134-1141.

Sugihara, A., O. Maeda, et al. (1998). "Expression of cytokines enhancing the osteoclast activity, and parathyroid hormone-related protein in prostatic cancers before and after endocrine therapy: an immunohistochemical study." Oncol Rep 5(6): 1389-94.

Stephens, R. J., Dearnaley, D. P., Cowan, R., Sydes, M., Naylor, S., Fallowfield, L., et al. (2007). The quality of life of men with locally advanced prostate cancer during neoadjuvant hormone therapy: data from the Medical Research Council RT01 trial (ISRCTN 47772397). BJU International, 99(2), 301-310.

Storey DJ, McLaren DB, Atkinson MA, Butcher I, Liggatt S, O'Dea R, et al. Clinically relevant fatigue in recurrence-free prostate cancer survivors. Ann Oncol. 2011.
Sydes MR, Parmar MK, James ND, Clarke NW, Dearnaley DP, Mason MD, Morgan RC, Sanders K, Royston P. Issues in applying multi-arm multi-stage methodology to a clinical trial in prostate cancer: the MRC STAMPEDE trial. Trials. 2009 Jun 11;10:39.

Symon Z, Griffith KA, McLaughlin PW, Sullivan M, Sandler HM. Dose escalation for localized prostate cancer: substantial benefit observed with 3D conformal therapy. Int J Radiat Oncol Biol Phys 2003;57:384-90.

Szymanski KM, Wei JT, Dunn RL, Sanda MG. Development and validation of an abbreviated version of the Expanded Prostate Cancer Index Composite instrument for measuring health-related quality of life among prostate cancer survivors. Urology. 2010 Mar 27. [Epub ahead of print]).

Taieb, J., B. Mathian, et al. (2003). "Testosterone measured by 10 immunoassays and by isotope-dilution gas chromatography-mass spectrometry in sera from 116 men, women, and children." Clin Chem 49(8): 1381-95.

Torres M, Liu T, Long Q, Mister D, Barsevick A, Brawley O, et al. Radiation-induced skin toxicity and cancer-related fatigue in women with breast cancer: mechanisms and mediators. Preliminary Data. 2011.

Truong, P.T., et al., Prospective evaluation of the prevalence and severity of fatigue in patients with prostate cancer undergoing radical external beam radiotherapy and neoadjuvant hormone therapy. *Canadian Journal of Urology*, 2006. 13(3): p. 3139-46.

U.S. Department of Health and Human Services, National Institutes of Health National Cancer Institute. Common Terminology Criteria for Adverse Events (CTCAE). Version 4.02. 28 May 2009.

van Andel G, Kurth KH. The impact of androgen deprivation therapy on health related quality of life in asymptomatic men with lymph node positive prostate cancer. *Eur Urol.* 44:209-214, 2003.

Voerman, B., Fischer, M., Visser, A., Garssen, B., van Andel, G., & Bensing, J. (2006). Health-related quality of life in Dutch men with prostate cancer. Journal of Psychosocial Oncology, 24(2), 49-64.

Wang, C., D. H. Catlin, et al. (2004). "Measurement of total serum testosterone in adult men: comparison of current laboratory methods versus liquid chromatography-tandem mass spectrometry." J Clin Endocrinol Metab 89(2): 534-43.

Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology 2000;56(6):899-905.

Wildi SM, Cox MH, Clark LL, Turner R, Hawes RH, Hoffman BJ, Wallace MB. Assessment of health state utilities and quality of life in patients with malignant esophageal Dysphagia. Am J Gastroenterol. 2004 Jun;99(6):1044-91

Wu MC, Bailey K. Analyzing changes in the presence of informative right censoring caused by death and withdrawal. Stat Med. 1988;7:337-46.

Wu AW, Jacobson KL, Frick KD, et al. Validity and responsiveness of the Euroqol as a measure of health related quality of life in people enrolled in an AIDS clinical trial. *Qual Life Res.* 11:273-282, 2002.

Zelen M. The randomization and stratification of patients to clinical trials. J Chronic Dis. 1974;27:365-75.

# APPENDIX I, STUDY PARAMETER TABLE: PRE-TREATMENT ASSESSMENTS (4/16/14)

| Note: See Sections 3.0 | and <u>4.0</u> (pre-s | tudy entry) fo | r details and/o | r exceptions to | this table. |
|---|---|---|---|---|---|
| Assessments (may be required for eligibility) | w/in 180<br>days prior to<br>registration | w/in 90 days<br>prior to<br>registration | w/in 60 days<br>prior to<br>registration | w/in 21 days<br>(3 weeks)<br>prior to<br>registration | w/in 14 days<br>(2 weeks)<br>prior to<br>registration |
| Biopsy | Χ | | | | |
| History/physical | | | Х | | |
| Ht/Wt/PS | | | | Х | |
| PSA | Х | | | | |
| CBC/diff | | | | | Х |
| Chemistry & liver panels | | | | Х | |
| Testosterone (standard assay unless otherwise noted) | | | | Х | |
| Note: Collect blood for<br>testosterone in the a.m. at<br>same time of day as<br>collection of fasting<br>insulin/ fasting glucose/<br>fasting lipids/hemoglobin<br>A1C | | | | | |
| Fasting glucose/ fasting lipids/ hemoglobin A1C | | | | X | |
| Note: Collect blood in the a.m. at same time of day as collection of testosterone | | | | | |
| Fasting insulin (ship specimen to UCSF BSR) | | | | X | |
| Note: Collect blood in the a.m. at same time of day as collection of testosterone | | | | | |
| MUGA scan or echocardiogram | | F | rior to registrat | ion | |
| Bone scan | | X | | | |
| CT or MRI | | Х | | | |
| Transrectal ultrasound and AUA | | | X (for<br>brachy<br>patients<br>only) | | |
| -Continued on next page- | | | | | |

| APPENDIX I, STUDY PARAMETER TABLE: PRE-TREATMENT ASSESSMENTS continued | | | | | |
|---|---|---|---|---|---|
| <u>Note</u> : See <u>Sections 3.0</u> and <u>4.0</u> (pre-study entry) for details and/or exceptions to this table. | | | | | |
| Assessments (may | w/in 180 | w/in 90 days | w/in 60 days | w/in 21 days | w/in 14 days |
| be required for | days prior to | prior to | prior to | (3 weeks) | (2 weeks) |
| eligibility) | registration | registration | registration | prior to | prior to |
| | | | | registration | registration |
| Review of | | | At registration | 1 | |
| medications | | | | | |
| *Clinical | | X* | | | |
| survivorship | | | | | |
| †PROMIS-fatigue, | | | | | |
| EPIC, EQ-5D, | Pre-treatment | | | | |
| PSQI/GLTEQ (if | | | | | |
| patient consents) | | | | | |
| Tissue for banking | | | | | |
| (if patient consents) | Pre-treatment | | | | |
| †Blood for | | | | | |
| banking/QOL (if | Pre-treatment (see also <u>Section 10.0</u> for specific collection requirements) | | | | |
| patient consents) | | | | | |
| *See Section 1.0 of pr | otocol under Ev | aluation of Clinic | cal and Chronic | Disease Outcome | es (1st |
| sentence). | | | | | |
| †Blood (Plasma & who | ole blood) collec | tion is mandator | y for patients pa | rticipating in QOL | |
| -Continued on next p | page- | | | | |

APPENDIX I, STUDY PARAMETER TABLE: ASSESSMENTS DURING TREATMENT (12/17/13)

Note: See Sections 10.0 (specimen collection), and 11.1 (during treatment) for details and/or exceptions to this table.

| Assessments During 24 months of ADT +/- TAK-700 30 months | | | | | |
|---|---|---|---|---|---|
| | q 1 | q 3 | 12 months | 24 months | 1 |
| | month | months | | | |
| History/physical | | Χ | | | |
| Ht/Wt/PS | | Χ | | | |
| PSA | | X | | | X |
| Chemistry & liver panels | <u>See</u><br>11.1 | <u>See</u><br>11.1 | | | |
| Testosterone (standard assay unless otherwise | | | X (by LC/MS/MS; ship specimen to | X (by LC/MS/MS; ship specimen to | Х |
| noted) | | | NRG Oncology Biospecimen | NRG Oncology Biospecimen | |
| Note: Collect blood for testosterone in the a.m. at | | | Bank) | Bank) | |
| same time of day as collection of fasting insulin/ | | | | | |
| fasting glucose/ fasting | | | | | |
| lipids/hemoglobin A1C Fasting glucose/ fasting | | | X | X | |
| lipids/hemoglobin A1C | | | X | ^ | |
| Note: Collect blood in the | | | | | |
| a.m. at same time of day as collection of testosterone | | | | | |
| Fasting insulin (ship | | | Х | Χ | |
| specimen to UCSF BSR) | | | | | |
| Note: Collect blood in the | | | | | |
| a.m. at same time of day as | | | | | |
| collection of testosterone | | | | | |
| Review of medications | | Χ | | | |
| AE evaluation | Χ | | | | |
| *Clinical survivorship | | Х | | | |
| †PROMIS-fatigue, EPIC,<br>EQ-5D, PSQI/GLTEQ (if<br>patient consents) | (1) In the week prior to RT start; (2) during the last week of RT; (3) at 1 year (12 months) after therapy starts | | | | |
| †Blood for banking/QOL (if patient consents) | At 1 year (12 months) after therapy starts (see also <u>Section 10.0</u> for specific collection requirements) | | | | |

<sup>\*</sup>See <u>Section 1.0</u> of protocol under Evaluation of Clinical and Chronic Disease Outcomes (1st sentence).

†Blood (Plasma & whole blood) collection is mandatory for patients participating in QOL.

-Continued on next page-

| ADDENDIY | CTUDY DADAMETED TABLE. FOLLOW III | D ACCECCMENTS (40/47/42) |
|---|---|---|
| | STUDY PARAMETER TABLE: FOLLOW UNITED IN 1981 11.0 (Specimen collection), and 11.1 (duals 11.1) | |
| <u>note</u> . See <u>Section</u> | exceptions to this table. | ing treatment, for details and/or |
| Assessments | Follow Up (beginning | g at 36 months) |
| | q 6 months for 3 years and then annually | q 12 months for 3 years |
| History/physical | X | |
| Ht/Wt/PS | X | |
| PSA | X | |
| Testosterone | | X |
| (standard assay | | |
| unless otherwise | | |
| noted) | | |
| Note: Collect blood | | |
| for testosterone in | | |
| the a.m. at same | | |
| time of day as | | |
| collection of fasting | | |
| insulin/ fasting | | |
| glucose/ fasting | | |
| lipids/hemoglobin | | |
| A1C | | |
| Fasting glucose/ | | X |
| fasting lipids/ | | |
| hemoglobin A1C | | |
| Note: Collect blood | | |
| in the a.m. at same | | |
| time of day as | | |
| collection of | | |
| testosterone | | |
| Fasting insulin (ship | | X |
| specimen to UCSF | | |
| BSR) | | |
| Note: Collect blood | | |
| in the a.m. at same | | |
| time of day as | | |
| collection of | | |
| testosterone | | |
| Bone scan | As clinically indicated, q 6 mc | onths after PSA relapse |
| AE evaluation | X | |

-Continued on next page-

APPENDIX I, STUDY PARAMETER TABLE: FOLLOW UP ASSESSMENTS continued (12/17/13)

Note: See Sections 10.0 (specimen collection), and 11.1 (during treatment) for details and/or exceptions to this table.

| | exceptions to tins tab | 101 |
|---|---|---|
| Assessments | Follow Up (beginning at 36 months) | |
| | q 6 months for 3 years and then annually | q 12 months for 3 years |
| *Clinical | X | |
| survivorship | | |
| †PROMIS-<br>fatigue, EPIC,<br>EQ-5D,<br>PSQI/GLTEQ<br>(if patient<br>consents) | At 2.5 years (30 months | s) after therapy starts |
| †Blood for<br>banking/QOL<br>(if patient<br>consents) | At 2.5 years (30 months) after therapy starts (see also <u>Section 10.0</u> for specific collection requirements) | |

<sup>\*</sup>See <u>Section 1.0</u> of protocol under Evaluation of Clinical and Chronic Disease Outcomes (1st sentence).

†Blood (Plasma and whole blood) collection is mandatory for patients participating in QOL.

# **APPENDIX II**

# **ZUBROD PERFORMANCE SCALE**

| 0 | Fully active, able to carry on all predisease activities without restriction |
|---|---|
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry work of a light or sedentary nature. For example, light housework, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair 50% or more of waking hours |
| 4 | Completely disabled. Cannot carry on self-care. Totally confined to bed |
| 5 | Death |

### APPENDIX III Staging System, Prostate, 7<sup>th</sup> Edition **DEFINITIONS OF TNM**

#### **Primary Tumor, Clinical (T)**

- Primary tumor cannot be assessed
- T0 No evidence of primary tumor
- T1 Clinically inapparent tumor neither palpable nor visible by imaging
  - T1a Tumor incidental histologic finding in 5% or less of tissue resected
  - T1b Tumor incidental histologic finding in more than 5% of tissue resected
  - Tumor identified by needle biopsy (e.g., because of elevated PSA) T1c
- T2 Tumor confined with prostate\*
  - T2a Tumor involves one-half of one lobe or less
  - T2b Tumor involves more than one-half of one lobe but not both lobes
  - T2c Tumor involves both lobes
- T3 Tumor extends through the prostate capsule\*\*
  - Extracapsular extension (unilateral or bilateral) T3a
  - T3b Tumor involves the seminal vesicle(s)
- T4 Tumor is fixed or invades adjacent structures other than seminal vesicles such as external sphincter, rectum, bladder, levator muscles and/or pelvic wall

\*Note: Tumor found in one or both lobes by needle biopsy, but not palpable or reliably visible by imaging, is classified as T1c

\*\*Note: Invasion into the prostatic apex or into (but not beyond) the prostatic capsule is classified not as T3 but as T2.

#### Primary Tumor, Pathologic (pT) \*

- pT2 Organ confined
  - pT2a Unilateral, one-half of one side or less
  - pT2b Unilateral, involving more than one-half of side but not both sides
  - pT2c Bilateral disease
- pT3 Extraprostatic extension
  - pT3a Extraprostatic extension or microscopic invasion of bladder neck\*\*
  - pT3b Seminal vesicle invasion
- pT4 Invasion of rectum, levator muscles, and/or pelvic wall

\*Note: There is no pathologic T1 classification

\*\*Note: Positive surgical margin should be indicated by an R1 descriptor (residual microscopic disease).

#### Regional Lymph Nodes (N)

#### Clinical

NX Regional lymph nodes were not assessed N0 No regional lymph node metastasis

Metastasis in regional lymph node(s) N1

#### **Pathologic**

Regional nodes not sampled pNX

No positive regional nodes pN0

pN1 Metastases in regional node(s)

# APPENDIX III Staging System, Prostate, 7<sup>th</sup> Edition DEFINITIONS OF TNM

#### Distant Metastasis (M)\*

M0 No distant metastasis
M1 Distant metastasis

M1a Nonregional lymph node(s)

M1b Bone(s)

M1c Other site(s) with or without bone disease

\*Note: When more than one site of metastasis is present, the most advanced category is used; pM1c is most advanced.

#### Histologic Grade (G)

 $\begin{array}{ll} \text{Gleason X} & \text{Gleason score cannot be processed} \\ \text{Gleason} \leq 6 & \text{Well-differentiated (slight anaplasia])} \end{array}$ 

Gleason 7 Moderately differentiated (moderate anaplasia)

Gleason 8-10 Poorly differentiated/undifferentiated (marked anaplasia)

# **Anatomic Stage/Prognostic Groups\***

| Stage I | T1a-c | N0 | M0 | PSA <10 | Gleason ≤6 |
|---|---|---|---|---|---|
| | T2a | N0 | M0 | PSA <10 | Gleason ≤6 |
| | T1-2a | N0 | M0 | PSA X | Gleason X |
| Stage IIA | T1a-c<br>T1a-c<br>T2a<br>T2b<br>T2b | N0<br>N0<br>N0<br>N0<br>N0 | M0<br>M0<br>M0<br>M0<br>M0 | PSA <20<br>PSA ≥10<20<br>PSA <20<br>PSA <20<br>PSA X | Gleason 7<br>Gleason ≤6<br>Gleason ≤7<br>Gleason X |
| Stage IIB | T2c | N0 | M0 | Any PSA | Any Gleason |
| | T1-2 | N0 | M0 | PSA ≥20 | Any Gleason |
| | T1-2 | N0 | M0 | Any PSA | Gleason ≥8 |
| Stage III | T3a-b | N0 | MO | Any PSA | Any Gleason |
| Stage IV | T4 | N0 | M0 | Any PSA | Any Gleason |
| | Any T | N1 | M0 | Any PSA | Any Gleason |
| | Any T | Any N | M1 | Any PSA | Any Gleason |

<sup>\*</sup>Note: When either PSA or Gleason is not available, grouping should be determined by T stage and/or either PSA or Gleason as available.

Source: Edge, SB, ed. AJCC Cancer Staging Manual. 7<sup>th</sup> ed. New York, NY: Springer; 2010.

# APPENDIX IV New York Heart Association Classification of Cardiac Disease

The following table presents the NYHA classification of cardiac disease.

| Class | Functional Capacity | Objective<br>Assessment |
|---|---|---|
| I | Patients with cardiac disease but without resulting limitations of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain. | No objective evidence of cardiovascular disease. |
| II | Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain. | Objective evidence of minimal cardiovascular disease. |
| III | Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. | Objective evidence of moderately severe cardiovascular disease. |
| IV | Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased. | Objective evidence of severe cardiovascular disease. |

Source: The Criteria Committee of New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th Ed. Boston, MA: Little, Brown & Co; 1994:253-256.

# APPENDIX V (12JUN2018) APPENDICES FOR NRG ONCOLOGY BIOSPECIMEN COLLECTION (as specified by the protocol)

#### **Shipping Instructions:**

U.S. Postal Service Mailing Address: For FFPE or Non-frozen Specimens Only NRG Oncology Biospecimen Bank University of California San Francisco Campus Box 1800 2340 Sutter Street, Room S341 San Francisco, CA 94143-1800

Courier Address (FedEx, UPS, etc.): <u>For ALL Frozen or Trackable Specimens</u> NRG Oncology Biospecimen Bank University of California San Francisco 2340 Sutter Street, Room S341 San Francisco, CA 94115

- □ Include all NRG Oncology paperwork in pocket of biohazard bag.
- □ Check that the Specimen Transmittal Form has the consent boxes checked off.
- □ Check that all samples are labeled with the RTOG (NRG) study and case number, and include date of collection as well as collection time point (e.g., pretreatment, post-treatment).

#### □ FFPE Specimens:

- Slides should be shipped in a plastic slide holder/slide box. Place a small wad of padding in top of the container. If you can hear the slides shaking it is likely that they will break during shipping.
- FFPE Blocks can be wrapped with paper towel, or placed in a cardboard box with padding. Do not wrap blocks with bubble wrap or gauze. Place padding in top of container so that if you shake the container the blocks are not shaking. If you can hear the block shaking, it might break during shipping.
- Slides, Blocks, or Plugs can be shipped ambient or with a cold pack either by United States Postal Service (USPS) to the USPS address (94143) or by Courier to the Street Address (94115). Do NOT ship on Dry Ice.

#### □ Frozen Specimens:

- Multiple cases may be shipped in the same cooler, but make sure each one is in a separate bag and clearly identified. If possible keep Serum, Plasma, Whole Bloods in separate bags.
- Place specimens and absorbent shipping material in Styrofoam cooler filled with dry ice (at least 7 lbs).
   There should be plenty of dry ice under and above the specimens. If the volume of specimens is greater than the volume of dry ice then ship in a larger Styrofoam box, or two separate boxes. Any Styrofoam box can be used, as long as it is big enough.
- Specimens received thawed due to insufficient dry ice or shipping delays will be discarded and the site will be notified.
- Send frozen specimens on Dry Ice via overnight courier to the address above. Specimens should only be shipped Monday through Wednesday (Monday-Tuesday for Canada) to prevent thawing due to delivery delays. Saturday or holiday deliveries cannot be accepted. Samples can be stored frozen at -80° C until ready to ship.
- □ For Questions regarding collection/shipping please contact the NRG Oncology Biospecimen Bank by e-mail: NRGBB@ucsf.edu or phone: 415-476-7864 or Fax: 415-476-5271.

### **APPENDIX V (continued)**

# NRG ONCOLOGY BLOOD COLLECTION KIT INSTRUCTIONS (12/17/13)

Note: There is a separate appendix for PBMC preparation not included in this instruction (See Appendix VI). This Kit is for collection, processing, storage, and shipping of serum, plasma, or whole blood (as specified by the protocol):

#### Kit contents:

- Red Top tubes for mandatory serum shipped separate (A)
- Three Purple Top EDTA tubes for plasma (B)
- One Purple Top EDTA tube for Whole Blood (C)
- Thirty-five (35) 1 ml cryovials
- Biohazard bags (2) and Absorbent shipping material (2)
- Styrofoam container (inner) and Cardboard shipping (outer) box
- UN1845 DRY Ice Sticker and UN3373 Biological Substance Category B Stickers
- Specimen Transmittal Form and Kit Instructions

### PREPARATION AND PROCESSING OF SERUM, PLASMA AND WHOLE BLOOD:

# (A) Serum (if requested): Red Top Tube

□ Label as many 1ml cryovials (5 to 10) as necessary for the serum collected. Label them with the RTOG (NRG) study and case number, collection date, time, and time point, and clearly mark cryovials "serum".

### **Process**:

- 1. Allow one red top tube to clot for 30 minutes at room temperature.
- 2. Spin in a standard clinical centrifuge at ~2500 RPM for 10 minutes at 4°C (preferred). If sites are unable to process samples at 4°C then spinning at room temperature is acceptable if done within 2 hours of draw but must be noted on the Specimen Transmittal Form.
- 3. Aliquot <u>0.5 ml serum</u> into as many cryovials as are necessary for the serum collected (5 to 10) labeled with RTOG (NRG) study and case numbers, collection date/time, protocol time-point collected (e.g. pretreatment, post-treatment), and clearly mark specimen as "serum".
- 4. Place cryovials into biohazard bag and immediately freeze at -70 to -90° C, and store frozen until ready to ship. See below for storage conditions.
- 5. Store serum at -70 to -90° C until ready to ship on dry ice. See below for storage conditions.

# PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED and include collection time point on the STF.

#### (B) Plasma (If requested): Purple Top EDTA tube #1

□ Label as many 1ml cryovials (5 to 10) as necessary for the plasma collected. Label them with the RTOG (NRG) study and case number, collection date, time, and time point, and clearly mark cryovials "plasma".

#### Process:

- 1. After collection, invert tube(s) multiple times to ensure adequate mixing of EDTA.
- 2. Centrifuge specimen(s) within one hour of collection in a standard clinical centrifuge at ~2500 RPM for 10 minutes at 4°C (preferred). If sites are unable to process samples at 4°C then spinning at room temperature is acceptable if done within 2 hours of draw but must be noted on the STF..
- 3. If the interval between specimen collection and processing is anticipated to be more than one hour, keep specimen on ice until centrifuging is performed.
- 4. Carefully pipette and aliquot <u>0.5 ml plasma</u> into as many cryovials as are necessary for the plasma collected (5 to 10) labeled with RTOG (NRG) study and case numbers, collection date/time, time point collected and clearly mark specimen as "plasma". Avoid pipetting up the buffy coat layer.
- 5. Place cryovials into biohazard bag and immediately freeze at -70 to -90°C.
- 6. Store frozen plasma until ready to ship on dry ice.
- 7. See below for storage conditions.

PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED and include collection time point on the Specimen Transmittal Form. (continued on next page)

#### **APPENDIX V**

### NRG ONCOLOGY BLOOD COLLECTION KIT INSTRUCTIONS (continued)



# (C) Whole Blood for DNA (if requested): Purple Top EDTA tube #2

□ Label as many 1ml cryovials (3 to 5) as necessary for the whole blood collected. Label them with the RTOG (NRG) study and case number, collection date/time, and time point, and clearly mark cryovials "blood".

#### **Process**:

- 1. After collection, invert tube(s) multiple times to ensure adequate mixing of EDTA. Blood can also be mixed for 5 minutes on a mixer at room temperature.
- 2. Carefully pipette and aliquot **1.0 ml blood** into as many cryovials as are necessary for the blood collected (3 to 5) labeled with RTOG (NRG) study and case numbers, collection date/time, time point collected and clearly mark specimen as "blood".
- 3. Place cryovials into biohazard bag and freeze immediately at -70 to -80° Celsius.
- 4. Store blood samples frozen until ready to ship on dry ice.
- 5. See below for storage conditions.

# PLEASE MAKE SURE THAT EVERY SPECIMEN IS LABELED and include collection time point on Specimen Transmittal Form.

#### Freezing and Storage:

- ☐ Freeze Blood samples in a -80°C Freezer or on Dry Ice or snap freeze in liquid nitrogen.
- $\,\square\,$  Store at –80°C (-70°C to -90°C) until ready to ship.

If a -80°C Freezer is not available,

 Samples can be stored short term in a -20°C freezer (non-frost free preferred) for up to one week (please ship out Monday-Wednesday only; Canada: Monday-Tuesday only).

#### OR:

Samples can be stored in plenty of dry ice for up to one week, replenishing daily (please ship out on Monday-Wednesday only; Canada: Monday-Tuesday only).

#### OR:

- Samples can be stored in liquid nitrogen vapor phase (ship out Monday-Wednesday only);
   Canada: Monday-Tuesday only).
- □ Please indicate on Specimen Transmittal Form the storage conditions used and time stored.

# **Shipping/Mailing:**

- Ship specimens on Dry Ice overnight **Monday-Wednesday (Monday-Tuesday from Canada)** to prevent thawing due to delivery delays. Saturday and holiday deliveries cannot be accepted.
- Include all NRG Oncology paperwork in a sealed plastic bag and tape to the outside top of the Styrofoam box.
- Wrap frozen specimens of same type (i.e., all serum together, plasma together and whole bloods together) in absorbent shipping material and place each specimen type in a separate biohazard bag.
   (continued on next page)

#### **APPENDIX V (12Jun2018)**

# RTOG BLOOD COLLECTION KIT INSTRUCTIONS (continued)

- □ Place specimen bags into the Styrofoam cooler and fill with plenty of dry ice (7-10 lbs/3.5kg minimum). *Add padding to avoid the dry ice from breaking the tubes.*
- Place Styrofoam coolers into outer cardboard box, and attach shipping label and UN3373 and UN1895 stickers to outer cardboard box.
- □ Multiple cases may be shipped in the same cooler, but make sure each one is in a separate bag and that there is enough room for plenty of dry ice. Add padding to avoid the dry ice from breaking the tubes.
- □ For questions regarding collection, shipping or to order a Blood Collection Kit, please e-mail NRGBB@ucsf.eduor call (415) 476-7864.

### **Shipping Address:**

Courier Address (FedEx, UPS, etc.): For all Frozen Specimens NRG Oncology Biospecimen Bank University of California San Francisco 2340 Sutter Street, Room S341 San Francisco, CA 94115 For questions, call 415-476-7864 or e-mail: NRGBB@ucsf.edu

### **APPENDIX VI** (12JUN2018)

# PBMC PREPARATION INSTRUCTIONS Peripheral blood mononuclear cell (PBMC) isolation

- 1. Collect whole blood into one lavender top tube (EDTA tube #3), invert to mix (total volume about 6 ml per tube). **Keep blood at room temperature (RT)**.
- 2. Within 10 mins if possible (no more than 2 hours), transfer the whole blood from collection tubes into a 50 ml conical tube. Note the volume of blood.
- 3. Dilute whole blood. Adjust blood volume to 1:1 with 1X Dulbeccos-PBS (CMF Free) (e.g. 6 whole blood + 6 ml 1X PBS), invert to mix.
- 4. Add 5 ml lymphocyte separation medium (LSM) per 15 ml conical tube.
- 5. Carefully add <u>the diluted whole blood</u> on the top of LSM using the disposable blunt tip transfer pipette, pipetting slowly alongside of the tube to get two layers. Do not mix diluted whole blood with LSM. <u>Note</u>: If you have more diluted blood than will fit in a single tube, you can divide it into two tubes so as not to waste any sample.
- 6. Carefully transfer the tube with diluted whole blood/LSM into a swing bucket centrifuge. Spin at 705 RCF for 10 minutes, RT, with the brake off. The figure below shows what to expect. (Note: Ficoll is another type of LSM).



- 7. Collect PBMCs with a disposable thin tip transfer pipet, and deposit to a new 15ml tube.
- 8. Wash cells: bring volume in the tubes up to 14ml with 1X PBS (still RT).
- 9. Centrifuge for 10 mins at 194 RCF, RT, brake on.

(continued on next page)

#### **APPENDIX VI**

# PBMC PREPARATION INSTRUCTIONS (continued) Peripheral blood mononuclear cell (PBMC) isolation

- 10. Discard supernatant and wash again with 14ml of 1X PBS, RT.
- 11. Centrifuge for 10 mins again at 194 RCF, RT, brake on.
- 12. Discard the supernatant. Re-suspend the pellet by gently flicking the bottom of the tube. Transfer the pellet by re-suspending it using 0.5-1.0 mL of the freezering serum mix and add this back to the cryovial containing the remaining freezing serum mix (FBS + 10% DMSO).
- 13. Store immediately at -80°C in 2 ml cryovial. Samples must then be kept at -80°C during storage and shipping.

#### 14. SHIPPING INSTRUCTIONS:

- □ Ship specimens on Dry Ice overnight **Monday-Wednesday (Monday-Tuesday from Canada)** to prevent thawing due to delivery delays. Saturday and holiday deliveries cannot be accepted.
- □ Include all NRG Oncology paperwork in a sealed plastic bag and tape to the outside top of the Styrofoam box.
- □ Wrap frozen specimens in absorbent shipping material, and place inside zip-lock biohazard bags. Place specimen bags into the Styrofoam cooler and fill with plenty of dry ice (7-10 lbs/3.5kg minimum). *Add padding to avoid the dry ice from breaking the tubes.*
- Place Styrofoam coolers into outer cardboard box, and attach shipping label and UN3373 and UN1895 stickers to outer cardboard box.
- □ For questions regarding *collection or processing of PBMC*'s please e-mail RTOG@emory.edu or call (404) 778-5564.
- □ To order a kit please contact the NRG Oncology Biospecimen Bank at NRGBB@ucsf.edu
- □ or call (415) 476-7864

#### **Shipping Address:**

Courier Address (FedEx, UPS, etc.): For all Frozen Specimens NRG Oncology Biospecimen Bank University of California San Francisco 2340 Sutter Street, Room S341 San Francisco, CA 94115 Phone: +1 415-476-7864

(continued on next page)

#### **APPENDIX VI**

# PBMC PREPARATION INSTRUCTIONS (continued) Peripheral blood mononuclear cell (PBMC) isolation

# PBMC Collection Kit Contents

Lavender top tubes: Becton Dickson 366450

1X PBS: Store at room temperature or 4C until ready for use. Keep sterile.

50 ml conical tube: Becton Dickson 352070

*lymphocyte separation medium:* Mediatech 25-072-CL - Store at room temperature.

disposable blunt tip transfer pipettes: Fisher 13-711-7M

disposable thin tip transfer pipettes: Thermo Scientific Samco 232

15 ml conical tubes: Becton Dickson 352097

1.5 mls Freezing medium in 2ml Cryovials: (store frozen until ready to use)(90% Fetal Bovine Serum, Hyclone SH30071.03; 10% DMSO, Sigma D2650)

### **APPENDIX VII**

# **MONTHLY PILL DIARY FOR RTOG 1115 TAK-700**

| Sunday | Monday | Tuesday | Wednesday | Thursday | Friday | Saturday |
|---|---|---|---|---|---|---|
| Date: | Date: | Date: | Date: | Date: | Date: | Date: |
| AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| Date: | Date: | Date: | Date: | Date: | Date: | Date: |
| AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| | | | _ | | _ | |
| Date: | Date: | Date: | Date: | Date: | Date: | Date: |
| AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| Date: | Date: | Date: | Date: | Date: | Date: | Date: |
| AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| Date: | Date: | Date: | Date: | Date: | Date: | Date: |
| AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE | AM DOSE |
| 300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |
| Journal Transfer of the Control of t | | | <u> </u> | | | |
| | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE | PM DOSE |
| PM DOSE<br>300mg | 300mg | 300mg | 300mg | 300mg | 300mg | 300mg |

# Patient Instructions:

Place a (✓) next to each dose taken on a daily basis. If you were instructed to take a different daily dose, write that dose in the box. If you missed a dose or a day, indicate that by placing an 'M' after the dose rather than a (✓).

Be sure to bring your <u>pill bottles and</u> <u>diaries</u> with you for your return appointment.

# Return appointment date:

| 1 | 1 |
|---|---|
| / | / |

| 1115/<br>Study number/case number | Date |
|-----------------------------------|------|
| Comments | |

<sup>\*\*</sup>Please file this diary in the patient's research chart. Do not mail to NRG Oncology.